The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for Study 201928: A randomised, double-blind, placebo-controlled study to evaluate the safety, efficacy and changes in induced sputum and blood biomarkers following daily repeat doses of inhaled GSK2269557 for 12 weeks in adult subjects diagnosed with an acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD). |
|---|---|---|
| <b>Compound Number</b> | : | GSK2269557 |
| Effective Date | : | 09-JAN-2019 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 201928.
- This RAP is intended to describe the pharmacodynamic/biomarker, safety, pharmacokinetic and efficacy analyses required for the study.
- This version of the RAP includes amendments to the originally approved RAP.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### RAP Author(s):

| Approver | |
|-----------------|----------------------|
| PPD | |
| Statistician (C | Clinical Statistics) |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Review Confirmation:**

| Approver | | Date | Approval Method |
|---|---|---|---|
| PPD | | | |
| - | ntable Person (Clinical | 09-Jan-2019 | Email |
| Development | ) | | |
| PPD | | 00 1 2010 | T:1 |
| Principal Programmer (Clinical Programming) | | 09-Jan-2019 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|--------------------------------|-------------|-----------------|
| Director (Clinical Statistics) | 09-Jan-2019 | eSignature |
| Manager (Clinical Programming) | 09-Jan-2019 | eSignature |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 6 |
| 2. | CLIMA | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objective(s) and Endpoint(s) | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.4. | Statistical Analyses | |
| | ۷.4. | 2.4.1. Primary Analyses | |
| | | 2.4.1. Filliary Ariaryses | 10 |
| 3. | PLAN | NED ANALYSES | 10 |
| | 3.1. | Final Analyses | 10 |
| 4. | ANAL | YSIS POPULATIONS | 10 |
| | 4.1. | Protocol Deviations | 11 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | 12 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.1.<br>5.2. | | |
| | 5.2.<br>5.3. | Baseline Definitions | |
| | 5.3. | Examination of Covariates and Subgroups | |
| | | 5.3.1. Covariates and Other Strata | |
| | - A | 5.3.2. Examination of Subgroups | 14 |
| | 5.4. | Other Considerations for Data Analyses and Data Handling Conventions | 14 |
| 6. | STUD | Y POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | 15 |
| 7. | PHAR | RMACODYNAMIC AND BIOMARKER ANALYSES | 15 |
| | 7.1. | Primary Pharmacodynamic and Biomarker Analyses | 15 |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | 16 |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Statistical Analyses / Methods | |
| | | 7.1.4.1. Statistical Methodology Specification | |
| | 7.2. | Exploratory Pharmacodynamic and Biomarker Analyses | |
| | | 7.2.1. Éndpoint / Variables | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Statistical Analyses / Methods | |
| 8. | FFFIC | CACY ANALYSES | 10 |
| ٥. | 8.1. | Secondary Efficacy Analyses (Not From HRCT Analyses) | |
| | 0.1. | 8.1.1. Endpoint / Variables | |
| | | 8.1.2. Summary Measure | |
| | | 8.1.3. Population of Interest | |
| | | 8.1.4. Statistical Analyses / Methods | |
| | | 8.1.4.1. Statistical Methodology Specification | |

| | 8.2. | Seconda<br>8.2.1.<br>8.2.2. | ary Efficacy Analyses (From HRCT Analyses) Endpoint / Variables | 21 |
|---|---|---|---|---|
| | | 8.2.2.<br>8.2.3. | Summary Measure Population of Interest | |
| | | 8.2.4. | Statistical Analyses / Methods | |
| | | 0.2.4. | 8.2.4.1. Statistical Methodology Specification | |
| | 8.3. | Explorate | ory Efficacy Analyses (From HRCT Analyses) | |
| | 0.0. | 8.3.1. | Endpoint / Variables | |
| | | 8.3.2. | Summary Measure | |
| | | 8.3.3. | Population of Interest | |
| | | 8.3.4. | Statistical Analyses / Methods | |
| | | | 8.3.4.1. Statistical Methodology Specification | |
| | 8.4. | Explorate | ory Efficacy Analyses (Not from HRCT Analyses) | 32 |
| | | 8.4.1. | Endpoint / Variables | |
| | | 8.4.2. | Summary Measure | |
| | | 8.4.3. | Population of Interest | 32 |
| | | 8.4.4. | Statistical Analyses / Methods | 33 |
| 9. | | | P BETWEEN THE PHARMACODYNAMIC AND | |
| | | | ATA AND THE HRCT DATA | |
| | 9.1. | Relations | ship between the mRNA data and the HRCT data | 33 |
| 40 | 0.455 | <del>-</del> \/ | YSES | 22 |
| 10. | | | Events Analyses | |
| | 10.1. | | _aboratory Analyses | |
| | 10.2. | | afety Analyses | |
| | 10.5. | Ourier Ge | alety Allalyses | |
| 11. | PHARMACOKINETIC ANALYSES | | | |
| | | | ary Pharmacokinetic Analyses | |
| | | 11.1.1. | Endpoint / Variables | |
| | | | 11.1.1.1 Drug Concentration Measures | 34 |
| | | | 11.1.1.2. Derived Pharmacokinetic Parameters | 34 |
| | | 11.1.2. | Summary Measure | 34 |
| | | 11.1.3. | Population of Interest | 34 |
| 12. | REFE | RENCES. | | 35 |
| 12 | ∧ DDE1 | VIDICES | | 36 |
| 13. | 13.1. | | x 1: Protocol Deviation Management | |
| | 10.1. | 13.1.1. | Important Protocol Deviations | |
| | 13.2. | - | x 2: Schedule of Activities | |
| | 10.2. | 13.2.1. | | |
| | 13.3. | | x 3: Assessment Windows | |
| | 10.0. | 13.3.1. | | |
| | 13.4. | | x 4: Study Phases and Treatment Emergent Adverse | |
| | | | , | 42 |
| | | 13.4.1. | Study Phases | 42 |
| | | | 13.4.1.1. Study Phases for Concomitant Medication | |
| | | 13.4.2. | Treatment States for Adverse Events | |
| | 13.5. | | x 5: Data Display Standards & Handling Conventions | |
| | | 13.5.1. | 1 5 | |
| | | 13.5.2. | Reporting Standards | 43 |

| | 13.5.3. | Reporting Standards for Pharmacokinetic | .44 |
|--------|----------|-------------------------------------------------|-----|
| 13.6. | Appendix | 6: Derived and Transformed Data | 45 |
| | 13.6.1. | General | 45 |
| | 13.6.2. | Study Population | .45 |
| | 13.6.3. | Efficacy | 46 |
| | 13.6.4. | Safety | 48 |
| | 13.6.5. | Pharmacodynamic and Biomarker | .49 |
| 13.7. | Appendix | 7: Reporting Standards for Missing Data | .60 |
| | 13.7.1. | Premature Withdrawals | |
| | 13.7.2. | Handling of Missing Data | 60 |
| | | 13.7.2.1. Handling of Missing and Partial Dates | .61 |
| 13.8. | Appendix | 8: Values of Potential Clinical Importance | .62 |
| | 13.8.1. | Laboratory Values | .62 |
| | 13.8.2. | ECG | .63 |
| | | Vital Signs | |
| 13.9. | Appendix | 3: Abbreviations & Trade Marks | 64 |
| | 13.9.1. | Abbreviations | 64 |
| | 13.9.2. | Trademarks | .66 |
| 13.10. | | : 10: List of Data Displays | |
| | 13.10.1. | Data Display Numbering | .67 |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | 13.10.5. | Efficacy Figures | .88 |
| | | Safety Tables | |
| | | Pharmacokinetic Tables | |
| | | Pharmacokinetic Figures | |
| | | Pharmacodynamic and Biomarker Tables | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 13 11 | Appendix | : 11: Example Mock Shells for Data Displays | 108 |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| GlaxoSmithKline Document Number | Date | Version |
| 2014N218070_00 | 2015-JUN-04 | Original |
| 2014N218070_01 | 2015-NOV-30 | Amendment No. 1 |
| Pomovo the specific equations for the prediction of percent predicted from spirometry | | |

Remove the specific equations for the prediction of percent predicted from spirometry from the inclusion criteria and in Section 7.7.2. At screening it may not be possible to identify which correction method was used, or modify the correction method used, at the time. It therefore is not valid to stipulate that lung function values be corrected using any particular method. Both FEV<sub>1</sub> and FVC measurements (which are not entry criteria for the study) collected during the study will be collected as absolute values (uncorrected), so that consistency will be obtained across all sites in the study, and percent predicted will be calculated using a standard approach in house at the end of the study.

| 2014N218070_02 | 2016-JAN-26 | Amendment No. 2 |
|----------------|-------------|-----------------|
|----------------|-------------|-----------------|

Increase the body mass index (BMI) range in the inclusion criteria from 18-32 kg/m<sup>2</sup> (inclusive) to 16- 35 kg/m<sup>2</sup> (inclusive). The original BMI range from 18-32 kg/m<sup>2</sup> is a typical range used in both healthy volunteer studies and general subject populations. The revised range is more appropriate for a COPD patient population.

To remove photo toxicity from the protocol and to include minor administrative and clarification changes.

| 2014N218070_04 | 2017-MAR-2 | Amendment No. 4 |
|----------------|------------|-----------------|
|----------------|------------|-----------------|

Replace the administration of GSK2269557 via the DISKUS<sup>TM</sup> device (1000  $\mu$ g) by a comparable dose administered via the ELLIPTA<sup>TM</sup> device (700  $\mu$ g). GSK2269557 is no longer manufactured for use with the DISKUS device which will be replaced with ELLIPTA Device. To increase the number of patients to be recruited to obtain sufficient completers. Minor updates and clarifications.

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Total lung capacity and lung lobar<br>volumes included in HRCT<br>secondary endpoint parameters | Total lung capacity and lung lobar<br>volumes dropped from HRCT<br>secondary endpoint parameters<br>included as an exploratory<br>endpoint parameter instead | The clinically relevant HRCT parameters are still to be decided. However, there was no clinical benefit seen in the comparison between GSK2269557 1000 mcg and Placebo in these parameters. |
| Analysis population: All Subject All randomised subjects who receive at least one dose of the study treatment. This population will be based on the treatment the subject actually received. Pharmacokinetic Subjects in the 'All subject' population for whom a pharmacokinetic sample was obtained and analysed. | <ul> <li>Analysis population: <ul> <li>All Subject</li> <li>All randomised subjects who receive at least one dose of the study treatment.</li> <li>This population will be based on the treatment the subject actually received.</li> <li>Pharmacokinetic Subjects in the 'All subject' population for whom a pharmacokinetic sample was obtained and analysed.</li> </ul> </li> <li>Note: The two subjects who were not compliant with inhaler instructions will be excluded from the outcome summaries if they received active treatment but will be included if they received placebo</li> </ul> | 2 subjects were not compliant with inhaler instructions and may not have received the full dose in amendment 4. Therefore, these subjects will be excluded from the outcome summaries if they received active treatment but will be included if they received placebo. Sensitivity analyses may be conducted including these subjects. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | | Endpoints | |
|---|---|---|---|
| Pri | Primary Objectives | | nary Endpoints |
| • | To establish the PI3Kδ-dependent changes in previously identified immune cell mechanisms specifically related to neutrophil function using mRNA in sputum from patients with an exacerbation of COPD, with or without treatment with GSK2269557. | • | Alterations in previously identified immune cell mechanisms specifically related to neutrophil function as determined by changes in mRNA transcriptomics in induced sputum after 12, 28 and 84 days of treatment. |
| Sec | condary Objectives | Sec | ondary Endpoints |
| • | To evaluate the effect of once daily repeat inhaled doses of GSK2269557 on lung parameters derived from HRCT scans in subjects with acute exacerbation of COPD, compared to placebo. | • | Change from baseline in siVaw, iVaw, iRaw, siRaw, total lung capacity, lung lobar volumes, trachea length and diameter at FRC and TLC after 12 days of treatment and after 28 days of treatment. |
| • | To assess the safety and tolerability of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. | • | Adverse events Haematology, clinical chemistry Vital signs 12-lead ECG |
| • | To evaluate the plasma PK of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD. | • | Day 1 plasma Cmax and trough (24 hours) post dose for inpatients. Trough concentration after 12 days, 28 days, 56 days and 84 days of treatment. |
| • | To evaluate the effect of once daily repeat inhaled doses of GSK2269557 on lung function parameters in subjects with acute exacerbation of COPD compared to placebo. | • | To evaluate the effect of once daily repeat inhaled doses of GSK2269557 on lung function parameters in subjects with acute exacerbation of COPD compared to placebo. |
| Exp | oloratory Objectives | Exp | loratory Endpoints |
| • | To establish any other PI3Kδ-dependent changes in mRNA in sputum or blood from patients with an exacerbation of COPD, with or without treatment with GSK2269557. | • | To establish any other PI3Kδ-dependent changes in mRNA in sputum or blood from patients with an exacerbation of COPD, with or without treatment with GSK2269557. To explore the pharmacodynamic effects in induced sputum of once daily repeat inhaled doses of GSK2269557 qPCR. |
| • | To explore the pharmacodynamic effects in induced sputum of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. | | |
| • | To assess the changes in other CT parameters such as low attenuation score after once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. | • | Change from baseline for other CT parameters including low attenuation score after 12 days of treatment and after 28 days of treatment |

### 2.3. Study Design



# 2.4. Statistical Analyses

## 2.4.1. Primary Analyses

To estimate differences in mRNA intensities within and between treatment groups, a repeated measures model will be fitted to the results of the analysis of each probe set at Day 12, Day 28 and Day 84 following a loge transformation of the data. The Day 1 response will be fitted as a baseline covariate.

Back transformed ratios versus screening along with 95% confidence intervals will be calculated for each treatment group and timepoint. Additionally, baseline adjusted ratios of the change between active treatment and placebo will be calculated along with 95% confidence intervals.

Further details are provided in Section 7.1.

#### 3. PLANNED ANALYSES

# 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Participants<br>Enrolled (APE) | All subjects who were screened for eligibility | Study Population |
| All Subjects | Comprised of all subjects who were randomised. This population will be based on the treatment the subject actually received. If participants receive >1 treatment, then they will be summarised according to the most frequently dosed treatment. In cases where the frequency is equal, the participant will be assigned the lowest dose strength of nemiralisib. If participants receive no treatment, then they will be summarised according to "No Treatment" | <ul> <li>Study Population</li> <li>Pharmacodynamics<br/>and Biomarker</li> <li>Safety</li> <li>Efficacy</li> </ul> |
| Pharmacokinetic (PK) | Subjects in the 'All Subjects' population for whom a pharmacokinetic sample was obtained and analysed. | • PK |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

Note: The two subjects who were not compliant with inhaler instructions will be excluded from the outcome summaries if they received active treatment but will be included if they received placebo

#### 4.1. Protocol Deviations

During the course of the study it was noted that two subjects did not complete dosing instructions as required. The primary plan is if the subjects received active treatment they will be excluded from the study outcome summaries; if the subject received placebo treatment, they will be included in the study outcome summaries. It has not yet been identified if they received placebo or active treatment. A footnote will be applied to all relevant displays stating the rationale, subject number, treatment and if they were excluded, e.g. "Subjects X & Y did not complete dosing instructions as required; subject X received nemiralisib and was therefore excluded, subject Y received placebo and was therefore included." The footnote may be tweaked for aesthetic purposes.

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan, refer to Appendix 1.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order in TLF |
| This will be derived as subjects who did not receive any treatment | | No Treatment | 1 |
| This will b | ne derived as subjects in RandALL<br>or C | All Placebo | 2 |
| This will be derived as subjects in RandALL codes B or D | | All NEMI | 3 |
| Α | Placebo | Placebo Diskus | 4 |
| B GSK2269557 1000 mcg | | NEMI Diskus | 5 |
| С | Placebo via Ellipta | Placebo Ellipta | 6 |
| D | GSK2269557 700 mcg | NEMI Ellipta | 7 |

#### NOTES:

- 1. The following footnote will be presented on displays which use the "Placebo Diskus", "NEMI Diskus", "Placebo Ellipta" or "NEMI Ellipta" treatment groups:
  - NEMI Diskus =1000 mcg Nemiralisib administered via the Diskus device; NEMI Ellipta =700 mcg Nemiralisib administered via the Ellipta device
- 2. Order represents treatments being presented in TFL, as appropriate

Treatment groups "Placebo" and "Placebo via Ellipta" (RandAll NG codes A and C) will be combined into "All Placebo" treatment group. Similarly, treatment groups "GSK2269557 700 mcg" and "GSK2269557 1000 mcg" (RandAll NG codes B and D) will be combined into "All NEMI" treatment group.

Treatment comparisons will be displayed as follows using the descriptors as specified:

#### 1. All NEMI vs All Placebo

#### Notes:

- The "All Placebo" and "All NEMI" groups and "All NEMI vs All Placebo" treatment comparison will be presented for Pharmacodynamic and biomarker, efficacy and study population summaries unless otherwise specified.
- The "Placebo Diskus", "NEMI Diskus", "Placebo Ellipta" or "NEMI Ellipta" treatment groups will be presented for Pharmacokinetic and safety summaries unless otherwise specified.
- The "Placebo Diskus", "NEMI Diskus", "Placebo Ellipta" or "NEMI Ellipta" treatment groups will be presented for all listings

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | St | Baseline | | | |
|---|---|---|---|---|---|
| | Screening | Day 1<br>(Pre-<br>Treatment) | Day 2<br>Within<br>48H/discharge<br>(On Treatment) | Day 12<br>(On<br>Treatment) | Used in Data<br>Display |
| Safety | | | | | |
| Labs including<br>Haematology | X | Х | | | Day 1 |
| ECG | Х | Х | | | Day 1 |
| Vitals | Х | Х | | | Day 1 |
| Efficacy | | | | | |
| HRCT Untrimmed | Х | | | | Screening |
| HRCT Scan<br>Trimmed | | | | | |
| Screening&Day12 | X | | | | Screening |
| Screening&Day28 | X | | | | Screening |
| Day12&Day28 | | | | Х | Day 12 |
| FEV₁ and FVC | | Х | Х | | Day 1 <sup>[1]</sup> |
| Daily PEF [2] | | Χ | | | Day 1 |
| | | | | | Mean of Days<br>1 to 3 |
| | | | | | Maximum of Days 1 to 3 |
| Pharmacodynamic | , | | | | <u>'</u> |
| Sputum and Blood | X | | | | Screening |
| Genetic sample (PGx) [3] | | | Х | | |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- [1] Baseline will be investigated to ensure there is sufficient data and will be footnoted as appropriate
- [2] For PEF 3 different baselines will be calculated: Day 1, mean of Days 1 to 3 and Maximum of Days 1 to 3. TFLs will be footnoted with the relevant baseline.
- [3] Collected at any time after randomisation

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Examination of Covariates and Subgroups

#### 5.3.1. Covariates and Other Strata

The list of covariates may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates of clinical interest may also be considered.

| Category | Details |
|------------|-------------------------------------------------------|
| Covariates | Age, Sex, BMI, Country, Primary exacerbation severity |

## **5.3.2.** Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories |
|-------------------------------|------------------------|
| Primary exacerbation severity | Moderate or Severe [1] |
| Country | Country |

#### NOTES:

[1] Exacerbations are defined as severe if they require hospitalisation, otherwise they are defined as moderate

# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 13.3 | Appendix 3: Assessment Windows |
| 13.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 13.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 13.6 | Appendix 6: Derived and Transformed Data |
| 13.7 | Appendix 7: Reporting Standards for Missing Data |
| 13.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "All Subjects" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

#### 7. PHARMACODYNAMIC AND BIOMARKER ANALYSES

# 7.1. Primary Pharmacodynamic and Biomarker Analyses

## 7.1.1. Endpoint / Variables

Sputum RNA will be extracted and hybridised using a balanced batch design. An appropriate microarray platform will be determined at the time of hybridisation, to allow for improvements in technology. The quality of the data will be assessed and then normalised using appropriate methodologies and software.

Microarray mRNA data will be normalised using gcRMA or RMA in Array Studio v5.0 or later. After normalisation, the data will be quality assessed and any samples deemed as QC fails will be excluded from any further analysis. This quality assessment will involve looking for outlying signals in both the normalised expression data and the MAS5 QC metrics generated from each sample. If any samples are excluded, the remaining data will be re-normalised. The output from the normalisation will be log2 transformed mRNA intensity data (measured in arbitrary units).

Since the data will be  $\log 2$  transformed prior to the analysis the treatment effects will be expressed as ratios after back transformation (2<sup>\(\circ\)</sup>). These ratios can be converted to fold change values as follows:

- If ratio ≥ 1 then fold change = ratio
- If ratio <1 then fold change = -1/ratio

Microarray data consists of expression values (log2-transformed) derived from individual probe sets designed against coding regions of individual genes. More than one probe set can exist per gene. This analysis will be conducted at the probe set level.

The mRNA data gives results from  $\sim$ 14000 genes encoded by  $\sim$ 54000 probe sets. To establish the PI3K $\delta$ -dependent changes in previously identified immune cell mechanisms specifically related to neutrophil function using mRNA, we identified 258 gene to subset our data on, refer to Section 13.6.5. The gene names were converted to Affymetrix probe IDs, this resulted in 638 probes refer to Section 13.6.5.

To compare the expression value between treatments for each probe set, linear repeated measures mixed effects model will be fitted to each probe set, with log2 (intensity) as the response variable. Note: log2 (intensity) may also be referred to as mRNA intensities (logarithm base 2 scale). Alteration in previously identified immune cell mechanisms specifically related to neutrophil function will be determined by changes in mRNA transcriptomics in induced sputum after 12, 28 and 84 days of treatment by the analysis of mRNA intensities (logarithm base 2 scale) subset by the 638 probes identified in Section 13.6.5.

### 7.1.2. Summary Measure

A repeated measures modelling analysis will be performed on the subset of 638 probes which have previously identified immune cell mechanisms specifically related to neutrophil function.

The model will be used to estimate the baseline adjusted fold changes for active treatment and placebo calculated for Day 12, Day 28 and Day 84 along with the corresponding 95% confidence intervals and unadjusted P-values. Additionally, baseline adjusted ratios of the change between active treatment and placebo will be calculated along with 95% confidence intervals and unadjusted P-values.

## 7.1.3. Population of Interest

The primary pharmacodynamic analyses will be based on the "All Subjects" population, unless otherwise specified.

#### 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.1.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

 Alterations in the previously identified immune cell mechanisms specifically related to neutrophil function as determined by changes in mRNA transcriptomics in induced sputum after 12, 28 and 84 days of treatment. The response variable will be mRNA intensities (logarithm base 2 scale).

#### **Model Specification**

The mRNA data gives results from ~14000 genes encoded by ~54000 probe sets. A subset of 638 probe sets specifically relating to the cell mechanisms of neutrophil function is specified in Section 13.6.5 This subset will comprise the primary statistical analysis dataset.

Each probe set will be analysed separately.

The log2 transformed mRNA intensities will be analysed in a repeated measures model under a Frequentist framework. The model will include a Treatment, Visit and Treatment\*Visit term. The Visit will consist of 4 levels: Screening (Baseline), Day 12, Day 28 and Day 84, and the Treatment will consist of three levels: Null (when Visit = Screening), All Placebo and All NEMI. An unstructured (UN) covariance structure will be fitted. The denominator degrees of freedom for use in significance testing will be computed using the Kenward Rogers approximation.

Back transformed baseline-adjusted ratios along with 95% CIs and two-sided unadjusted p-values will be calculated for each Visit for the All NEMI and All Placebo Treatments, i.e. Day 84, Day 28 and Day 12 in the All NEMI Treatment group vs Screening and Day 84, Day 28 and Day 12 in the All Placebo Treatment group vs Screening. Additionally, baseline adjusted ratios between All NEMI vs All Placebo will be calculated for Day 12, Day 28 and Day 84 along with 95% CI and two-sided unadjusted p-values, i.e. Day 84 in the All NEMI Treatment group vs Day 84 in the All Placebo Treatment group, similarly for Day 28 and Day 12. Other comparisons of interest may also be calculated such as means for each Visit and Treatment, i.e. Screening (Null Treatment), Day 12, 28 and 84 (All NEMI Treatment) Day 12, 28 and 84 (All Placebo Treatment).

To enable review by the study team, csv files will be created containing the output for all probe sets in scope for the primary statistical analysis will be generated sorted alphabetically by probe set ID. Separate csv files may be created containing only probe sets where the p-value for the comparisons is <0.05. Such probe sets will be ranked by fold change, with the expectation that, in general, a greater than a 1.5-fold change is scientifically meaningful. To comply with guidance regarding QC, csv files will be stored as a SAS dataset to ensure QC can be audited.

Following review by the study team of the results, a subset of probe sets may be identified and may be used for further reporting.

#### **Model Checking & Diagnostics**

- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - In the event that this model fails to converge, alternative correlation structures may be considered

#### **Model Results Presentation**

Output from the repeated measures modelling detailed above will be tabulated. In particular, the estimated baseline adjusted fold changes, 95% CI, standard error (on the logarithm base 2 scale), unadjusted p-values at each time point and for the active treatment comparison with placebo. The probe set, gene/gene description will be included in the outputs.

# 7.2. Exploratory Pharmacodynamic and Biomarker Analyses

#### 7.2.1. Endpoint / Variables

In addition to the primary analysis, there is an exploratory objective to establish any other PI3K $\delta$ -dependent changes in mRNA in sputum or blood from patients with an exacerbation of COPD, with or without treatment with GSK2269557. To address this

blood and sputum mRNA data, as described in Section 7.1,but analyses will be conducted on the complete mRNA data, i.e. the results from  $\sim$ 14000 genes encoded by  $\sim$ 54000 probe sets.

To explore the pharmacodynamic effects in induced sputum of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. Endpoints may include, but not limited to, cytokines (IL-6, IL-8, TNFα), microbiome (by 16SrRNA), bacterial qPCR, total cell counts and PMNs differentials.

To explore the pharmacodynamic effects in blood of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. Endpoints may include, but not limited to, total cell counts and PMNs differentials.

# 7.2.2. Summary Measure

To establish any other PI3K $\delta$ -dependent changes in mRNA in sputum or blood from patients with an exacerbation of COPD, with or without treatment with GSK2269557. A repeated measures modelling analysis will be performed on the complete probe set. The model will be used to estimate the baseline adjusted fold changes for active treatment and placebo calculated for Day 12, Day 28 and Day 84 along with the corresponding 95% confidence intervals and unadjusted P-values. Additionally, baseline adjusted ratios of the change between active treatment and placebo will be calculated along with 95% confidence intervals and unadjusted P-values.

To explore the pharmacodynamic effects in induced sputum of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. Summary statistics of endpoints may include, but not limited to, cytokines (IL-6, IL-8, TNF $\alpha$ ), microbiome (by 16SrRNA), bacterial qPCR, total cell counts and PMNs differentials.

To explore the pharmacodynamic effects in blood of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. Summary statistics of endpoints may include, but not limited to, total cell counts and PMNs differentials.

#### 7.2.3. Population of Interest

The exploratory pharmacodynamic analyses will be based on the "All Subjects" population, unless otherwise specified.

As previously discussed for the two subjects that did not follow inhalation instructions, if the subjects received active treatment they will be excluded from the study outcome summaries; if the subject received placebo treatment, they will be included in the study outcome summaries.

#### 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Refer to Section 7.1.4.1 for statistical methodology specification, however, for the exploratory analysis, the models will be fitted but on the complete dataset ~14000 genes encoded by ~54000 probe sets; sputum and blood data will be analysed separately. Note: only a subset of the results will be presented as it is not feasible to present all ~54,000 probe sets for the sputum and blood data. Biostatistics will await guidance following unblinded regarding which, if any, probe sets should be presented for the exploratory analysis and confirmation if a cut off criteria other than p-value<0.05 AND (fold change> 1.5 OR fold change< -1.5) should be used in determining which comparisons for the probe sets should be presented.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed. For each endpoint, the values will be inspected to determine whether a data transformation is required. It is expected that: cytokines may require a transformed on the natural logarithm scale

#### 8. EFFICACY ANALYSES

# 8.1. Secondary Efficacy Analyses (Not From HRCT Analyses)

## 8.1.1. Endpoint / Variables

To evaluate the effect of once daily repeat inhaled doses of nemiralisib on lung function parameters in subjects with acute exacerbation of COPD compared to placebo. Lung function parameters including:

- PEF
- FEV<sub>1</sub> and FVC at clinic prior to sputum induction
- reliever usage

#### 8.1.2. Summary Measure

For PEF, summary statistics for the change from baseline PEF will be presented in tabular form, mean and 95% CIs of AM PEF readings will be plotted by study treatment vs. Study Day.

For  $FEV_1$  (L) and FVC (L), a change from baseline statistical analysis will be conducted and presented via tables of predicted adjusted medians for each Treatment arm at each visit, and the difference between treatment arms at each visit.

For reliever use, bronchodilator use recorded in the diary will be summarised as the mean number of occasions of rescue use per day and the percentage of rescue-free days in four-week interval periods as described in Section 13.6.3, where a rescue-free day is defined as a 24-hour period in which the number of occasions bronchodilator taken is zero. Summary tables will display estimates for each 4-weekly period for mean number of occasions of rescue use per day and percentage of rescue-free days separately.

#### 8.1.3. Population of Interest

The primary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

#### 8.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 8.1.4.1. Statistical Methodology Specification

NOTE: The description below describes the current thinking of how to analyse these endpoints. The proposed models will be assessed, and if not appropriate alternative models could be used.

## **Endpoint / Variables**

• FEV1 (L), FVC(L)

#### **Model Specification**

- The data will be inspected during statistical analysis to determine whether a data transformation is required. It is likely no transformations will be required
- The analysis will include all available values. If there are values which were recorded within 4h after the subject had taken relief medication, a sensitivity analysis may be done which excludes these values.
- The endpoints (FEV<sub>1</sub> and FVC) will be analysed in separate models. The change from baseline in the endpoint will be analysed in a Bayesian repeated measures model, with a baseline by Visit covariate and Treatment by Visit class parameter. Note that the model will not include an intercept. The Treatment will have two levels: All NEMI and All Placebo, and the Visit will have two levels: Day 28 and Day 84. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e. covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The change from baseline at each of the Visits will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in a tabular format.
- The difference between the treatment arms, for the change from baseline will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular format.
- The probabilities that the treatment difference is greater or less than 0 (depending on direction
  of the endpoint), in addition to other values appropriately selected based on the data, will also
  be computed for each Visit. These results will be presented in tabular format.

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data. For example, if data do not approximately follow a normal distribution then attempt will be made to find a suitable transformation.
- A comprehensive investigation into a suitable model should be initiated. For example, additional covariates will be investigated
- An unstructured covariance structure will be used. However, in the event that this model fails to converge, alternative correlation structures may be considered.
- Models with a Bayesian Framework will use vague priors. If appropriate, conjugate priors will be used. For example, for a multivariate model, the prior for the variance covariance matrix will be an inverse Wishart distribution.

#### **Model Results Presentation**

 Output from the repeated measures modelling detailed above will be tabulated. In particular, the estimated change from baseline, 95% CI, standard error, and posterior probabilities at each time point and for the active treatment comparison with placebo.

#### **Subgroup Analyses**

- For FEV1, a subgroup analysis will be conducted by index exacerbation severity (refer to Section 5.3 Examination of Covariates and Subgroups). A similar model as described in Model specification will be fitted but will also include a Severity\*Treatment\*Visit term within the model.
- The results of the subgroup analysis will be reported in a separate table.

# 8.2. Secondary Efficacy Analyses (From HRCT Analyses)

#### 8.2.1. Endpoint / Variables

To evaluate the effect of once daily repeat inhaled doses of nemiralisib on lung parameters derived from HRCT scans in subjects with acute exacerbation of COPD, compared to placebo. Ratio from baseline in siVaw, iVaw, iRaw, siRaw, trachea length and diameter at FRC and TLC after 12 days of treatment and after 28 days of treatment.

#### 8.2.2. Summary Measure

Each HRCT scan will be conducted at two lung volumes: total lung capacity (TLC) and functional residual capacity (FRC); these will be referred to as scan conditions. The HRCT images will be processed to derive the HRCT parameters at FRC and TLC, however these conditions are not applicable for all parameters.

The HRCT scans will be conducted at Screening, Day 12 and Day 28. The 3 HRCT images will then be processed to derive the HRCT parameters at each scan; this data will be referred to as the untrimmed data. The untrimmed data measures all airways that are present in each scan.

However partially due to positioning of subjects whilst taking a scan, it can be that some airways are visible in some scans and not in other scans. For these reasons, some HRCT

imaging endpoints will be calculated to include only airways that are visible in both scans. Therefore, the scans were grouped into three scan trimming pairs where, within each scan trimming pair, the airways that were not present in both scans were removed/trimmed.

The three scan trimming pairs, and subsequent timepoints, are:

- The scan trimming pair SCRD28, which contains the Screening (SCRD28:SCR) and Day 28 (SCRD28:D28) timepoints, where only airways that were present in both screening and day 28 scans are accounted for.
- The scan trimming pair SCRD12, which contains the Screening (SCRD12:SCR) and Day 12 (SCRD12:D12) timepoints where only airways that were present in both screening and day 12 scan are accounted for.
- The scan trimming pair (D12D28), which contains the Day 12 (D12D28:D12) and Day 28 (D12D28:D28) timepoints, where only airways that were present in both day 12 and day 28 scans are accounted for.

These 6 HRCT images were then processed to derive the HRCT parameters at each of these scan-trimming pair time points; this data will be referred to as the scan trimmed data. The scan trimmed data considers only airways that were present in both scans within the scan trimming pair. This ensures the airway models are the same length although the cross-sectional area of the airway may vary. For example, the schematic below shows visible airways on Screening alone and Day 12 alone. It then shows the airways that are visible on both Screening & Day 12 scans, through removing/trimming airways that are not present in both scans.



The HRCT scans can identify the 5 different lobes of the lungs and these lobes can then be categorized into and up to 5 regions depending on the endpoint. The 5 lobes are Right Upper Lobe (RUL), Left Upper Lobe (LUL), Right Middle Lobe (RML), Right Lower Lobe (RLL) and Left Lower Lobe (LLL). The 5 regions are Upper (comprising of RUL, RML and LUL), Lower (comprising of RLL and LLL), Central (the main bronchi between the lobes and the trachea), Distal (comprising of Upper and Lower) and Total (comprising of Distal and Central).

The endpoints for which the 5 regions apply include:

- Specific imaging airway volume (siVaw)
- Imaging airway volume (iVaw)
- Specific imaging airway resistance (siRaw)
- Imaging airway resistance (iRaw)
- Specific imaging airway wall volume (siVaww)
- Imaging airway wall volume (iVaww)

The endpoints for which only 3 regions (upper, lower & total) apply include:

- Imaging lobe volume (iVlobe)
- Percent predicted lobar volume (iVlobepred)
- Low attenuation score (LAS)
- Air trapping score (AT)
- Blood vessel density (BVD)

The endpoint for which only 2 regions (upper & lower) apply is:

• Internal airflow lobar distribution (IALD)

For the measures iVaw, iRaw and iVaww, standardization within a subject for the size of the lobar volume was conducted. These specific measures can be adjusted for the individual's lobar volume by correcting for the corresponding lobe/region. Note the central region is not applicable for lobar volumes, instead the corresponding region for the central, distal and total regions is the total lobar volume region. For example:

- To calculate siVaw, the lobes/regions of iVaw being divided by the corresponding lobes/regions of iVlobe to calculate the lobes/regions of siVaw, thus siVaw can be defined as a measure of volume in an individual's airways, corrected for the individual's lobar volume.
- To calculate siRaw, the lobes/regions of iRaw were multiplied by the corresponding lobes/regions of iVlobe.
- To calculate siVaww, the lobes/regions of iVaww were divided by the corresponding lobes/regions of iVlobe.

For such reasons, the table below shows the HRCT endpoints and the results that will be captured:

Table 2 HRCT Endpoints (and results that will be captured)

| | | Untrimmed | | Scan Trimming, based on: | | | |
|---|---|---|---|---|---|---|---|
| Endpoints | Units | Screening | Day<br>12 | Day 28 | Screening<br>and Day 12<br>scans | Screening<br>and Day 28<br>scans | Day 12 and<br>Day 28 scans |
| iVaw | mL | Х | Х | Х | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| siVaw | mL/L | х | Х | Х | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| iRaw | KPa*s/L | | | | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| siRaw | KPa*s | | | | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| iVlobe | L | Х | х | Х | | | |
| Percent<br>Predicted iVlobe | % of<br>Predicted<br>value | х | х | Х | | | |
| IALD [3] | % | Х | х | Х | | | |
| LAS [1] | % of iVlobe | х | Х | Х | | | |
| AT [2] | % of iVlobe | х | Х | Х | | | |
| BVD [1] | % of iVlobe | х | Х | Х | | | |
| iVaww <sup>[1]</sup> | mL | Х | Х | Х | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| siVaww <sup>[1]</sup> | mL/L | х | Х | Х | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| Trachea length | mm | Х | х | Х | | | |
| Trachea<br>Diameter | mm | х | Х | х | | | |
| Trachea<br>Length/Diameter | mm/mm | Х | Х | Х | | | |

All these endpoints will be measured at TLC and FRC, except:

- [1] These endpoints will only be measured at TLC
- [2] This endpoint will be measured only at FRC [3] The state (TLC/FRC) is not applicable

For the endpoints siVaw, iVaw, iRaw and siRaw appropriate transformations will be applied prior to summaries and statistical analyses, likely a log transformation. Summary statistics will be presented for absolute data and change from baseline. An attempt will be made to fit separate statistical models for each endpoint, scan trimming condition (Untrimmed or Scan Trimmed), lung volume (FRC or TLC) and Lobes (RUL, LUL, RML, RLL and LLL) or Regions (Upper, Lower, Central, Distal and Total) combination as appropriate. The primary plan for statistical analyses will be to fit separate statistical models for:

#### • siVaw

- o Untrimmed at FRC for all lobes, i.e. RUL, LUL, RML, RLL and LLL in one model.
- Untrimmed at FRC for all regions, i.e. Upper, Lower, Central, Distal and Total in one model.
- o Scan Trimmed at FRC for Distal region only.

#### siRaw

o Scan Trimmed at FRC for Distal region only.

For untrimmed data, the ratio from baseline across the different Regions (accounting for the average baseline associated to the Region of interest) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). In addition, the placebo-adjusted ratio from baseline across the different Regions will be represented via adjusted posterior medians, as well as their associated 95% HPD-tailed credible intervals and posterior probabilities. These results will be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

For scan trimmed data, the change from baseline across the different Regions (accounting for the average baseline associated to the Region of interest) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). In addition, the placebo-adjusted change from baseline across the different Regions will be represented via adjusted posterior medians, as well as their associated 95% HPD-tailed credible intervals and posterior probabilities. These results will be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

For the tracheal endpoints, absolute data and change from baseline summary statistics will be provided for each lung volume (FRC or TLC) for trachea length, diameter and length/diameter.

#### 8.2.3. Population of Interest

The primary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

#### 8.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8.2.4.1. Statistical Methodology Specification

NOTE: The description below describes the current thinking of how to analyse these endpoints. The proposed models will be assessed, and if not appropriate alternative models could be used.

#### **Endpoint / Variables**

Imaging Untrimmed endpoint siVaw at FRC

#### **Model Specification**

- The data will be inspected prior to analysis to determine whether a data transformation is required. It is likely that the data will approximately follow a log normal distribution; however, the most appropriate distribution should be used.
- It is thought that the use of bronchodilators could affect the HRCT results. The database will contain information on whether relief medication was used in the 4 hours prior to each scan, and this information may be used in the sensitivity analyses of the HRCT results.
- An attempt will be made to fit a statistical model for all Lobes (RUL, LUL, RML, RLL and LLL) and a separate statistical model for all Regions (Upper, Lower, Central, Distal and Total), i.e. two models; one for lobes, one for regions. However, should this model fail to converge or be deemed unsuitable potentially due to sample size, separate statistical models will be fitted for each Lobe/Region (RUL, LUL, RML, RLL, LLL, Upper, Lower, Central, Distal and Total), i.e. ten models in total, one for each lobe/region endpoint.
- The log of (or other transformation as appropriate) the ratio from baseline will be analysed in a multivariate model), under a Bayesian framework. The model will include a Baseline\*Region term and a Treatment\*Visit\*Region term, as well as any co-variates of interest. Note that the model will not include an intercept. The Visit will consist of two levels: Day 12 and Day 28, and the Treatment will consist of two levels: All NEMI and All Placebo. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e. covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The change from baseline (accounting for the average baseline) across the different Visits will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable).
- The difference between the treatment arms, for the change from baseline across the different

- Visits will be represented via adjusted medians, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable)
- The probabilities that the treatment ratio is greater than 1 (depending on direction of the endpoint), in addition to other values appropriately selected based on the data, will also be computed for each Visit. These results will be presented in tabular format

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data. For example, if data do not approximately follow a normal distribution then attempt will be made to find a suitable transformation.
  - Note: Should parameters require a log transformation with an offset, for each posterior sample (i) appropriately back transformed values will be calculated for each treatment arm, and then (ii) using these back transformed values, the ratio of the treatment arms (All NEMI/All Placebo) will be calculated for each posterior sample, and finally summarised accordingly
- A comprehensive investigation into a suitable model should be initiated. For example, additional covariates will be investigated such as age, BMI, gender etc. Note: when investigating fitting separate statistical models for Lobes (RUL, LUL, RML, RLL and LLL) and Regions (Upper, Lower, Central, Distal and Total), i.e. two models; one for lobes, one for regions. If there are convergence issues an alternative structure of fitting separate statistical models for each Lobe (RUL, LUL, RML, RLL and LLL) and each Region (Upper, Lower, Central, Distal and Total), i.e. ten models; five for lobes, five for regions. a similar model as described in Model Specification should be tested but will include a baseline and a Treatment\*Visit term instead of a Baseline\*Region term and a Treatment\*Visit\*Region term, respectively.

Note: It may also be prudent to investigate a model fitting baseline as a timepoint in which case the log of (or other transformation as appropriate) the absolute results will be analysed in a multivariate model, under a Bayesian framework. The model could include a Treatment\*Visit\*Region parameter, as well as any co-variates of interest. Note that this model would not include an intercept. The Visit would consist of three levels: Baseline, Day 12 and Day 28, and the Treatment would consist of three levels: Null (when Visit = Screening), NEMI and Placebo. With assumptions as described in Model Specification.

- An unstructured covariance structure will be used. However, in the event that this model fails to converge, alternative correlation structures may be considered.
- Models with a Bayesian Framework will use vague priors. If appropriate, conjugate priors will be used. For example, for a multivariate model, the prior for the variance covariance matrix will be an inverse Wishart distribution.

#### **Model Results Presentation**

 Output from the repeated measures modelling detailed above will be tabulated. In particular, the estimated ratio to baseline (or change from baseline if appropriate), 95% CI, standard error (on the appropriate scale, likely logarithm base e), and posterior probabilities at each time point and for the active treatment comparison with placebo. The scan trimming condition, lung volume and lobe or region description will be included in the outputs.

## **Sensitivity and Supportive Analyses**

• It is thought that the use of bronchodilators could affect the HRCT results. The database will contain information on if relief medication was used in the 4 hours prior to each scan, and this

information may be used in the sensitivity analyses of the HRCT results including only those who did not take bronchodilator relief medication in the 4 hours prior to HRCT scan.

#### **Endpoint / Variables**

• Imaging Scan Trimmed endpoints siVaw and siRaw at FRC in the Distal Region only.

#### **Model Specification**

- It is likely that the data will approximately follow a log normal distribution; however, the most appropriate distribution should be used.
- Separate statistical models will be fitted for each endpoint, i.e. two models; one for siVaw (scan trimmed at FRC in Distal region), one for siRaw (scan trimmed at FRC in Distal region).
- The responses of interest are the change from baseline based on (i) Airways present on scans taken at Screening and Day 12, (ii) Airways present on scans taken at Screening and Day 28, and (iii) Airways present on scans taken at Day 12 and Day 28. The baselines for each of these endpoints are provided in the table below.

| | ` , | (ii) Screening & Day28<br>Scan trimming | (iii) Day 12 & Day 28<br>Scan trimming |
|---|---|---|---|
| Screening Result | ✓ (baseline) | ✓ (baseline) | |
| Day 12 Result | ✓ (post dose) | | ✓ (baseline) |
| Day 28 Result | | ✓ (post dose) | ✓ (post dose) |

- The modelling below assumes that the Scan trimming endpoints (Screening&Day12, Screening&Day28 and Day12&Day28) will be analysed in a single multivariate model. This is subject to sensitivity analysis.
- The log of (or other transformation as appropriate) the change from baseline (where baseline is defined in the table above) will be analysed in a multivariate model to account for the correlation between the multiple Scan Trimmings (Screening&Day12, Screening&Day28 and Day12&Day28), under a Bayesian framework. The model will have a separate intercept for each Scan Trimming combination (by fitting a class parameter Scan Trimming, and having no overall intercept), and will also include a baseline\*Scan Trimming and a Treatment\*Scan Trimming parameter. The Visit will consist of two levels: Day 12 and Day 28, the scan trimming will consist of three levels Screening&Day12, Screening&Day28 and Day12&Day28, and the Treatment will consist of two levels: All NEMI and All Placebo. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e. covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The change from baseline across the different Scan Trimming pairs (accounting for the average baseline) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be

- presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable).
- The difference between the treatment arms, for the change from baseline across the different Scan Trimming pairs will be represented via adjusted medians, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (if applicable). For parameters that require a log transformation with an offset, for each posterior sample (i) appropriately back transformed values will be calculated for each treatment arm, and then (ii) using these back transformed values, the ratio of the treatment arms (Active/Placebo) will be calculated for each posterior sample, and finally summarised accordingly.

The probabilities that the treatment ratio is greater than 1 (for siVaw) and less than 1 (for siRaw), in addition to other values appropriately selected based on the data, will also be computed for each Visit. These results will be presented in tabular format.

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data. For example if data do not approximately follow a normal distribution then an attempt will be made to find a suitable transformation.
  - Note: Should parameters require a log transformation with an offset, for each posterior sample (i) appropriately back transformed values will be calculated for each treatment arm, and then (ii) using these back transformed values, the ratio of the treatment arms (All NEMI/All Placebo) will be calculated for each posterior sample, and finally summarised accordingly
- A comprehensive investigation into a suitable model should be initiated. For example, additional covariates will be investigated
- An unstructured covariance structure will be used. However, in the event that this model fails to converge, alternative correlation structures may be considered.
- Models with a Bayesian Framework will use vague priors. If appropriate, conjugate priors will be used. For example, for a multivariate model, the prior for the variance covariance matrix will be an inverse Wishart distribution.

#### **Model Results Presentation**

 Output from the repeated measures modelling detailed above will be tabulated. In particular, the estimated ratio to baseline (or change from baseline if appropriate), 95% CI, standard error (on the appropriate scale, likely logarithm base e), and posterior probabilities at each time point and for the active treatment comparison with placebo. The scan trimming condition, lung volume and lobe or region description will be included in the outputs.

### Sensitivity and Supportive Analyses

• It is thought that the use of bronchodilators could affect the HRCT results. The database will contain information on if relief medication was used in the 4 hours prior to each scan, and this information may be used in the sensitivity analyses of the HRCT results including only those who did not take bronchodilator relief medication in the 4 hours prior to HRCT scan.

## 8.3. Exploratory Efficacy Analyses (From HRCT Analyses)

#### 8.3.1. Endpoint / Variables

To assess the changes in other HRCT parameters such as low attenuation score after once daily repeat inhaled doses of nemiralisib administered to subjects with acute exacerbation of COPD, compared to placebo. Change from baseline for other CT parameters including low attenuation score after 12 days of treatment and after 28 days of treatment.

### 8.3.2. Summary Measure

The structure of HRCT endpoints is as described in Section 8.2.2, exploratory endpoints include:

- iVlobe
- Percent Predicted iVlobe
- IALD
- LAS
- AT
- BVD
- iVaww
- siVaww

For all endpoints, the data will be inspected prior to analyses to determine whether a data transformation is required. Appropriate transformations will be applied prior to summaries and statistical analyses. It is likely a log transformation will be required for iVlobe, LAS, IALD, BVD iVaww and siVaww, and that no transformation will be required for Percent Predicted iVlobe and AT, however, the most appropriate distribution should be used

Summary statistics will be presented for absolute data and change from baseline. Separate statistical models will be fitted for each scan trimming condition (Untrimmed or Scan Trimmed), lung volume (FRC or TLC) and Regions (Upper, Lower, Central, Distal and Total) combination as appropriate, note: statistical analyses will only be conducted on:

- IALD for upper and lower regions only (within the same model)
- LAS at TLC for total region only
- AT at FRC for total region only
- BVD at TLC for total region only
- siVaww untrimmed data at TLC for distal region only

For the endpoints: LAS, AT and BVD, separate statistical models will be fitted for the Total region only. The change from baseline (accounting for the average baseline associated to the region) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). The difference between the treatment arms, for the change from baseline will be represented via adjusted medians, as

well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

For the endpoint IALD, a statistical model will be fitted for both the Upper and Lower regions. The change from baseline across the different regions (accounting for the average baseline associated to the region of interest) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). The difference between the treatment arms, for the change from baseline across the different regions will be represented via adjusted medians, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

For the endpoint siVaww, a statistical model will be fitted for the distal region using untrimmed data. The change from baseline (accounting for the average baseline associated to the region) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). The difference between the treatment arms, for the change from baseline will be represented via adjusted medians, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

#### 8.3.3. Population of Interest

The secondary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

#### 8.3.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.3.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8.3.4.1. Statistical Methodology Specification

For statistical analyses of IALD in the upper and lower regions refer to Section 8.2.4.1 for the analysis of untrimmed siVaw but note that it is likely only 1 statistical model would be fitted for the upper and lower regions only. If appropriate this could be adapted into two models; one for upper, one for lower. The probability that the treatment ratio is greater than 1 will be presented for the lower region and the probability that the treatment ratio is less than 1 will be presented for the upper region, in addition to other values appropriately selected based on the data.

For statistical analyses of LAS at TLC in the total region only, refer to Section 8.2.4.1 for the analysis of untrimmed siVaw but note only 1 statistical model would be fitted for the Total regions only. The probability that the treatment ratio is less than 1 will be presented, in addition to other values appropriately selected based on the data.

For statistical analyses of AT at FRC in the total region only, refer to Section 8.2.4.1 for the analysis of untrimmed siVaw however it is likely that no transformation will be required for this endpoint in which case the absolute change from baseline will be fitted and probabilities that the true treatment difference is less than 1, in addition to other values appropriately selected based on the data, will also be computed for each Visit. Note only 1 statistical model would be fitted for the Total regions only.

For statistical analyses of BVD at TLC in the total region only, refer to Section 8.2.4.1 for the analysis of untrimmed siVaw but note only 1 statistical model would be fitted for the Total regions only.

For statistical analyses of siVaww at TLC in the distal region only, refer to Section 8.2.4.1 for the analysis of untrimmed siVaw but note only 1 statistical model would be fitted for the Distal regions only. The probability that the treatment ratio is less than 1, in addition to other values appropriately selected based on the data will be presented.

### 8.4. Exploratory Efficacy Analyses (Not from HRCT Analyses)

#### 8.4.1. Endpoint / Variables

Additional exploratory endpoints include the severity of index exacerbation, where exacerbations requiring hospitalisations are defined as severe and those not requiring hospitalisation are defined as moderate.

## 8.4.2. Summary Measure

For the severity of index exacerbation, a summary table detailing the number and percentage of subjects who had moderate or severe index exacerbations. Note: exacerbations requiring hospitalisations are defined as severe and those not requiring hospitalisation are defined as moderate.

If available, data on exacerbations occurring during the study will be summarised. This may include investigator defined exacerbations (including information on moderate or severe) and/or concomitant medication defined exacerbations. Concomitant medication defined exacerbations may be defined as treatment with systemic/oral corticosteroids and/or antibiotics where the exacerbation is deemed to have ended if no additional treatment with systemic/oral corticosteroids and/or antibiotics is required within < 7days from the end of treatment for the primary exacerbation.

#### 8.4.3. Population of Interest

The secondary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

#### 8.4.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.4.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 9. RELATIONSHIP BETWEEN THE PHARMACODYNAMIC AND BIOMARKER DATA AND THE HRCT DATA

# 9.1. Relationship between the mRNA data and the HRCT data

The relationship between a selection of the mRNA data and the HRCT data may be performed as an exploratory analysis. This may include scatter plots of individual participant data, linear regression lines, Pearson's correlation coefficient and 95% confidence intervals plots as appropriate. This data will be produced following SAC.

#### 10. SAFETY ANALYSES

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

## 10.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

# 10.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

# 10.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

## 11. PHARMACOKINETIC ANALYSES

## 11.1. Secondary Pharmacokinetic Analyses

#### 11.1.1. Endpoint / Variables

## 11.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3 Reporting Standards for Pharmacokinetic)

#### 11.1.1.2. Derived Pharmacokinetic Parameters

No non-compartmental analysis will be conducted for this study as such there will be no derived pharmacokinetic parameters.

## 11.1.2. Summary Measure

The concentrations of the samples will be summarised.

#### 11.1.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

# 12. REFERENCES

Quanjer Ph.H, Tammeling G.J, Cotes J.E., Pedersen O.F, Peslin R, Yernault J-C. Lung volumes and forced ventilatory flows; *European Respiratory Journal* 1993 6: 5-40

# 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management

# 13.1.1. Important Protocol Deviations

Based on an assessment of the important protocol deviations listed in the PDMP, partial data exclusions or time-point exclusions may occur which may not remove a subject from the analysis population, but may exclude a portion of the subject's data.
## 13.2. Appendix 2: Schedule of Activities

## 13.2.1. Protocol Defined Schedule of Events

## **Screening and Follow Up Visits**

| Procedure | Screening (up to 3 days prior to Visit 1) | Follow-up (7-14 days post-last dose) | Notes |
|---|---|---|---|
| Informed consent | X | | |
| Demography | X | | |
| Inclusion and exclusion criteria | X | | |
| Full physical exam, including height and weight | X | | |
| Brief physical examination, including weight | | X | |
| Chest X-Ray | X | | To be done before baseline HRCT to exclude significant pneumonia and other incidental serious underlying pathology. |
| Medical history (includes substance usage and Family history of premature CV disease) | Х | | Substances: Drugs, Alcohol, tobacco via history. No drug, alcohol screening is required. |
| Past and current medical conditions (including cardiovascular medical history and therapy history) | X | | |
| Laboratory assessments (include Hematology and biochemistry) <sup>1</sup> | X | X | Historical values analysed by local lab to be used for eligibility assessment. Another sample must be collected and sent to central lab as soon as informed consent is obtained. |
| Hep B and Hep C screen <sup>2</sup> | X | | |
| Urine pregnancy test (only WCBP) | X | | Before conducting the HRCT. Done locally at the site. |
| 12-lead ECG | X | X | Single assessment |
| Vital signs | X | X | Single assessment |
| HRCT (at TLC and FRC) | X | | Within 48 h of diagnosis, if subject otherwise eligible. Includes electronic monitoring of breathing (if applicable). Baseline HRCT will be reviewed by the local site's radiologist to identify any significant occurring underlying medical conditions that require further clinical management or monitoring. |

| Procedure | Screening (up to 3 days prior to Visit 1) | Follow-up<br>(7-14 days post-last dose) | Notes |
|---|---|---|---|
| Induced Sputum <sup>3</sup> | X <sup>4</sup> | | To include sputum culture pre-first dose. Culture to be done by the local site laboratory. |
| Blood sample for mRNA Analysis | X <sup>4</sup> | | Collected at any time on specified days |
| AE/SAE collection and review | | X | |
| Concomitant medication review | Х | Х | |

- 1. Due to the short screening window, central laboratory analysis results will not be available on time. Therefore, the local laboratory results should be used for eligibility assessment (to exclude severe subjects and underlying medical conditions). If local laboratory results are already available from diagnosis of current exacerbation, there is no need to take another sample for local analysis. A sample for central laboratory analysis should also be obtained. See Section 7.8.6 of Protocol Amendment 4 for further details.
- 2. If test otherwise performed within 3 months prior to first dose of study treatment, testing at screening is not required. Because of the short window for screening, treatment with GSK2269557 may start before receiving the result of the hepatitis tests. If subsequently the test is found to be positive, the subject may be withdrawn, as judged by the Principal Investigator in consultation with the Medical Monitor.
- 3. Induced sputum collection may be attempted on several occasions if an adequate sample is not produced at the first attempt.
- 4. To be collected at any time point before randomisation.

## **Treatment Period**

| Procedure | Treatment Period | | | | Notes | | |
|---|---|---|---|---|---|---|---|
| Visit | 1 | 21 | 3 | 4 | 5 | 6 | |
| Day | 1 | Within 48h<br>/ discharge | 12 | 28 | 56 | 84 | |
| Visit window | N/A | ±1 days | ±2 days | ±2 days | - 4 / +2 days | - 4 / +2 days | |
| SAFETY ASSESSMENTS | | | | | | | |
| AE/SAE collection and review | ←==== | | ======= | ======= | ======== | ====→ | |
| Concomitant medication review | ←==== | ======== | ======= | ======= | ======== | ====→ | |
| Reliever usage | ←==== | ======== | | | | | |
| Brief physical exam, including weight | X <sup>2</sup> | | Χ | Χ | X | Χ | Pre-dose |
| Laboratory assessments (include haematology and biochemistry) | X <sup>2</sup> | | Χ | Х | Х | Χ | Pre-dose |
| 12-lead ECG | <b>X</b> <sup>2</sup> | | Χ | Χ | X | Χ | Pre-dose. Single assessment |
| Vital signs | X <sup>2</sup> | | Χ | Х | Х | Χ | Pre-dose. Single assessment |
| Urine pregnancy test (only WCBP) | | | Χ | Х | | | Before conducting the HRCT |
| STUDY TREATMENT | | | | | | | |
| ELLIPTA™ Inhaler Training | X | | | | | | Training conducted by reviewing the Patient Information Leaflet with the subject (no device will be used). Additional training may be conducted at the discretion of the investigator |
| Randomisation | X | | | | | | |
| Study drug administration | <b>←===</b> = | | | | | · | Daily in the morning before breakfast, (with the exception of days when the subjects have a planned visit to the clinic. On those days, they will be dosed at the clinic). |
| Assessment of study treatment compliance | | | Х | Х | Х | Х | |
| Diary Card dispense and review at clinic | Χ | | Χ | Χ | Х | Χ | Refer to SRM for details. |

| Procedure | | Treatment Period | | | | | | Notes |
|---|---|---|---|---|---|---|---|---|
| | Visit | 1 | 21 | 3 | 4 | 5 | 6 | |
| | Day | 1 | Within 48h<br>/ discharge | 12 | 28 | 56 | 84 | |
| , | Visit window | N/A | ±1 days | ±2 days | ±2 days | - 4 / +2 days | - 4 / +2 days | |
| EFFICACY ASSESSMENTS | | | | | | | | |
| HRCT (at TLC and FRC) | | | | X | X | | | At any time on specified days. Includes electronic monitoring of breathing (if applicable). The radiologist may review any of the scan(s) if they wish, but this is NOT required for the study. A formal review is required at screening only by the radiologist. |
| FEV₁ and FVC | | X | Х | Х | Χ | Х | Χ | In clinic only for all visits where possible. |
| PEF | | <b>←===</b> | ======== | ======= | ======= | | ==== <del>)</del> | Daily before drug administration at home. If subject in hospital, this may be collected using the handheld device provided prior to drug administration. |

| OTHER ASSESSMENTS | | | | | | | |
|---|---|---|---|---|---|---|---|
| Blood sample for PK | X | | Х | X | X | X | Day 1: 5 min and 24 h post-dose. The 24 h post-dose time-point is optional for subjects not hospitalised. Pre-dose at all other time-points. |
| Sputum induction <sup>3</sup> | | | Χ | Х | | Χ | |
| Blood sample for mRNA analysis | | | Х | Х | | Χ | |
| Genetic sample (PGx) <sup>4</sup> | | X | | | | | Collected at any time after randomisation |

- 1. On discharge if the subject was hospitalized. Within 48 hours of first dose administration if the subject was not hospitalised. See Section 4.2 of Protocol Amendment 4
- Assessments do not need to be completed if screening assessments conducted within 48 hours
   Induced sputum collection may be repeated on several occasions if an adequate sample is not produced at the first attempt
- 4. Informed consent for optional sub-studies (e.g. genetics research) must be obtained before collecting a sample. May be obtained at any visits.

## 13.3. Appendix 3: Assessment Windows

## 13.3.1. Definitions of Assessment Windows for Analyses

| Population | Target | Analysis V | /indow | Analysis |
|---|---|---|---|---|
| | | Beginning Timepoint | Ending Timepoint | Timepoint |
| Screening | NA | 3 days prior to Visit 1 (Day 1) | Day 1 | Screening |
| Safety, | NA – Day of first dose | NA | NA | Visit 1 |
| Efficacy, Study<br>population and<br>all other<br>assessments | If subject was hospitalised: Target = On discharge If subject wasn't hospitalised: Target = Within 48 hours of first dose administration | Target -1 day | Target +1 day | Visit 2 |
| | Day 12 | Target -2 day | Target +3 day | Visit 3 |
| | Day 28 | Target -4 day | Target +2 day | Visit 4 |
| | Day 56 | Target -7 day | Target +6 day | Visit 5 |
| | Day 84 | Target -8 day | Target +4 day | Visit 6 |
| Follow-up | NA | 1 week following last day of dose | 4 weeks following the last day of dose | Follow-up |

# 13.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

### 13.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the study treatment, unless otherwise specified

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

### 13.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

### 13.4.2. Treatment States for Adverse Events

| Flag | Definition |
|---|---|
| Pre-Treatment | If AE onset date is before the treatment start date. |
| | AE Start Date < Study Treatment Start Date |
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date. |
| (On-Treatment) | • Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date. |
| Post-Treatment | If AE onset date is after the treatment stop date. |
| | AE Start Date > Study Treatment Stop Date |
| Onset Time Since<br>1st Dose (Days) | If Treatment Start Date > AE Onset Date, then Onset Time = AE Onset Date - Treatment Start Date |
| | <ul> <li>If Treatment Start Date ≤ AE Onset Date, then Onset Time = AE Onset Date - Treatment Start Date +1</li> <li>Missing otherwise.</li> </ul> |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing]. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 13.5. Appendix 5: Data Display Standards & Handling Conventions

### 13.5.1. Reporting Process

| Software | |
|---|---|
| The currently sup | The currently supported versions of SAS software (version 9.4) will be used. |
| Reporting Area | |
| HARP Server | : UK1SALX00175.corpnet2.com |
| HARP Compound | : ARPROD/GSK2269557/mid201928 |
| | Note: the current planned reporting effort is final_01, this may be superseded. |
| <b>Analysis Datasets</b> | |
| <ul> <li>Analysis datasets will be created according to Legacy GSK A&amp;R dataset standards and Integrated Data<br/>Standards Library</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be g | generated for all tables |

## 13.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- A project wide decision was made to present GSK2269557 as Nemiralisib (abbreviated to NEMI) refer to Section 5.1 for further details.

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| | <ul> <li>Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be<br/>included in listings but omitted from figures, summaries and statistical analyses.</li> </ul> |
|---|---|
| Unscheduled Visits | |
| <ul> <li>Unscheduled visits</li> </ul> | s will not be included in summary tables. |
| <ul> <li>Unscheduled visits</li> </ul> | s will not be included in summary figures |
| All unscheduled vi | sits will be included in listings. |
| <b>Descriptive Summary</b> | Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |
| All graphics will be | done using the SGPLOT/SGPANEL/SG template procedures |

## 13.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. Note: Use the separate NEMI DISKUS and NEMI ELLIPTA treatment groups |
| NONMEM/Pop PK<br>File | Not applicable. |
| NONMEM/PK/PD<br>File | Not applicable. |

## 13.6. Appendix 6: Derived and Transformed Data

#### 13.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 13.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 13.6.2. Study Population

### **Treatment Compliance**

- Treatment compliance will be calculated based on the formula:
  - Treatment Compliance = Counter Readings / (Actual Treatment Duration in Days \* Frequency)
- Treatment compliance could be greater than 100% if there are events of overdose.

### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

Cumulative Dose = Sum of (Counter Readings x Study Drug Dose)

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age at Screening where birth date will be imputed as follows:
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Refer to IDSL standards for age range categories.

#### Body Mass Index (BMI)

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

### 13.6.3. **Efficacy**

### **HRCT**

### Endpoints provided by FluidDA

Y = Endpoints will be provided by FluidDA.

| | | | | | | | Lobes | & Regions | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | LLL | LUL | RML | RUL | RLL | 니 | UL | CENTRAL | DISTAL | TOTAL | TRACHEA |
| iVaw | Υ | Υ | Υ | Υ | Υ | С | С | Y | С | С | N/A |
| siVaw | С | С | С | С | С | С | С | С | С | С | N/A |
| iRaw | Υ | Υ | Υ | Υ | Υ | С | С | Υ | Υ | Υ | N/A |
| siRaw | С | C | С | C | С | C | С | С | С | С | N/A |
| iVlobe | Υ | Υ | Υ | Υ | Υ | С | С | N/A | N/A | С | N/A |
| iVlobepred | Υ | Υ | Υ | Υ | Υ | Υ | Υ | N/A | N/A | Υ | N/A |
| LAS | Υ | Υ | Υ | Υ | Υ | Υ | Υ | N/A | N/A | Υ | N/A |
| IALD | С | C | С | C | С | C | С | N/A | N/A | N/A | N/A |
| AT | Υ | Υ | Υ | Υ | Υ | Υ | Υ | N/A | N/A | Υ | N/A |
| BVD | Υ | Υ | Υ | Υ | Υ | Υ | Υ | N/A | N/A | Υ | N/A |
| iVaww | Υ | Υ | Υ | Υ | Υ | С | С | Υ | С | С | N/A |
| siVaww | С | С | С | С | С | С | С | С | С | С | N/A |
| Diameter | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | Υ |
| Length | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | Υ |
| Length/Diameter | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | С |

C = Endpoints will be Calculated by GSK (see Derived Data below)

#### Imaging Endpoints Calculated by GSK

iVaw LL = iVaw RLL + iVaw LLL

iVaw UL = iVaw RUL + iVaw RML + iVaw LUL

iVaw DISTAL = iVaw LL + iVaw UL

iVaw TOTAL = iVaw CENTRAL + iVaw DISTAL

iRaw LL = 1/ (1/iRaw RLL + 1/iRaw LLL)

iRaw UL = 1/ (1/iRaw RUL + 1/iRaw RML + 1/iRaw LUL)

iVlobe LL = iVlobe RLL + iVlobe LLL

iVlobe UL = iVlobe RUL + iVlobe RML + iVlobe LUL

iVlobe TOTAL = iVlobe LL + iVlobe UL

iVaww LL = iVaww RLL + iVaww LLL

iVaww UL = iVaww RUL + iVaww RML + iVaww LUL

iVaww DISTAL = iVaww LL + iVaww UL

iVaww TOTAL = iVaww CENTRAL + iVaww DISTAL

siVaw LLL = iVaw LLL / iVlobe LLL

siVaw LUL = iVaw LUL / iVlobe LUL

siVaw RML = iVaw RML / iVlobe RML

siVaw RUL = iVaw RUL / iVlobe RUL

siVaw RLL = iVaw RLL / iVlobe RLL

siVaw LL = iVaw LL / iVlobe LL

siVaw UL = iVaw UL / iVlobe UL

siVaw CENTRAL = iVaw CENTRAL / iVlobe TOTAL

siVaw DISTAL = iVaw DISTAL / iVlobe TOTAL

siVaw TOTAL = iVaw TOTAL / iVlobe TOTAL

siRaw LLL = iRaw LLL \* iVlobe LLL

siRaw LUL = iRaw LUL \* iVlobe LUL

siRaw RML = iRaw RML \* iVlobe RML

siRaw RUL = iRaw RUL \* iVlobe RUL

siRaw RLL = iRaw RLL \* iVlobe RLL

siRaw LL = iRaw LL \* iVlobe LL

siRaw UL = iRaw UL \* iVlobe UL

siRaw CENTRAL = iRaw CENTRAL \* iVlobe TOTAL siRaw DISTAL = iRaw DISTAL \* iVlobe TOTAL

siRaw TOTAL = iRaw TOTAL \* iVlobe TOTAL

siVaww LLL = iVaww LLL / iVlobe LLL

siVaww LUL = iVaww LUL / iVlobe LUL

siVaww RML = iVaww RML / iVlobe RML

siVaww RUL = iVaww RUL / iVlobe RUL

siVaww RLL = iVaww RLL / iVlobe RLL

siVaww LL = iVaww LL / iVlobe LL

siVaww UL = iVaww UL / iVlobe UL

siVaww CENTRAL = iVaww CENTRAL / iVlobe TOTAL

siVaww DISTAL = iVaww DISTAL / iVlobe TOTAL

siVaww TOTAL = iVaww TOTAL / iVlobe TOTAL

IALD LLL = 100 \* (iVlobe LLL TLC - iVlobe LLL FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD LUL = 100 \* (iVlobe LUL TLC - iVlobe LUL FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD RML = 100 \* (iVlobe RML TLC - iVlobe RML FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD RUL = 100 \* (iVlobe RUL TLC - iVlobe RUL FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD RLL = 100 \* (iVlobe RLL TLC - iVlobe RLL FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD LL = IALD RLL + IALD LLL

IALD UL = IALD RUL + IALD RML + IALD LUL

#### **Lung Function Parameters**

#### **Lung Function Parameters Calculated by GSK**

- FEV1 % Predicted (Men) = 4.30\*Height 0.029\*Age 2.49
- FEV1 % Predicted (Women) = 3.95\*Height 0.025\*Age 2.60

Formulas have been taken from Quanjer, 1993 Lung volumes and forced ventilator flows [accessed: 23rd July 2015] where height is measured in metres and age in years at screening.

#### **Rescue Medication Endpoints**

### Number of occasions bronchodilator taken in the last 24 per hours 4-week period derived by GSK

- Number of occasions bronchodilator taken in the last 24 hours were collected in the daily diary
- The table below shows which daily diary records are used to calculate the daily diary endpoints for each analysis time period. Any diary data collected in the post-treatment phase of the study will not be slotted.

| Daily | Record | |
|---------------------------|---------------------------|----------------------|
| Beginning Timepoint (day) | Ending Timepoint<br>(day) | Analysis Time Period |
| 1 | 28 | Weeks 1 – 4 |
| 29 | 56 | Weeks 5 – 8 |
| 57 | 84 | Weeks 9 – 12 |

Note: There is no Day 0. Any records with actual day>84 will not be assigned to a time period. Any records with actual day<0 may be assigned to a Week -1 (Baseline) time period

Note: Daily diary records that were not assigned to a time period will not be used in calculation of daily diary endpoints.

- For a subject to be counted in any time period for a given endpoint they must have at least one diary entry recorded for that endpoint during that time period.
- Any daily diary data that were collected post-study treatment discontinuation will be excluded from analysis, including four weekly period data summaries.
- If a subject has more than one daily diary record for any given day, the worst-case response on that day for each endpoint will be used in the summaries and analyses. i.e.

- the maximum number of occasions of bronchodilator use reported will be counted for the day in question and used to determine if it was a rescue-free day
- The mean number of occasions of rescue use per day and percentage of rescue-free days, will be calculated for each subject during the four weekly periods defined above.

## 13.6.4. Safety

#### **ECG Parameters**

#### **RR** Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value then do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Laboratory Values**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Places = '< x' becomes x 0.01
  - Example 2: 1 Decimal Places = '> x' becomes x + 0.1
  - Example 3: 0 Decimal Places = '< x' becomes x 1</li>

## 13.6.5. Pharmacodynamic and Biomarker

| Biomarker Category | Analyte | Method | Lab | Matrix | Total samples |
|---|---|---|---|---|---|
| Inflammatory Cytokine | IL-8 | MSD | Quest | Sputum | 4 |
| | IL-6 | MSD | Quest | Sputum | 4 |
| | $TNF\alpha$ | MSD | Quest | Sputum | 4 |
| Microbiome | Bacterial DNA | 16SRNA | GSK-RTP | Sputum | 4 |
| | Bacterial DNA | qPCR | GSK-RTP | Sputum | 4 |
| | Viral DNA | qPCR | GSK-RTP | Sputum | 4 |
| Transcriptomics | Human RNA | Affymetrix | Expression<br>Analysis | Blood | 4 |

#### NOTES:

- Sampling times: Screening, day 12, day 28 and day 84
- Inflammatory cytokine biomarkers are elevated in COPD patients. Expected to reduce with treatment.
- Microbiome biomarkers are drivers of exacerbations in COPD and are inhibited in preclinical disease studies
- PI3Kδ transcriptome analysis in FTIH study has 16 genes identified (sputum) showing a consistent response with dose – all are down regulated.

#### Pharmacodynamic and Biomarker

#### **Pharmacodynamic**

#### **PMNs Differentials**

- Percentage data may be arc-sine transformed especially if many of the percentage values are smaller than 20% or larger than 80%. The response variable, y, measured in radians, is sin-1sqrt{0.01\*p} where p is the differential percentage.
- If transformations are used then the results will be reported on the back-transformed scale, except where a transformed value:
  - o exceeds 0.01\*p/2 then the back-transformed value will be set equal to 100%
  - o is less than 0 then the back-transformed value will be set equal to 0%.

#### **Biomarkers**

## **Inflammatory Cytokines**

- In general, it is assumed that biomarker endpoints will require variance stabilising transformations, such as taking a
  loge transformation prior to analysis (and that summary statistics appropriate to loge normally distributed data will
  apply for all summaries). However, this assumption will be considered for each endpoint Individually prior to the
  generation of summary tables or statistical analysis, and if deemed more appropriate, a loge transformation will not
  be applied, or non-parametric methods may be employed.
- If transformations are used, then the results will be reported on the back-transformed scale unless otherwise stated.

#### **RNA** transcriptome

- Affymetrix microarray mRNA data will be normalised using RMA in ARRAY STUDIO v8.0 or later by the Statistical
  Consultancy Group (SCG) within GSK. After normalisation, the data will be quality assessed and any samples
  deemed as QC fails will be excluded from any further analysis. This quality assessment will involve looking for
  outlying signals in both the normalised expression data and the MAS5 QC metrics generated from each sample. If
  any samples are excluded, the remaining data will be re-normalised. The output from the normalization will be log2
  transformed mRNA intensity data.
- Summary mRNA data will be reviewed and a decision made on which probe sets are to be included in the SI dataset.
- Treatment ratios from the statistical analyses of mRNA intensity data will be converted to fold changes as follows:
  - o If ratio ≥ 1 then fold change = ratio
  - If ratio < 1 then fold change = -1/ratio</li>

The primary pharmacodynamic endpoint is based on a subset of probe sets defined as those that have previously identified immune cell mechanisms specifically related to neutrophil function.

The gene list that meets this criterion based on PII115119 D14 vs D1 gene changes, PII115117 and Metacore neutrophil pathways identified in PII115119 study. This gene list identified 258 genes in total after filtering for redundancy and was agreed by the study team is presented in Table 3.

Table 3 Gene List that have previously identified immune cell mechanisms specifically related to neutrophil function

| Gene | Source | Gene | Source |
|---|---|---|---|
| CD177 | PII115119 - Neutrophil migration | ITGAL | Metacore: IL8 Neutrophil migration |
| CXCR1 | PII115119 - Neutrophil migration | ADAM17 | Metacore: Inhibition of neutrophil migration |
| CXCR2 | PII115119 - Neutrophil migration | C5 | Metacore: Inhibition of neutrophil migration |
| FPR2 | PII115119 - Neutrophil migration | C5AR1 | Metacore: Inhibition of neutrophil migration |
| LTB4R | PII115119 - Neutrophil migration | CCR5 | Metacore: Inhibition of neutrophil migration |
| PAK1 | PII115119 - Neutrophil migration | CD34 | Metacore: Inhibition of neutrophil migration |
| PXN | PII115119 - Neutrophil migration | CALM1 | Metacore: Inhibition of neutrophil migration |
| PREX1 | PII115119 - Neutrophil migration | CALM2 | Metacore: Inhibition of neutrophil migration |
| TLN1 | PII115119 - Neutrophil migration | CALM3 | Metacore: Inhibition of neutrophil migration |
| SSH2 | PII115119 - Neutrophil migration | FPR1 | Metacore: Inhibition of neutrophil migration |
| F2RL1 | PII115119 - Neutrophil infection response | ICAM2 | Metacore: Inhibition of neutrophil migration |
| TLR10 | PII115119 - Neutrophil infection response | IL1B | Metacore: Inhibition of neutrophil migration |
| CEACAM3 | PII115119 - Neutrophil infection response | IL1R1 | Metacore: Inhibition of neutrophil migration |
| TREML2 | PII115119 - Neutrophil infection response | ITPR1 | Metacore: Inhibition of neutrophil migration |
| DEFB124 | PII115119 - Neutrophil infection response | ITPR2 | Metacore: Inhibition of neutrophil migration |
| CLEC4C | PII115119 - Neutrophil infection response | ITPR3 | Metacore: Inhibition of neutrophil migration |
| IFITM1 | PII115119 - Neutrophil infection response | SELL | Metacore: Inhibition of neutrophil migration |
| CR1 | PII115119 - Neutrophil infection response | MSN | Metacore: Inhibition of neutrophil migration |
| PMAIP1 | FTIH - GSK'557 response | NFKB1 | Metacore: Inhibition of neutrophil migration |
| S100P | FTIH - GSK'557 response | NFKB2 | Metacore: Inhibition of neutrophil migration |
| PTGS2 | FTIH - GSK'557 response | REL | Metacore: Inhibition of neutrophil migration |
| CCL20 | FTIH - GSK'557 response | RELA | Metacore: Inhibition of neutrophil migration |
| EGR3 | FTIH - GSK'557 response | RELB | Metacore: Inhibition of neutrophil migration |
| H1F0 | FTIH - GSK'557 response | PECAM1 | Metacore: Inhibition of neutrophil migration |
| NCOA3 | FTIH - GSK'557 response | PRKCA | Metacore: Inhibition of neutrophil migration |
| TARP | FTIH - GSK'557 response | PRKCB | Metacore: Inhibition of neutrophil migration |
| CEACAM1 | FTIH - GSK'557 response | PRKCD | Metacore: Inhibition of neutrophil migration |
| TTPAL | FTIH - GSK'557 response | PRKCE | Metacore: Inhibition of neutrophil migration |
| VPS37B | FTIH - GSK'557 response | PRKCG | Metacore: Inhibition of neutrophil migration |
| SYAP1 | FTIH - GSK'557 response | PRKCH | Metacore: Inhibition of neutrophil migration |
| SPTBN1 | FTIH - GSK'557 response | PRKCI | Metacore: Inhibition of neutrophil migration |

| Gene | Source | Gene | Source |
|---|---|---|---|
| EGR1 | FTIH - GSK'557 response | PRKCQ | Metacore: Inhibition of neutrophil migration |
| OSM | FTIH - GSK'557 response | PRKD1 | Metacore: Inhibition of neutrophil migration |
| TBC1D22A | FTIH - GSK'557 response | PRKD2 | Metacore: Inhibition of neutrophil migration |
| AKT1 | Metacore: IL8 Neutrophil migration | PRKD3 | Metacore: Inhibition of neutrophil migration |
| AKT2 | Metacore: IL8 Neutrophil migration | PLCB2 | Metacore: Inhibition of neutrophil migration |
| AKT3 | Metacore: IL8 Neutrophil migration | PTAFR | Metacore: Inhibition of neutrophil migration |
| ACTA1 | Metacore: IL8 Neutrophil migration | TLR2 | Metacore: Inhibition of neutrophil migration |
| ACTA2 | Metacore: IL8 Neutrophil migration | TLR4 | Metacore: Inhibition of neutrophil migration |
| ACTB | Metacore: IL8 Neutrophil migration | TNFRSF1A | Metacore: Inhibition of neutrophil migration |
| ACTC1 | Metacore: IL8 Neutrophil migration | TNFRSF1B | Metacore: Inhibition of neutrophil migration |
| ACTG1 | Metacore: IL8 Neutrophil migration | TNF | Metacore: Inhibition of neutrophil migration |
| ACTG2 | Metacore: IL8 Neutrophil migration | VAV1 | Metacore: Inhibition of neutrophil migration |
| MYH1 | Metacore: IL8 Neutrophil migration | EZR | Metacore: Inhibition of neutrophil migration |
| MYH10 | Metacore: IL8 Neutrophil migration | VCL | Metacore: Inhibition of neutrophil migration |
| MYH11 | Metacore: IL8 Neutrophil migration | ITGAM | Metacore: Inhibition of neutrophil migration |
| MYH13 | Metacore: IL8 Neutrophil migration | ABL1 | Metacore: Inhibition of neutrophil migration |
| MYH14 | Metacore: IL8 Neutrophil migration | JUN | Metacore: Inhibition of neutrophil migration |
| MYH15 | Metacore: IL8 Neutrophil migration | FOS | Metacore: Inhibition of neutrophil migration |
| MYH16 | Metacore: IL8 Neutrophil migration | MAPK11 | Metacore: Inhibition of neutrophil migration |
| MYH2 | Metacore: IL8 Neutrophil migration | MAPK12 | Metacore: Inhibition of neutrophil migration |
| MYH3 | Metacore: IL8 Neutrophil migration | MAPK13 | Metacore: Inhibition of neutrophil migration |
| MYH4 | Metacore: IL8 Neutrophil migration | MAPK14 | Metacore: Inhibition of neutrophil migration |
| MYH6 | Metacore: IL8 Neutrophil migration | BDKRB1 | Metacore: Neutrophil migration in Asthma |
| MYH7 | Metacore: IL8 Neutrophil migration | CCL15 | Metacore: Neutrophil migration in Asthma |
| MYH8 | Metacore: IL8 Neutrophil migration | CCL2 | Metacore: Neutrophil migration in Asthma |
| MYH9 | Metacore: IL8 Neutrophil migration | CCL5 | Metacore: Neutrophil migration in Asthma |
| MYL1 | Metacore: IL8 Neutrophil migration | CCL7 | Metacore: Neutrophil migration in Asthma |
| MYL12A | Metacore: IL8 Neutrophil migration | CCR1 | Metacore: Neutrophil migration in Asthma |
| MYL12B | Metacore: IL8 Neutrophil migration | CCR2 | Metacore: Neutrophil migration in Asthma |
| MYL2 | Metacore: IL8 Neutrophil migration | CCR3 | Metacore: Neutrophil migration in Asthma |
| MYL3 | Metacore: IL8 Neutrophil migration | CXCL5 | Metacore: Neutrophil migration in Asthma |
| MYL4 | Metacore: IL8 Neutrophil migration | CXCL1 | Metacore: Neutrophil migration in Asthma |
| MYL5 | Metacore: IL8 Neutrophil migration | CXCL2 | Metacore: Neutrophil migration in Asthma |
| MYL6 | Metacore: IL8 Neutrophil migration | CXCL3 | Metacore: Neutrophil migration in Asthma |
| MYL6B | Metacore: IL8 Neutrophil migration | HSPA14 | Metacore: Neutrophil migration in Asthma |
| MYL7 | Metacore: IL8 Neutrophil migration | HSPA1A | Metacore: Neutrophil migration in Asthma |
| MYL9 | Metacore: IL8 Neutrophil migration | HSPA1B | Metacore: Neutrophil migration in Asthma |
| MYLPF | Metacore: IL8 Neutrophil migration | HSPA1L | Metacore: Neutrophil migration in Asthma |
| ACTN1 | Metacore: IL8 Neutrophil migration | HSPA2 | Metacore: Neutrophil migration in Asthma |
| ACTN2 | Metacore: IL8 Neutrophil migration | HSPA4 | Metacore: Neutrophil migration in Asthma |
| ACTN3 | Metacore: IL8 Neutrophil migration | HSPA5 | Metacore: Neutrophil migration in Asthma |

| Gene | Source | Gene | Source |
|---|---|---|---|
| ACTN4 | Metacore: IL8 Neutrophil migration | HSPA6 | Metacore: Neutrophil migration in Asthma |
| ACTR2 | Metacore: IL8 Neutrophil migration | HSPA7 | Metacore: Neutrophil migration in Asthma |
| ACTR3 | Metacore: IL8 Neutrophil migration | HSPA8 | Metacore: Neutrophil migration in Asthma |
| ACTR3B | Metacore: IL8 Neutrophil migration | HSPA9 | Metacore: Neutrophil migration in Asthma |
| ARPC1A | Metacore: IL8 Neutrophil migration | MIF | Metacore: Neutrophil migration in Asthma |
| ARPC1B | Metacore: IL8 Neutrophil migration | CCL3 | Metacore: Neutrophil migration in Asthma |
| ARPC2 | Metacore: IL8 Neutrophil migration | PGF | Metacore: Neutrophil migration in Asthma |
| ARPC3 | Metacore: IL8 Neutrophil migration | TAC1 | Metacore: Neutrophil migration in Asthma |
| ARPC4 | Metacore: IL8 Neutrophil migration | TACR1 | Metacore: Neutrophil migration in Asthma |
| ARPC5 | Metacore: IL8 Neutrophil migration | KLK1 | Metacore: Neutrophil migration in Asthma |
| CFL1 | Metacore: IL8 Neutrophil migration | KLK10 | Metacore: Neutrophil migration in Asthma |
| CFL2 | Metacore: IL8 Neutrophil migration | KLK11 | Metacore: Neutrophil migration in Asthma |
| MAPK1 | Metacore: IL8 Neutrophil migration | KLK12 | Metacore: Neutrophil migration in Asthma |
| MAPK3 | Metacore: IL8 Neutrophil migration | KLK13 | Metacore: Neutrophil migration in Asthma |
| GNAI1 | Metacore: IL8 Neutrophil migration | KLK14 | Metacore: Neutrophil migration in Asthma |
| GNAI2 | Metacore: IL8 Neutrophil migration | KLK15 | Metacore: Neutrophil migration in Asthma |
| GNAI3 | Metacore: IL8 Neutrophil migration | KLK2 | Metacore: Neutrophil migration in Asthma |
| GNAO1 | Metacore: IL8 Neutrophil migration | KLK3 | Metacore: Neutrophil migration in Asthma |
| GNAZ | Metacore: IL8 Neutrophil migration | KLK4 | Metacore: Neutrophil migration in Asthma |
| GNB1 | Metacore: IL8 Neutrophil migration | KLK5 | Metacore: Neutrophil migration in Asthma |
| GNB2 | Metacore: IL8 Neutrophil migration | KLK6 | Metacore: Neutrophil migration in Asthma |
| GNB3 | Metacore: IL8 Neutrophil migration | KLK7 | Metacore: Neutrophil migration in Asthma |
| GNB4 | Metacore: IL8 Neutrophil migration | KLK8 | Metacore: Neutrophil migration in Asthma |
| GNB5 | Metacore: IL8 Neutrophil migration | KLK9 | Metacore: Neutrophil migration in Asthma |
| GNG10 | Metacore: IL8 Neutrophil migration | FLT1 | Metacore: Neutrophil migration in Asthma |
| GNG11 | Metacore: IL8 Neutrophil migration | RUNX1 | Metacore: Transcription regulation of granulocytes |
| GNG12 | Metacore: IL8 Neutrophil migration | CEBPA | Metacore: Transcription regulation of granulocytes |
| GNG13 | Metacore: IL8 Neutrophil migration | CEBPE | Metacore: Transcription regulation of granulocytes |
| GNG2 | Metacore: IL8 Neutrophil migration | ANPEP | Metacore: Transcription regulation of granulocytes |
| GNG3 | Metacore: IL8 Neutrophil migration | PTPRC | Metacore: Transcription regulation of granulocytes |
| GNG4 | Metacore: IL8 Neutrophil migration | E2F1 | Metacore: Transcription regulation of granulocytes |
| GNG5 | Metacore: IL8 Neutrophil migration | CSF3 | Metacore: Transcription regulation of granulocytes |
| GNG7 | Metacore: IL8 Neutrophil migration | CSF3R | Metacore: Transcription regulation of granulocytes |
| GNG8 | Metacore: IL8 Neutrophil migration | GATA1 | Metacore: Transcription regulation of granulocytes |
| GNGT1 | Metacore: IL8 Neutrophil migration | JAK1 | Metacore: Transcription regulation of granulocytes |
| GNGT2 | Metacore: IL8 Neutrophil migration | JAK2 | Metacore: Transcription regulation of granulocytes |
| ICAM1 | Metacore: IL8 Neutrophil migration | LRG1 | Metacore: Transcription regulation of granulocytes |
| CXCL8 | Metacore: IL8 Neutrophil migration | LTF | Metacore: Transcription regulation of granulocytes |
| ITGB2 | Metacore: IL8 Neutrophil migration | ELANE | Metacore: Transcription regulation of granulocytes |
| LIMK1 | Metacore: IL8 Neutrophil migration | LYZ | Metacore: Transcription regulation of granulocytes |
| MYLK | Metacore: IL8 Neutrophil migration | MXD1 | Metacore: Transcription regulation of granulocytes |

| Gene | Source | Gene | Source |
|---|---|---|---|
| MYLK2 | Metacore: IL8 Neutrophil migration | MAX | Metacore: Transcription regulation of granulocytes |
| MYLK3 | Metacore: IL8 Neutrophil migration | PRTN3 | Metacore: Transcription regulation of granulocytes |
| PPP1CB | Metacore: IL8 Neutrophil migration | MPO | Metacore: Transcription regulation of granulocytes |
| PPP1R12A | Metacore: IL8 Neutrophil migration | SPI1 | Metacore: Transcription regulation of granulocytes |
| PDPK1 | Metacore: IL8 Neutrophil migration | RARA | Metacore: Transcription regulation of granulocytes |
| PIK3CG | Metacore: IL8 Neutrophil migration | RXRA | Metacore: Transcription regulation of granulocytes |
| PIK3R5 | Metacore: IL8 Neutrophil migration | SOCS3 | Metacore: Transcription regulation of granulocytes |
| PIP5K1A | Metacore: IL8 Neutrophil migration | STAT3 | Metacore: Transcription regulation of granulocytes |
| PIP5K1B | Metacore: IL8 Neutrophil migration | STAT5A | Metacore: Transcription regulation of granulocytes |
| PIP5K1C | Metacore: IL8 Neutrophil migration | STAT5B | Metacore: Transcription regulation of granulocytes |
| PRKCZ | Metacore: IL8 Neutrophil migration | FES | Metacore: Transcription regulation of granulocytes |
| PLD1 | Metacore: IL8 Neutrophil migration | MYB | Metacore: Transcription regulation of granulocytes |
| PLPP6 | Metacore: IL8 Neutrophil migration | MYC | Metacore: Transcription regulation of granulocytes |
| RAC1 | Metacore: IL8 Neutrophil migration | CYBB | Metacore: Transcription regulation of granulocytes |
| RAC2 | Metacore: IL8 Neutrophil migration | NCF1 | Metacore: Transcription regulation of granulocytes |
| TLN2 | Metacore: IL8 Neutrophil migration | NCF2 | Metacore: Transcription regulation of granulocytes |

Gene names converted to Affymetrix probe ID, resulted in 638 probes in total, these are presented in Table 4.

Table 4 Probe Set that have previously identified immune cell mechanisms specifically related to neutrophil function

| Gene | Probe ID | Gene | Probe ID |
|-------|-------------------------|--------|--------------|
| ABL1 | 202123_s_at | KLK7 | 239381_at |
| ACTA1 | 203872_at | KLK8 | 1552319_a_at |
| ACTA2 | 200974_at | KLK8 | 206125_s_at |
| ACTA2 | 215787_at | KLK9 | 233687_s_at |
| ACTA2 | 243140_at | LIMK1 | 204356_at |
| ACTB | 200801_x_at | LIMK1 | 204357_s_at |
| ACTB | 213867_x_at | LIMK1 | 208372_s_at |
| ACTB | 224594_x_at | LRG1 | 228648_at |
| ACTB | AFFX-HSAC07/X00351_3_at | LTB4R | 210128_s_at |
| ACTB | AFFX-HSAC07/X00351_5_at | LTB4R | 216388_s_at |
| ACTB | AFFX-HSAC07/X00351_M_at | LTB4R | 236172_at |
| ACTC1 | 205132_at | LTF | 202018_s_at |
| ACTG1 | 201550_x_at | LYZ | 1555745_a_at |
| ACTG1 | 211970_x_at | LYZ | 213975_s_at |
| ACTG1 | 211983_x_at | MAPK1 | 1552263_at |
| ACTG1 | 211995_x_at | MAPK1 | 1552264_a_at |
| ACTG1 | 212363_x_at | MAPK1 | 208351_s_at |
| ACTG1 | 212988_x_at | MAPK1 | 212271_at |
| ACTG1 | 213214_x_at | MAPK1 | 224620_at |
| ACTG1 | 221607_x_at | MAPK1 | 224621_at |
| ACTG1 | 224585_x_at | MAPK1 | 229847_at |
| ACTG2 | 202274_at | MAPK11 | 206040_s_at |
| ACTG2 | 241148_at | MAPK11 | 211499_s_at |

| Gene | Probe ID | Gene | Probe ID |
|--------|--------------|--------|--------------|
| ACTN1 | 208636 at | MAPK11 | 211500 at |
| ACTN1 | 208637_x_at | MAPK12 | 1556340 at |
| ACTN1 | 211160_x_at | MAPK12 | 1556341 s at |
| ACTN1 | 237401 at | MAPK12 | 206106_at |
| ACTN1 | 203861_s_at | MAPK13 | 210058_at |
| ACTN2 | 203862_s_at | MAPK13 | 210059_s_at |
| ACTN2 | 203863_at | MAPK14 | 202530_at |
| ACTN2 | 203864_s_at | MAPK14 | 210449_x_at |
| ACTN2 | 206891 at | MAPK14 | 211087_x_at |
| ACTN3 | 200601_at | MAPK14 | 211561_x_at |
| ACTR2 | 1554390_s_at | MAPK3 | 212046_x_at |
| ACTR2 | 1558015_s_at | MAX | 208403_x_at |
| ACTR2 | 200727_s_at | MAX | 209331_s_at |
| ACTR2 | 200728_at | MAX | 209331_s_at |
| ACTR2 | 200729 s at | MAX | 210734_x_at |
| ACTR2 | 234210_x_at | MAX | 214108_at |
| ACTR2 | 234212 at | MIF | 217871_s_at |
| ACTR3 | 200996 at | MPO | 203948 s at |
| ACTR3 | 213101_s_at | MPO | 203949 at |
| ACTR3 | 213102_at | MSN | 200600 at |
| ACTR3 | 228603 at | MSN | 233749 at |
| ACTR3 | 239170 at | MXD1 | 206877_at |
| ACTR3B | 1555487_a_at | MXD1 | 226275 at |
| ACTR3B | 218868_at | MXD1 | 228846_at |
| ADAM17 | 205745_x_at | MYB | 204798 at |
| ADAM17 | 205746_s_at | MYB | 215152_at |
| ADAM17 | 213532_at | MYC | 202431 s at |
| ADAM17 | 237897 at | MYH1 | 205951_at |
| AKT1 | 207163_s_at | MYH10 | 212372_at |
| AKT2 | 1560689_s_at | MYH10 | 213067_at |
| AKT2 | 203808 at | MYH11 | 1568760 at |
| AKT2 | 203809_s_at | MYH11 | 201495_x_at |
| AKT2 | 211453_s_at | MYH11 | 201496_x_at |
| AKT2 | 225471_s_at | MYH11 | 201497_x_at |
| AKT2 | 226156 at | MYH11 | 207961_x_at |
| AKT2 | 236664_at | MYH11 | 228133_s_at |
| AKT3 | 212607_at | MYH11 | 228134_at |
| AKT3 | 212609_s_at | MYH11 | 239307 at |
| AKT3 | 219393_s_at | MYH13 | 208208_at |
| AKT3 | 222880_at | MYH14 | 217545_at |
| AKT3 | 224229_s_at | MYH14 | 217660_at |
| AKT3 | 242876_at | MYH14 | 219946_x_at |
| AKT3 | 242879_x_at | MYH14 | 226988_s_at |
| ANPEP | 202888_s_at | MYH14 | 232977_x_at |
| ANPEP | 234458_at | MYH14 | 234290_x_at |
| ANPEP | 234576_at | MYH15 | 215331_at |
| ARPC1A | 200950_at | MYH16 | 1564072_at |
| ARPC1B | 201954_at | MYH2 | 204631_at |
| ARPC2 | 207988_s_at | MYH3 | 205940_at |
| ARPC2 | 208679_s_at | MYH4 | 208148_at |
| ARPC2 | 213513_x_at | MYH6 | 214468_at |
| ARPC3 | 208736_at | MYH7 | 204737_s_at |
| ARPC4 | 211672_s_at | MYH7 | 216265_x_at |
| ARPC4 | 217817_at | MYH8 | 206717_at |

| Gene | Probe ID | Gene | Probe ID |
|---------|--------------|--------|--------------|
| ARPC4 | 217818_s_at | MYH8 | 34471 at |
| ARPC5 | 1555797 a at | MYH9 | 211926 s at |
| ARPC5 | 1569325 at | MYL1 | 209888_s_at |
| ARPC5 | 211963_s_at | MYL12A | 1555976_s_at |
| ARPC5 | 237387 at | MYL12A | 1555977_at |
| BDKRB1 | 207510_at | MYL12A | 1555978_s_at |
| C5 | 205500_at | MYL12A | 201318_s_at |
| C5AR1 | 220088_at | MYL12A | 201319_at |
| CCL15 | 210390_s_at | MYL12B | 221474_at |
| CCL2 | 216598_s_at | MYL2 | 209742_s_at |
| CCL20 | 205476_at | MYL3 | 205589_at |
| CCL3 | 205114_s_at | MYL4 | 210088_x_at |
| CCL5 | 1405_i_at | MYL4 | 210395_x_at |
| CCL5 | 1555759_a_at | MYL4 | 216054_x_at |
| CCL5 | 204655 at | MYL4 | 217274_x_at |
| CCL7 | 208075 s at | MYL5 | 205145 s at |
| CCR1 | 205098 at | MYL6 | 212082_s_at |
| CCR1 | 205099_s_at | MYL6 | 214002 at |
| CCR2 | 206978_at | MYL6B | 204173_at |
| CCR2 | 207794 at | MYL7 | 219942_at |
| CCR3 | 208304 at | MYL9 | 201058_s_at |
| CCR5 | 206991_s_at | MYL9 | 244149 at |
| CD177 | 219669 at | MYLK | 1563466 at |
| CD34 | 209543 s at | MYLK | 1568770 at |
| CEACAM1 | 206576_s_at | MYLK | 1569956 at |
| CEACAM1 | 209498_at | MYLK | 202555 s at |
| CEACAM1 | 210610_at | MYLK | 224823_at |
| CEACAM1 | 211883_x_at | MYLK2 | 231792_at |
| CEACAM1 | 211889_x_at | MYLK3 | 1562411_at |
| CEACAM3 | 208052_x_at | MYLK3 | 1568925_at |
| CEACAM3 | 210789_x_at | MYLK3 | 1568926_x_at |
| CEACAM3 | 217209_at | MYLK3 | 217623_at |
| CEBPA | 204039_at | MYLK3 | 238834_at |
| CEBPE | 214523_at | MYLPF | 205163_at |
| CFL1 | 1555730_a_at | NCF1 | 204961_s_at |
| CFL1 | 200021_at | NCF1 | 214084_x_at |
| CFL1 | 230870_at | NCF2 | 209949_at |
| CFL1 | 236792_at | NCOA3 | 1562439_at |
| CFL2 | 224352_s_at | NCOA3 | 207700_s_at |
| CFL2 | 224663_s_at | NCOA3 | 209060_x_at |
| CFL2 | 233496_s_at | NCOA3 | 209061_at |
| CLEC4C | 1552552_s_at | NCOA3 | 209062_x_at |
| CLEC4C | 1555687_a_at | NCOA3 | 211352_s_at |
| CR1 | 206244_at | NFKB1 | 209239_at |
| CR1 | 208488_s_at | NFKB2 | 207535_s_at |
| CR1 | 217484_at | NFKB2 | 209636_at |
| CR1 | 217552_x_at | NFKB2 | 211524_at |
| CR1 | 244313_at | OSM | 214637_at |
| CSF3 | 207442_at | OSM | 230170_at |
| CSF3R | 1553297_a_at | PAK1 | 1565772_at |
| CSF3R | 203591_s_at | PAK1 | 209615_s_at |
| CXCL1 | 204470_at | PAK1 | 226507_at |
| CXCL2 | 1569203_at | PAK1 | 230100_x_at |
| CXCL2 | 209774_x_at | PDPK1 | 204524_at |

| Gene | Probe ID | Gene | Probe ID |
|---|---|---|---|
| CXCL2 | 230101 at | PDPK1 | 221244 s at |
| CXCL3 | 207850 at | PDPK1 | 224986 s at |
| CXCL5 | 207852 at | PDPK1 | 244629_s_at |
| CXCL5 | 214974_x_at | PDPK1 | 244630_at |
| CXCL5 | 215101_s_at | PDPK1 | 32029_at |
| CXCL8 | 202859_x_at | PECAM1 | 1558397_at |
| CXCL8 | 211506_s_at | PECAM1 | 1559921 at |
| CXCR1 | 207094_at | PECAM1 | 208981 at |
| CXCR2 | 207008_at | PECAM1 | 208982 at |
| CYBB | 203922_s_at | PECAM1 | 208983_s_at |
| CYBB | 203923_s_at | PGF | 209652_s_at |
| CYBB | 217431_x_at | PGF | 215179_x_at |
| CYBB | 233538_s_at | PIK3CG | 206369_s_at |
| DEFB124 | 1568375_at | PIK3CG | 206370_at |
| DEFB124 | 1568377_x_at | PIK3CG | 239294_at |
| E2F1 | 2028_s_at | PIK3R5 | 220566_at |
| E2F1 | 204947_at | PIK3R5 | 227553_at |
| EGR1 | 201693_s_at | PIK3R5 | 227645_at |
| EGR1 | 201694_s_at | PIP5K1A | 207391_s_at |
| EGR1 | 227404_s_at | PIP5K1A | 210256_s_at |
| EGR3 | 206115_at | PIP5K1A | 211205_x_at |
| ELANE | 206871_at | PIP5K1B | 205632_s_at |
| EZR | 208621_s_at | PIP5K1B | 217477_at |
| EZR | 208622_s_at | PIP5K1C | 212518_at |
| EZR | 208623_s_at | PLCB2 | 204046_at |
| EZR | 217230_at | PLCB2 | 210388_at |
| EZR | 217234_s_at | PLD1 | 1557126_a_at |
| FES | 205418_at | PLD1 | 177_at |
| FLT1 | 204406_at | PLD1 | 205203_at |
| FLT1 | 210287_s_at | PLD1 | 215723_s_at |
| FLT1 | 222033_s_at | PLD1 | 215724_at |
| FLT1 | 226497_s_at | PLD1 | 226636_at |
| FLT1 | 226498_at | PLD1 | 232530_at |
| FLT1 | 232809_s_at | PLPP6 | 227385_at |
| FOS | 209189_at | PMAIP1 | 204285_s_at |
| FPR1 | 205118_at | PMAIP1 | 204286_s_at |
| FPR1 | 205119_s_at | PPP1CB | 201407_s_at |
| FPR2 | 210772_at | PPP1CB | 201408_at |
| FPR2 | 210773_s_at | PPP1CB | 201409_s_at |
| GATA1 | 1555590_a_at | PPP1CB | 228222_at |
| GATA1 | 210446_at | PPP1R12A | 201602_s_at |
| GNAI1 | 209576_at | PPP1R12A | 201603_at |
| GNAI1 | 227692_at | PPP1R12A | 201604_s_at |
| GNAI2 | 201040_at | PREX1 | 224909_s_at |
| GNAI2 | 215996_at | PREX1<br>PRKCA | 224925_at |
| GNAI2 | 217271_at | | 1560074_at |
| GNAI3<br>GNAI3 | 201179_s_at | PRKCA | 206923_at |
| GNAI3<br>GNAI3 | 201180_s_at | PRKCA<br>PRKCA | 213093_at |
| GNA01 | 201181_at | PRKCA | 215194_at |
| GNAO1 | 204762_s_at<br>204763_s_at | PRKCB | 215195_at<br>207957_s_at |
| GNAO1 | 215912_at | PRKCB | 209685_s_at |
| GNAO1 | 231951_at | PRKCB | 227817_at |
| GNAZ | 204993_at | PRKCB | 227824 at |
| UNAL | 20 <del>1</del> 333_at | LUVOD | 221024_al |

| Gene | Probe ID | Gene | Probe ID |
|---------------|----------------------------|--------------|--------------|
| GNB1 | 200744_s_at | PRKCB | 228795 at |
| GNB1 | 200745_s_at | PRKCB | 230437 s at |
| GNB1 | 200746_s_at | PRKCD | 202545 at |
| GNB2 | 200852_x_at | PRKCE | 206248 at |
| GNB3 | 206047_at | PRKCE | 226101 at |
| GNB4 | 223487_x_at | PRKCE | 234089 at |
| GNB4 | 223488_s_at | PRKCE | 236459_at |
| GNB4 | 225710_at | PRKCE | 239011 at |
| GNB5 | 1554346_at | PRKCG | 206270 at |
| GNB5 | 204000_at | PRKCG | 236195_x_at |
| GNB5 | 207124_s_at | PRKCH | 206099 at |
| GNB5 | 211871_x_at | PRKCH | 218764_at |
| GNB5 | 242404_at | PRKCH | 230124_at |
| GNG10 | 201921 at | PRKCI | 209677_at |
| GNG11 | 204115_at | PRKCI | 209678_s_at |
| GNG11 | 239942 at | PRKCI | 213518_at |
| GNG12 | 1555240_s_at | PRKCQ | 210038_at |
| GNG12 | 212294 at | PRKCQ | 210039_s_at |
| GNG12 | 222834_s_at | PRKCZ | 1569748 at |
| GNG13 | 220806_x_at | PRKCZ | 202178 at |
| GNG2 | 1555766_a_at | PRKD1 | 205880_at |
| GNG2 | 223943_s_at | PRKD1 | 217705_at |
| GNG2 | 224964_s_at | PRKD2 | 209282 at |
| GNG2 | 224965 at | PRKD2 | 241669_x_at |
| GNG3 | 222005_s_at | PRKD2 | 38269 at |
| GNG4 | 1555765_a_at | PRKD3 | 1554910 at |
| GNG4 | 1555867 at | PRKD3 | 211084_x_at |
| GNG4 | 1566513 a at | PRKD3 | 218236_s_at |
| GNG4 | 205184 at | PRKD3 | 222565_s_at |
| GNG5 | 207157_s_at | PRKD3 | 242549_at |
| GNG7 | 206896_s_at | PRTN3 | 207341 at |
| GNG7 | 214227_at | PTAFR | 206278_at |
| GNG7 | 228831_s_at | PTAFR | 211661_x_at |
| GNG7 | 232043_at | PTAFR | 227184 at |
| GNG7<br>GNG8 | 233416_at | PTGS2 | 1554997_a_at |
| GNG8 | 234284_at | PTGS2 | 204748_at |
| GNG0<br>GNGT1 | 207166_at | PTPRC | 1552480_s_at |
| GNGT2 | 235139_at | PTPRC | 1569830_at |
| H1F0 | 208886_at | PTPRC | 207238_s_at |
| HSPA14 | 219212_at | PTPRC | 212587_s_at |
| HSPA14 | 226887_at | PTPRC | 212588 at |
| HSPA14 | 227650_at | PXN | 201087_at |
| HSPA1L | 210189_at | PXN | 211823_s_at |
| HSPA1L | 233694_at | RAC1 | 1567457_at |
| HSPA2 | 211538 s at | RAC1 | 1567458 s at |
| HSPA4 | 208814_at | RAC1 | 208640_at |
| HSPA4 | 208815_x_at | RAC1 | 208641_s_at |
| HSPA4 | 211015_s_at | RAC2 | 207419_s_at |
| HSPA4 | 211015_s_at<br>211016_x_at | RAC2 | 213603_s_at |
| HSPA5 | 211936_at | RAC2<br>RARA | 1565358_at |
| HSPA5 | 230031_at | RARA | 203749_s_at |
| HSPA6 | 230031_at | RARA | 203750_s_at |
| HSPA6 | 213418_at | RARA | 211605_s_at |
| HSPA8 | | RARA | 216300_x_at |
| ПЭГАО | 208687_x_at | KAKA | 210000_X_at |

| Gene | Probe ID | Gene | Probe ID |
|--------------|--------------------------|----------|--------------|
| HSPA8 | 210338_s_at | REL | 206035 at |
| HSPA8 | 221891_x_at | REL | 206036_s_at |
| HSPA8 | 224187_x_at | REL | 228812 at |
| HSPA9 | 200690 at | REL | 235242 at |
| HSPA9 | 200691_s_at | REL | 239486 at |
| HSPA9 | 200692_s_at | RELA | 201783_s_at |
| HSPA9 | 232200 at | RELA | 209878_s_at |
| ICAM1 | 202637_s_at | RELA | 230202 at |
| ICAM1 | 202638_s_at | RELB | 205205 at |
| ICAM1 | 215485_s_at | RXRA | 202426_s_at |
| ICAM2 | 204683 at | RXRA | 202449_s_at |
| ICAM2 | 213620_s_at | S100P | 204351 at |
| IFITM1 | 201601 x at | SELL | 204563 at |
| IFITM1 | 214022_s_at | SOCS3 | 206359 at |
| IL1B | 205067 at | SOCS3 | 206360_s_at |
| IL1B | 39402 at | SOCS3 | 214105 at |
| IL1R1 | 202948 at | SOCS3 | 227697 at |
| IL1R1 | 215561_s_at | SPI1 | 205312_at |
| ITGAL | 1554240_a_at | SPTBN1 | 200671_s_at |
| ITGAL | 213475 s at | SPTBN1 | 200671_5_dt |
| ITGAM | 205785 at | SPTBN1 | 212071_s_at |
| ITGAM | 205786 s at | SPTBN1 | 213914 s at |
| ITGB2 | 1555349_a_at | SPTBN1 | 214856 at |
| ITGB2 | 202803 s at | SPTBN1 | 215918 s at |
| ITGB2 | 236988 x at | SPTBN1 | 226342 at |
| ITPR1 | 1562373_at | SPTBN1 | 226765 at |
| ITPR1 | 203710 at | SPTBN1 | 228246 s at |
| ITPR1 | 211323 s at | SPTBN1 | 230540 at |
| ITPR1 | 216944 s at | SPTBN1 | 242220 at |
| ITPR1 | 240052 at | SSH2 | 1554114 s at |
| ITPR2 | 202660 at | SSH2 | 1555423 at |
| ITPR2 | 202661 at | SSH2 | 1555425 x at |
| ITPR2 | 202662_s_at | SSH2 | 1560306 at |
| ITPR2 | 211360_s_at | SSH2 | 226080 at |
| ITPR3 | 201187_s_at | STAT3 | 208991 at |
| ITPR3 | 201188 s at | STAT3 | 208992 s at |
| ITPR3 | 201189_s_at | STAT3 | 225289_at |
| ITPR3 | 239542_at | STAT3 | 243213_at |
| JAK1 | 1552610 a at | STAT5A | 203010_at |
| JAK1 | 1552611_a_at | STAT5B | 1555086_at |
| JAK1 | 201648_at | STAT5B | 1555088_x_at |
| JAK1 | 239695_at | STAT5B | 205026_at |
| JAK1 | 240613_at | STAT5B | 212549_at |
| JAK1<br>JAK2 | 1562031_at | STAT5B | 212550 at |
| JAK2 | | SYAP1 | 225154_at |
| JAK2 | 205841_at<br>205842_s_at | TAC1 | 206552_s_at |
| JUN | 201464_x_at | TACR1 | 208048_at |
| JUN | 201465_s_at | TACR1 | 208049_s_at |
| JUN | 201466_s_at | TACR1 | 210637_at |
| JUN<br>KLK1 | 213281_at | TACR1 | 230908_at |
| | 216699_s_at | TARP | 211144_x_at |
| KLK10 | 209792_s_at | TARP | 216920_s_at |
| KLK10 | 215808_at | TARP | 217381_s_at |
| KLK11 | 205470_s_at | TBC1D22A | 209650_s_at |

| Gene | Probe ID | Gene | Probe ID |
|-------|--------------|----------|--------------|
| KLK12 | 220782_x_at | TBC1D22A | 210144_at |
| KLK12 | 233586_s_at | TBC1D22A | 33778_at |
| KLK12 | 234316_x_at | TLN1 | 203254_s_at |
| KLK13 | 205783_at | TLN1 | 232763_at |
| KLK13 | 216670_at | TLN1 | 236132_at |
| KLK13 | 217315_s_at | TLN2 | 212701_at |
| KLK14 | 220573_at | TLN2 | 212703_at |
| KLK15 | 221462_x_at | TLN2 | 232625_at |
| KLK15 | 233477_at | TLR10 | 223750_s_at |
| KLK15 | 234495_at | TLR10 | 223751_x_at |
| KLK15 | 234966_at | TLR2 | 204924_at |
| KLK2 | 1555545_at | TLR4 | 1552798_a_at |
| KLK2 | 209854_s_at | TLR4 | 221060_s_at |
| KLK2 | 209855_s_at | TLR4 | 224341_x_at |
| KLK2 | 210339_s_at | TLR4 | 232068_s_at |
| KLK3 | 204582_s_at | TNF | 1563357_at |
| KLK3 | 204583_x_at | TNF | 207113_s_at |
| KLK3 | 231629_x_at | TNFRSF1A | 207643_s_at |
| KLK4 | 1555697_at | TNFRSF1B | 203508_at |
| KLK4 | 1555737_a_at | TREML2 | 219748_at |
| KLK4 | 224062_x_at | TTPAL | 219633_at |
| KLK4 | 231782_s_at | TTPAL | 228031_at |
| KLK4 | 233854_x_at | VAV1 | 206219_s_at |
| KLK5 | 222242_s_at | VCL | 200930_s_at |
| KLK6 | 204733_at | VCL | 200931_s_at |
| KLK7 | 205778_at | VPS37B | 221704_s_at |

## 13.7. Appendix 7: Reporting Standards for Missing Data

## 13.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as Subject whom have completed their final visit (day 84).</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 13.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| Outliers | <ul> <li>Any participants excluded from the summaries and/or statistical analyses will be<br/>documented along with the reason for exclusion in the clinical study report.</li> </ul> |
| PD | <ul> <li>Any values below the Lower Limit of Quantification (LLQ) will be assigned a value of ½ LLQ for display purposes in Figures and for computation of summary statistics. Any values above the Upper Limit of Quantification (ULQ) will be assigned to the ULQ for display purposes in Figures and for computation of summary statistics. Where biomarker concentrations are from an assay of an increased dilution factor the LLQ and ULQ will be multiplied by this factor. Note: Values sent to biostatistics are raw and have not taken into account dilution factor. LLQ and ULQ need to be taken into account prior to dilution factor and then imputed. Then Dilution factor needs to be applied. E.g. if raw value is 10 and dilution factor is 1:2 and ULD is 15, then this value is valid, but the final value should be 20.</li> <li>If the number of LLQ (and/or ULQ) values is large for an individual biomarker then an alternative analysis method, such as TOBIT analysis, may be required. "Large" is hard to define prospectively and may depend upon the dataset in question. Any such methodology will be documented in the statistical contributions to the study report.</li> <li>Imputed values will be used in tables and figures, unless the proportion of imputed values at a given time point is large, in which case the summary statistics may not be presented for that time point and/or alternative actions will be taken and documented in the study report.</li> <li>Where values are imputed, the number of such imputations will be included as a summary statistic in the relevant summary tables.</li> </ul> |
| HRCT | <ul> <li>No missing data imputation methods will be used.</li> <li>Note that for the HRCT data, there may be instances such that measurements from a particular Lobe cannot be distinguished between another Lobe, for example the iVlobe may be measured from both the LLL and LUL lobes. In such a case, the Lobe will be denoted as LLL + LUL. Therefore, for the statistical analysis purpose, since analysis is</li> </ul> |

| Element | Reporting Det | ail | | | | |
|---|---|---|---|---|---|---|
| | therefore n | on a lobar level, the LLL and LUL Lobes will be set to missing and will not be included in the analysis. Below is a table of all possible scenarios, data is set to missing and not used in the statistical analysis: | | | | |
| | | | | Lobes | | Label |
| | | RUL | RUL RML RLL LUL LLL | | LLL | Labei |
| | | Х | X X | | | RUL + RML |
| | | x x RML + RLL | | | | |
| | | Х | x RUL + RLL | | | |
| | | | 1 | İ | 1 | DIU - DIU - DII |
| | | Χ | Χ | Χ | | RUL + RML + RLL |

## 13.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

## 13.8. Appendix 8: Values of Potential Clinical Importance

## 13.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units Category Clinical Concern Range | | cern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Hematocrit | Ratio of | Male | | 0.54 |
| Hematocht | 1 | Female | | 0.54 |
| Llaamadahin | g/L | Male | | 180 |
| Haemoglobin | | Female | | 180 |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | ≥1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 13.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-----------------------|-------|------------------------|-----------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 500 [1] |
| Absolute PR Interval | msec | < 110 [1] | > 220 [2] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [2] |

### NOTES:

## 13.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

<sup>[1]</sup> An upper limit of 450 would represent standard ECG values of PCI for HV studies, this has been extended to 500 as often with exacerbations the treatment can result in a short term prolongation of QTc up to 500.

<sup>[2]</sup> Represent standard ECG values of PCI for HV studies

## 13.9. Appendix 9: Abbreviations & Trade Marks

## 13.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| A&R | Analysis and Reporting |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| AT | Air Trapping Score (% of iVlobe) |
| BVD | Blood Vessel Density (% of iVlobe) |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CENTRAL | Central lung region |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CT | Computed tomography |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| Diameter | Diameter |
| DISTAL | Distal lung region |
| DLco | Diffusion capacity |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FEV <sub>1</sub> | Forced expiratory volume in 1 second |
| FRI | Functional respiratory imaging |
| FRC | Functional residual capacity |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| HRCT | High Resolution Computed Tomography |
| IA | Interim Analysis |
| IALD | Internal Airflow Lobar Distribution |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IL-8 | Interleukin 8 |
| IL-6 | Interleukin 6 |

| Abbreviation | Description |
|---|---|
| IMMS | International Modules Management System |
| IP | Investigational Product |
| iRaw | Imaging Airway Resistance |
| ITT | Intent-To-Treat |
| iVlobe | Lobar Volume |
| iVlobepred<br>iVaw | Percent Predicted Lobar Volume |
| | Imaging Airway Volume |
| iVaww | Airway Wall Volume |
| LAS | Low Attenuation Score (% of iVlobe) |
| Length | Length |
| LL | Lung, lower lobes |
| LLL | Lung, left lower lobe |
| LOC | Last Observation Carries Forward |
| LUL | Lung, left upper lobe |
| LUL+LLL | Lung, left upper and lower lobe |
| MMP9 | Matrix metallopeptidase 9 |
| MMRC | Modified Medical Research Council |
| MMRM | Mixed Model Repeated Measures |
| NQ | Non-quantifiable |
| OTU | Operational Taxonomic Unit |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PEF | peak expiratory flow |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| qPCR | Quantitative polymerase chain reaction |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RLL | Lung, right lower lobe |
| RML | Lung, right middle lobe |
| RML+RLL | Lung, right middle and lower lobe |
| RUL | Lung, right upper lobe |
| RUL+RLL | Lung, right upper and lower lobe |
| RUL+RML | Lung, right upper and middle lobe |
| RUL+RML+RLL | Lung, right upper, middle and lower lobe |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| sGaw | Specific conductance |
| siRaw | Specific Imaging Airway Resistance |
| | epocino inaging / in ray i toolotanoo |

| Abbreviation | Description |
|--------------|--------------------------------|
| siVaw | Specific Imaging Airway Volume |
| siVaww | Specific Airway Wall Volume |
| SoC | Standard of Care |
| SOP | Standard Operation Procedure |
| sRaw | Specific Resistance |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TLC | Total lung capacity |
| TNFα | Tumor necrosis factor alpha |
| TOTAL | Total lung region |
| TRACHEA | Trachea |
| UL | Lung, upper lobes |

## 13.9.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| ELLIPTA |
| HARP |
| RAMOS NG |
| RANDALL NG |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|
| FluidDA |
| Quest |
| SAS |
| WinNonlin |

## 13.10. Appendix 10: List of Data Displays

## 13.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|---------|
| Study Population | 1.1 to 1.17 | N/A |
| Efficacy | 2.1 to 2.68 | 2.1 |
| Safety | 3.1 to 3.20 | N/A |
| Pharmacokinetic | 4.1 to 4.4 | 4.1 |
| Pharmacodynamic and / or Biomarker | 6.1 to 6.21 | 6.1 |
| Section | List | ings |
| ICH Listings 1 to 34 | | |
| Other Listings | 35 t | o 49 |

## 13.10.2. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

## 13.10.3. Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1.1. | All Subjects | ES1 | Summary of Subject Disposition | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | All Subjects | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC |
| 1.3. | APE | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| 1.4. | All Subjects | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Protoc | ol Deviation | | | | |
| 1.5. | All Subjects | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Popula | tion Analysed | | | | |
| 1.6. | APE | SP1 | Summary of Study Populations | IDSL | SAC |
| 1.7. | All Subjects | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.8. | All Subjects | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.9. | APE | DM11 | Summary of Age Ranges | EudraCT | SAC |
| 1.10. | All Subjects | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |
| 1.11. | All Subjects | DM6 | Summary of Race and Racial Combinations Details | | SAC |
| 1.12. | All Subjects | PII116678/final/<br>Table 2.109 | Summary of Index Exacerbation Severity | | |

| Study | Population Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Prior a | nd Concomitan | t Medications | | | |
| 1.13. | All Subjects | MH1 | Summary of Current Medical Conditions | ICH E3 | SAC |
| 1.14. | All Subjects | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC |
| 1.15. | All Subjects | CM1 | Summary of Prior Medications | ICH E3 | SAC |
| 1.16. | All Subjects | CM1 | Summary of Concomitant Medications | ICH E3 | SAC |
| Exposi | ure and Treatme | ent Compliance | | | |
| 1.17. | All Subjects | EX1 | Summary of Exposure to Study Treatment | ICH E3 Include Daily Dose, Cumulative does and Days on study drug per template. | SAC |
| Family | Family History of Cardiovascular Risk Factors | | | | |
| 1.18. | All Subjects | FH1 | Summary of Family History of Cardiovascular Risk Factors | | SAC |

## 13.10.4. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| HRCT | maging Endpo | ints | | | |
| 2.1. | All Subjects | PII116678/ final/<br>Table 2.1 | Summary of iVaw (mL) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used | SAC |
| 2.2. | All Subjects | PII116678/ final/<br>Table 2.2 | Summary of iVaw (mL) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.3. | All Subjects | PII116678/ final/<br>Table 2.3 | Summary of iVaw (mL) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used | SAC |
| 2.4. | All Subjects | PII116678/ final/<br>Table 2.4 | Summary of iVaw (mL) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used Footnote baseline | SAC |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.5. | All Subjects | PII116678/ final/<br>Table 2.9 | Summary of siVaw (mL/L) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used | SAC |
| 2.6. | All Subjects | PII116678/ final/<br>Table 2.10 | Summary of siVaw (mL/L) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.7. | All Subjects | PII116678/final/<br>Table 2.11 | Summary of siVaw (mL/L) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used | SAC |
| 2.8. | All Subjects | PII116678/final/<br>Table 2.12 | Summary of siVaw (mL/L) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.9. | All Subjects | PII116678/final/<br>Table 2.17 | Summary of iRaw (kPa*s/L) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No longitudinal endpoints Footnote any transformations used | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.10. | All Subjects | PII116678/final/<br>Table 2.18 | Summary of iRaw (kPa*s/L) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No longitudinal endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.11. | All Subjects | PII116678/final/<br>Table 2.19 | Summary of iRaw (kPa*s/L) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page No longitudinal endpoints Footnote any transformations used | SAC |
| 2.12. | All Subjects | PII116678/final/<br>Table 2.20 | Summary of iRaw (kPa*s/L) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page No longitudinal endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.13. | All Subjects | PII116678/final/<br>Table 2.25 | Summary of siRaw (kPa*s) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No longitudinal endpoints Footnote any transformations used | SAC |
| Efficac | Efficacy: Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable | | | |
| 2.14. | All Subjects | PII116678/final/<br>Table 2.26 | Summary of siRaw (kPa*s) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No longitudinal endpoints Footnote any transformations used Footnote baseline | SAC | | | |
| 2.15. | All Subjects | PII116678/final/<br>Table 2.27 | Summary of siRaw (kPa*s) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page No longitudinal endpoints Footnote any transformations used | SAC | | | |
| 2.16. | All Subjects | PII116678/final/<br>Table 2.28 | Summary of siRaw (kPa*s) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page No longitudinal endpoints Footnote any transformations used Footnote baseline | SAC | | | |
| 2.17. | All Subjects | PII116678/final/<br>Table 2.33 | Summary of iVlobe (L) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC | | | |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.18. | All Subjects | PII116678/final/<br>Table 2.34 | Summary of iVlobe (L) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.19. | All Subjects | PII116678/final/<br>Table 2.35 | Summary of iVlobe (L) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.20. | All Subjects | PII116678/final/<br>Table 2.36 | Summary of iVlobe (L) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.21. | All Subjects | PII116678/final/<br>Table 2.41 | Summary of Percent Predicted iVlobe (%) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Note in HARP to output (%) it may be necessary to input (%%) | SAC |
| 2.22. | All Subjects | PII116678/final/<br>Table 2.42 | Summary of Percent Predicted iVlobe (%) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline Note in HARP to output (%) it may be necessary to input (%%) | SAC |
| 2.23. | All Subjects | PII116678/final/<br>Table 2.43 | Summary of Percent Predicted iVlobe (%) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Note in HARP to output (%) it may be necessary to input (%%) | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.24. | All Subjects | PII116678/final/<br>Table 2.44 | Summary of Percent Predicted iVlobe (%) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline Note in HARP to output (%) it may be necessary to input (%%) | SAC |
| 2.25. | All Subjects | PII116678/final/<br>Table 2.49 | Summary of LAS (% of iVlobe) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.26. | All Subjects | PII116678/final/<br>Table 2.50 | Summary of LAS (% of iVlobe) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.27. | All Subjects | PII116678/final/<br>Table 2.51 | Summary of LAS (% of iVlobe) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.28. | All Subjects | PII116678/final/<br>Table 2.52 | Summary of LAS (% of iVlobe) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.29. | All Subjects | PII116678/final/<br>Table 2.55 | Summary of IALD (%) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.30. | All Subjects | PII116678/final/<br>Table 2.56 | Summary of IALD (%) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.31. | All Subjects | PII116678/final/<br>Table 2.57 | Summary of IALD (%) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central, Distal and Total do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.32. | All Subjects | PII116678/final/<br>Table 2.58 | Summary of IALD (%) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central, Distal and Total do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.33. | All Subjects | PII116678/final/<br>Table 2.61 | Summary of AT (% of iVlobe) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.34. | All Subjects | PII116678/final/<br>Table 2.62 | Summary of AT (% of iVlobe) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.35. | All Subjects | PII116678/final/<br>Table 2.63 | Summary of AT (% of iVlobe) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.36. | All Subjects | PII116678/final/<br>Table 2.64 | Summary of AT (% of iVlobe) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.37. | All Subjects | PII116678/final/<br>Table 2.67 | Summary of BVD (% of iVlobe) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.38. | All Subjects | PII116678/final/<br>Table 2.68 | Summary of BVD (% of iVlobe) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.39. | All Subjects | PII116678/final/<br>Table 2.69 | Summary of BVD (% of iVlobe) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.40. | All Subjects | PII116678/final/<br>Table 2.70 | Summary of BVD (% of iVlobe) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.41. | All Subjects | PII116678/final/<br>Table 2.73 | Summary of iVaww (mL) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used | SAC |
| 2.42. | All Subjects | PII116678/final/<br>Table 2.74 | Summary of iVaww (mL) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used Footnote baseline | SAC |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.43. | All Subjects | PII116678/final/<br>Table 2.75 | Summary of iVaww (mL) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used | SAC |
| 2.44. | All Subjects | PII116678/final/<br>Table 2.76 | Summary of iVaww (mL) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.45. | All Subjects | PII116678/final/<br>Table 2.79 | Summary of siVaww (mL/L) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used | SAC |
| 2.46. | All Subjects | PII116678/final/<br>Table 2.80 | Summary of siVaww (mL/L) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.47. | All Subjects | PII116678/final/<br>Table 2.81 | Summary of siVaww (mL/L) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.48. | All Subjects | PII116678/final/<br>Table 2.82 | Summary of siVaww (mL/L) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.49. | All Subjects | PII116678/final/<br>Table 2.85 | Summary of Trachea Length (mm), Diameter (mm) and Length /Diameter (mm/mm) (Absolute) | Footnote any transformations used | SAC |
| 2.50. | All Subjects | PII116678/final/<br>Table 2.86 | Summary of Trachea Length (mm), Diameter (mm) and Length /Diameter (mm/mm) (Change from Baseline) | Footnote any transformations used Footnote baseline | SAC |
| 2.51. | All Subjects | PII116678/final/<br>Table 2.14 | Summary of Statistical Analysis for siVaw (mL/L), for Individual Lobes at FRC using Untrimmed Data | Ensure no overlapping information across pages for each Lobe Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.52. | All Subjects | PII116678/final/<br>Table 2.16 | Summary of Statistical Analysis for siVaw (mL/L), for Individual Regions at FRC using Untrimmed Data | Ensure no overlapping information across pages for each Lobe Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.53. | All Subjects | Refer to:<br>PII116678/final/<br>Table 2.16<br>Note: there will<br>be less regions | Summary of Statistical Analysis for siVaw (mL/L), for Distal Region at FRC using Scan Trimmed Data | Ensure no overlapping information across pages for each Lobe Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.54. | All Subjects | Refer to:<br>PII116678/final/<br>Table 2.29<br>Note: there will<br>be less regions | Summary of Statistical Analysis for siRaw (kPa*s), for Distal Region at FRC | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.55. | All Subjects | Refer to:<br>PII116678/final/<br>Table 2.54<br>Note: there will<br>be less regions | Summary of Statistical Analysis for LAS (% of iVlobe), for Total Region at TLC | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.56. | All Subjects | Refer to:<br>PII116678/final/<br>Table 2.60<br>Note: there will<br>be less regions | Summary of Statistical Analysis for IALD (%), for Upper and Lower Regions | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.57. | All Subjects | Refer to:<br>PII116678/final/<br>Table 2.66<br>Note: there will<br>be less regions | Summary of Statistical Analysis for AT (% of iVlobe), for Total Region at FRC | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.58. | All Subjects | Refer to:<br>PII116678/final/<br>Table 2.72<br>Note: there will<br>be less regions | Summary of Statistical Analysis for BVD (% of iVlobe), for Total Region at TLC | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.59. | All Subjects | Refer to: PII116678/final/ Table 2.84 Note: there will be less regions | Summary of Statistical Analysis for siVaww (mL/L), for Distal Region at TLC using Untrimmed Data | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| Lung F | unction | | | | |
| 2.60. | All Subjects | PII115119/<br>Part_A /Table<br>3.18 | Summary of FEV1 (L) and FVC (L) (Absolute Values) | Summaries by Visit<br>Footnote any transformations used | SAC |
| 2.61. | All Subjects | PII115119/<br>Part_A /Table<br>3.19 | Summary of FEV1 (L) and FVC (L) (Change from Baseline) | Summaries by Visit Footnote any transformations used Footnote Baseline | SAC |
| 2.62. | All Subjects | PII116678/ final<br>/Table 2.88 | Summary of Statistical Analysis for FEV1 (L) (Change from Baseline) | Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.63. | All Subjects | PII116678/<br>postcsr_2017_01<br>/Table 2.1 | Sub Group Analysis: by Index Exacerbation Severity<br>Summary of Statistical Analysis for FEV1 (L) (Change from<br>Baseline) | Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.64. | All Subjects | PII116678/ final<br>/Table 2.88 | Summary of Statistical Analysis for FVC (L) (Change from Baseline) | Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| Relief N | Medication | | | | |
| 2.65. | All Subjects | Refer to programming notes | Summary of Rescue Medication Free Days | Use the standard tu_sumstatsinrows to summarise Rescue Medication Free days by time period and treatment. Include columns for time period, treatment, N, n, mean, 95% CI, SD, median, min and max | SAC |
| 2.66. | All Subjects | Refer to programming notes | Summary of Mean Number of Occasions of Rescue Use per Day | Use the standard tu_sumstatsinrows to summarise Mean Number of Occasions of Rescue Use per Day by time period and treatment. Include columns for timeperiod, treatment, N, n, mean, 95% CI, SD, median, min and max | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Exacer | bations | | | | |
| 2.67. | All Subjects | Refer to PII116678/ final /Table 2.97 And programming notes | Summary of Investigator Defined Exacerbations | Update rows to be consistent with data i.e. include 6, 7, etc exacerbations as appropriate | SAC |
| 2.68. | All Subjects | Refer to PII116678/ final /Table 2.116 And programming notes | Summary of Investigator Reported Exacerbations<br>Requiring Concomitant Medication Treatment | Update rows to be consistent with data i.e. include 6, 7, etc exacerbations as appropriate | SAC |

# 13.10.5. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Lung F | unction | | | | |
| 2.1. | All Subjects | Refer to PII116678/final/ Table 2.2 but update the number of plots based on the data as appropriate | Summary of PEF (morning) | X-axis to contain each Day, with Means and confidence intervals, grouped by Treatment. Include baseline as a subheading per example shell | SAC |

# 13.10.6. Safety Tables

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Adverse Ev | ents (AEs) | | | | |
| 3.1. | All<br>Subjects | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.2. | All<br>Subjects | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | ICH E3 | SAC |
| 3.3. | All<br>Subjects | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3<br>Include flag for serious | SAC |
| 3.4. | All<br>Subjects | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT | SAC |
| Serious and | Other Signific | ant Adverse Ev | vents | | |
| 3.5. | All<br>Subjects | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC |
| 3.6. | All<br>Subjects | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | IDSL | SAC |
| Laboratory: | Chemistry | | | | |
| 3.7. | All<br>Subjects | LB1 | Summary of Chemistry | ICH E3 | SAC |

| Safety: Tabl | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.8. | All<br>Subjects | LB15 | Summary of Worst Case Emergent Laboratory Chemistry Results Post-Baseline Relative to Baseline | | SAC |
| Laboratory: | Hematology | | | - | |
| 3.9. | All<br>Subjects | LB1 | Summary of Hematology | ICH E3 | SAC |
| 3.10. | All<br>Subjects | LB15 | Summary of Worst Case Emergent Laboratory Hematology Results Post-Baseline Relative to Baseline | | SAC |
| Laboratory: | Hepatobiliary | (Liver) | | <u></u> | |
| 3.11. | All<br>Subjects | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC |
| 3.12. | All<br>Subjects | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC |
| ECG | | | | | |
| 3.13. | All<br>Subjects | EG1 | Summary of ECG Findings | IDSL | SAC |
| 3.14. | All<br>Subjects | EG2 | Summary of ECG Values by Visit | | SAC |
| 3.15. | All<br>Subjects | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC |
| Vital Signs | | | | | |
| 3.16. | All<br>Subjects | VS1 | Summary of Vital Signs | | SAC |

| Safety: Tabl | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.17. | All<br>Subjects | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3<br>Includes Baseline Values | SAC |
| 3.18. | All<br>Subjects | VS7 | Summary of Worst Case Vital Sign Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline | | SAC |

# 13.10.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Plasma | Concentration | n | | | • |
| 4.1. | PK | PK01<br>PII116678/final/Table<br>4.1 | Summary of Plasma Nemiralisib Pharmacokinetic Concentration – Time Data (ng/mL) | All visits/timepoints, include a column for visit. Summarise PK data on original scale. Produce 95% CIs Note: Use the separate NEMI Diskus and NEMI ELLIPTA treatment groups Excluding the two subjects who were noted to not comply with inhalation instructions – include | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.2. | PK | PK01<br>PII116678/final/Table<br>4.2 | Summary of Plasma Nemiralisib Pharmacokinetic Concentration – Time Data (ng/mL) Including All PK Concentrations Analysed | All visits/timepoints, include a column for visit. Summarise PK data on original scale. Produce 95% CIs Note: Use the separate NEMI Diskus and NEMI ELLIPTA treatment groups | SAC |
| | | | | Including the two subjects who were noted to not comply with inhalation instructions – include footnote | |
| | | | | All visits/timepoints, include a column for visit and planned time. Summarise PK data on original scale. Produce n, No. imputed, geometric mean and corresponding 95% Cis SD Logs and %CVb | |
| 4.3. | PK | PII116678/final/Table<br>4.3 | Summary of Log-Transformed Plasma Nemiralisib<br>Pharmacokinetic Concentration – Time Data (ng/mL) | Note: Use the separate NEMI<br>Diskus and NEMI ELLIPTA<br>treatment groups | SAC |
| | | | | Excluding the two subjects who were noted to not comply with inhalation instructions – include footnote | |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.4. | PK | PII116678/final/Table<br>4.4 | Summary of Log-Transformed Plasma Nemiralisib Pharmacokinetic Concentration – Time Data (ng/mL) Including All PK Concentrations Analysed | All visits/timepoints, include a column for visit and planned time. Summarise PK data on original scale. Produce n, No. imputed, geometric mean and corresponding 95% Cis SD Logs and %CVb Note: Use the separate NEMI Diskus and NEMI ELLIPTA treatment groups Including the two subjects who were noted to not comply with inhalation instructions – include footnote | SAC |

# 13.10.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Plasma | Concentration | ) | | | |
| 4.1. | PK | Refer to PII116678/ final/ Figure 4.1 But include additional timepoints per programming notes | Box and Whisker Plot of Plasma Concentration | Two figures to be created: 1st: Plasma Concentration at Day 1 (5 min and 24 hours post-dose) and Day 12 2nd: Plasma Concentration at Day 12, Day 28, Day 56 and Day 84 Note: Use the separate NEMI Diskus and NEMI ELLIPTA | SAC |

# 13.10.9. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| MRNa | | | | | |
| 6.1. | All Subjects | PII115119/<br>Part A/<br>Listing 40 | Summary of Statistical Analysis of mRNA Transcriptome in Induced Sputum (Selected Probe Sets Related to Neutrophil Function) | Summarise ratio, 95% CI and p-<br>values. Sort alphabetically on probe<br>set ID | SAC |
| 6.2. | All Subjects | PII115119/<br>Part A/<br>Listing 40 | Summary of Statistical Analysis of mRNA Transcriptome in Blood (All Probe Sets) | Biostatistics will await guidance following unblinded regarding which, if any, probe sets should be presented for the exploratory analysis and confirmation if a cut off criteria other than p-value<0.05 AND (fold change> 1.5 OR fold change< -1.5) should be used in determining which comparisons for the probe sets should be presented. Summarise ratio, 95% CI and p-values. | SAC |

| Pharma | acodynamic an | d Biomarker: Tab | es | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.3. | All Subjects | PII115119/<br>Part A/<br>Listing 40 | Summary of Additional Statistical Analysis of mRNA<br>Transcriptome in Induced Sputum (All Probe Sets) | Biostatistics will await guidance following unblinded regarding which, if any, probe sets should be presented for the exploratory analysis and confirmation if a cut off criteria other than p-value<0.05 AND (fold change> 1.5 OR fold change< -1.5) should be used in determining which comparisons for the probe sets should be presented. Summarise ratio, 95% CI and p-values. | SAC |
| Cell Co | unt Data and P | MN Differentials | | | |
| 6.4. | All Subjects | PII115119/<br>Part A/Table<br>5.7 | Summary Statistics (Absolute): Total Cell Count Data in Sputum by Treatment and Time. | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.5. | All Subjects | PII115119/<br>Part A/Table<br>5.8 | Summary Statistics (Change from Baseline): Total Cell Count Data in Sputum by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.6. | All Subjects | PII115119/<br>Part A/Table<br>5.9 | Summary Statistics (Absolute): PMNs Differentials in Sputum by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.7. | All Subjects | PII115119/<br>Part A/Table<br>5.10 | Summary Statistics (Change from Baseline): PMNs Differentials in Sputum by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.8. | All Subjects | PII115119/<br>Part A/Table<br>5.11 | Summary Statistics (Absolute): Total Cell Count Data in Blood by Treatment and Time. | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.9. | All Subjects | PII115119/<br>Part A/Table<br>5.12 | Summary Statistics (Change from Baseline): Total Cell Count Data in Blood by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.10. | All Subjects | PII115119/<br>Part A/Table<br>5.13 | Summary Statistics (Absolute): PMNs Differentials in Blood by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |

| Pharma | acodynamic an | d Biomarker: Tabl | es | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.11. | All Subjects | PII115119/<br>Part A/Table<br>5.14 | Summary Statistics (Change from Baseline): PMNs Differentials in Blood by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| Inflamn | natory Biomark | ers | | | |
| 6.12. | All Subjects | PII115119/<br>Part A/Table<br>5.17 | Summary Statistics (Absolute): Inflammatory Biomarkers by Treatment and Time | It is expected that no transformation will be required for this Table (6.12) and a log transformation will be required for Table 6.14. However appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.13. | All Subjects | PII115119/<br>Part A/Table<br>5.18 | Summary Statistics (Change from Baseline): Inflammatory Biomarkers by Treatment and Time | It is expected that no transformation will be required for this Table (6.13) and a log transformation will be required for Table 6.15. However appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |

| Pharma | acodynamic an | d Biomarker: Tabl | es | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.14. | All Subjects | PII115119/<br>Part A/Table<br>5.19 | Summary Statistics (Log-Transformed Absolute) Inflammatory Biomarkers by Treatment and Time | It is expected that no transformation will be required for Table 6.12 and a log transformation will be required for this Table (6.14). However appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.15. | All Subjects | PII115119/<br>Part A/Table<br>5.20 | Summary Statistics (Log-Transformed Change from Baseline) Inflammatory Biomarkers by Treatment and Time | It is expected that no transformation will be required for Table 6.13 and a log transformation will be required for this Table (6.15). However appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| Microb | iome (16S rRNA | A) and qPCR | | , | |
| 6.16. | All Subjects | PD4<br>and Refer to<br>programming<br>notes | Summary Statistics (Absolute): Microbiome (16S rRNA) Relative Abundance by Treatment and Time | If Data available Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |

| Pharma | acodynamic an | d Biomarker: Tabl | es | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.17. | All Subjects | PD4<br>and Refer to<br>programming<br>notes | Summary Statistics (Percentage Change from Baseline): Microbiome (16S rRNA) Relative Abundance by Treatment and Time | If Data available. Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.18. | All Subjects | PII115119/<br>Part A/Table<br>5.24 | Summary Statistics (Absolute): qPCR delta Ct by Treatment and Time | If Data available. Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.19. | All Subjects | PII115119/<br>Part A/Table<br>5.25 | Summary Statistics (Log-Transformed Absolute): qPCR fold change by Treatment and Time | If Data available. Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| Bacteri | al Culture | | | | |
| 6.20. | All Subjects | PII115119/<br>Part A/Table<br>5.26 | Frequency Table of Bacterial Culture (Presence) by Treatment and Time | | SAC |

# 13.10.10. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1. | APE | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | All Subjects | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | All Subjects | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 4. | All Subjects | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| 5. | All Subjects | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 6. | All Subjects | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | All Subjects | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 8. | APE | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | All Subjects | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 10. | All Subjects | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | All Subjects | CM3 | Listing of Concomitant Medications | IDSL | SAC |
| Expos | ure and Treatmo | ent Compliance | | | • |
| 12. | All Subjects | EX3 | Listing of Exposure Data | ICH E3 | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events | | | | |
| 13. | All Subjects | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| 14. | All Subjects | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 15. | All Subjects | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Serious | and Other Sig | nificant Adverse l | Events | | |
| 16. | All Subjects | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| 17. | All Subjects | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| 18. | All Subjects | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 19. | All Subjects | AE8 | Listing of Adverse Events Leading to Withdrawal from Study or<br>Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | |
| 20. | All Subjects | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 21. | All Subjects | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC |
| 22. | All Subjects | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC |
| 23. | All Subjects | LIVER7 | Listing of Liver Biopsy Details | | SAC |
| 24. | All Subjects | LIVER8 | Listing of Liver Imaging Details | | SAC |
| All Lab | oratory | | | | |
| 25. | All Subjects | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 26. | All Subjects | LB5 | Listing of Laboratory Values of Potential Clinical Importance | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 27. | All Subjects | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| ECG | | | | | |
| 28. | All Subjects | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 29. | All Subjects | EG3 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC |
| 30. | All Subjects | CP_EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |
| 31. | All Subjects | EG5 | Listing of Abnormal ECG Findings | IDSL | SAC |
| Vital Si | gns | | | | |
| 32. | All Subjects | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 33. | All Subjects | VS4 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC |

# 13.10.11. Non-ICH Listings

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Demog | raphy and Bas | eline Characteristi | cs | | |
| 34. | All Subjects | FH1 | Summary of Family History of Cardiovascular Risk Factors | | SAC |
| 35. | All Subjects | Refer to<br>Programming<br>notes | COPD Disease duration and Exacerbation Duration | Include investigator ID, subject ID, country, treatment group, COPD Disease Duration (in years and months) and Exacerbation History (number requiring oral/systemic corticosteroids and/or antibiotics and number requiring hospitalisation) as columns | SAC |
| 36. | All Subjects | PREG1a | Listing of Subjects Who Became Pregnant During the Study | Also indicate if the female partners of subjects became pregnant during the study | SAC |
| Labs | | | | | |
| 37. | All Subjects | LB13 | Listing of Laboratory Reference Ranges | | SAC |
| 38. | All Subjects | CP_LB5 | Listing of Laboratory Values Outside Normal Reference Range | | SAC |
| PK | | | | | |
| 39. | PK | PK07 | Listing of Individual Subjects Plasma Concentrations at all time points | | SAC |
| PD/Bio | markers | | | · · · | |
| 40. | All Subjects | PII115119/<br>Part A/Listing 25 | Listing of Sputum Collection | Include sample ID if available | SAC |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 41. | All Subjects | PII115119/<br>Part A/Listing 26 | Listing of Blood Collection for RNA | | SAC |
| 42. | All Subjects | PII115119/<br>Part A/Listing 31 | Listing of Cell Count Data | | SAC |
| 43. | All Subjects | PII115119/<br>Part A/Listing 32 | Listing of PMNs Differentials | | SAC |
| 44. | All Subjects | PII115119/<br>Part A/Listing 34 | Listing of Individual Subject Inflammatory Cytokine Biomarker Data | | SAC |
| 45. | All Subjects | PII115119/<br>Part A/Listing 35 | Listing of Microbiome (16S rRNA) Biomarker Data | | SAC |
| 46. | All Subjects | PII115119/<br>Part A/Listing 36 | Listing of qPCR Data | | SAC |
| 47. | All Subjects | PII115119/<br>Part A/Listing 37 | Listing of Bacterial Culture Data | | SAC |
| Compli | ance and Drug | Accountability | | | |
| 48. | All Subjects | Example Shell POP_L1 | Listing of Overall Compliance | Adaptation of IDSL Shell COMP2 | SAC |
| 49. | All Subjects | POP_L2 | Listing of Drug Accountability Data | Adaptation of IDSL Shell COMP3A | SAC |
| Patient | Profiles | | | | |
| 50. | All Subjects | CVEND1 | Patient Profile for Congestive Heart Failure | Listing for subject with Myocardial infarction/unstable angina | SAC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 51. | All Subjects | Refer to IDSL<br>Library<br>Arrythmias<br>Statistical<br>Display<br>Standards | Patient Profile for Arrythmias | Listing for subject with<br>Arrhythmias | SAC |
| 52. | All Subjects | Refer to IDSL Library Cerebrovascular Events, Stroke And Transient Ischemic Attack Statistical Display Standards | Patient Profile for Cerebrovascular Events, Stroke and Transient Ischemic Attack | Listing for subject with<br>Cerebrovascular events/stroke<br>and transient ischemic attack | SAC |

# 13.11. Appendix 11: Example Mock Shells for Data Displays

Available Upon Request
### The GlaxoSmithKline group of companies

201928

| Division | | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for Study 201928: A randomised, double-blind, placebo-controlled study to evaluate the safety, efficacy and changes in induced sputum and blood biomarkers following daily repeat doses of inhaled GSK2269557 for 12 weeks in adult subjects diagnosed with an acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD).

Compound Number : GSK2269557

Effective Date : 26-JUN-2018

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 201928.
- This RAP is intended to describe the pharmacodynamic/biomarker, safety, pharmacokinetic and efficacy analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

# RAP Author(s):

# Approver PPD Statistician (Clinical Statistics)

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

201928

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | 44 | |
| Study Accountable Person (Clinical Development) | 11-JUN-2018 | Email |
| PPD | 14-JUN-2018 | Email |
| Study Manager (Clinical Development) | 11,001, 2010 | Dilluii |
| Head (Respiratory HUB) | 20-JUN-2018 | Email |
| PPD PPD | | |
| Medical Director (Safety Lead) | 19-JUN-2018 | Email |
| PPD | 11 HD1 2010 | F11 |
| Data Quality Lead (Data Management) | 11-JUN-2018 | Email |
| PPD | 15 HIN 2010 | E |
| Clinical Pharmacokineticist (PK) | 15-JUN-2018 | Email |
| PPD | | |
| Director (Human Translational Models and Biomarkers) | 11-JUN-2018 | Email |
| PPD | | |
| Senior Director (Target Sciences Computational Biology) | 19-JUN-2018 | Email |
| PPD | 11 HDI 2010 | F11 |
| Principal Programmer (Clinical Programming) | 11-JUN-2018 | Email |

Notes:

[1] Approval of the gene list

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|--------------------------------|-------------|-----------------|
| PPD | 20 HIN 2019 | email |
| Director (Clinical Statistics) | 20-JUN-2018 | eman |
| PPD | 26-JUN-2018 | omoi1 |
| Manager (Clinical Programming) | 20-JUN-2018 | email |

201928

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRODUCTIO | ON | 6 |
| 2. | SLIMMARY OF | F KEY PROTOCOL INFORMATION | 6 |
| ۷. | | es to the Protocol Defined Statistical Analysis Plan | |
| | | Objective(s) and Endpoint(s) | |
| | | Design | |
| | | cal Analyses | |
| | 2.4.1. | | |
| 3. | PLANNED ANA | ALYSES | 11 |
| | 3.1. Final A | nalyses | 11 |
| 4. | | PULATIONS | |
| | 4.1. Protoco | ol Deviations | 11 |
| 5. | | IONS FOR DATA ANALYSES AND DATA HANDLING | 10 |
| | 5.1. Study T | Freatment & Sub-group Display Descriptors | ۱۵<br>12 |
| | | le Definitions | |
| | | nation of Covariates and Subgroups | |
| | 5.3.1 | Covariates and Other Strata | |
| | 5.3.1.<br>5.3.2. | Examination of Subgroups | |
| | | Considerations for Data Analyses and Data Handling | 10 |
| | Conver | ntions | 15 |
| 6. | CTUDY DODL | LATION ANALYSES | 16 |
| 0. | | ew of Planned Study Population Analyses | |
| 7. | | YNAMIC AND BIOMARKER ANALYSES | |
| | | Pharmacodynamic and Biomarker Analyses | |
| | 7.1.1. | | |
| | 7.1.2. | | |
| | 7.1.3. | | |
| | 7.1.4. | Statistical Analyses / Methods | |
| | | 7.1.4.1. Statistical Methodology Specification | |
| | 7.2. Explora | atory Pharmacodynamic and Biomarker Analyses | 19 |
| | 7.2.1. | Endpoint / Variables | 19 |
| | 7.2.2. | Summary Measure | |
| | 7.2.3. | Population of Interest | <mark>20</mark> |
| | 7.2.4. | Statistical Analyses / Methods | 21 |
| 8. | | IALYSES | |
| | | dary Efficacy Analyses (Not From HRCT Analyses) | |
| | 8.1.1. | Endpoint / Variables | |
| | 8.1.2. | Summary Measure | |
| | 8.1.3. | Population of Interest | |
| | 8.1.4. | Statistical Analyses / Methods | |
| | | 8.1.4.1. Statistical Methodology Specification | <mark>22</mark> |

| | | | | 201928 |
|---|---|---|---|---|
| | 8.2. | Seconda | ry Efficacy Analyses (From HRCT Analyses) | 24 |
| | | 8.2.1. | Endpoint / Variables | |
| | | 8.2.2. | Summary Measure | |
| | | 8.2.3. | Population of Interest | |
| | | 8.2.4. | Statistical Analyses / Methods | 28 |
| | 0.0 | | 8.2.4.1. Statistical Methodology Specification | 28 |
| • | 8.3. | | ory Efficacy Analyses (From HRCT Analyses) | |
| | | 8.3.1.<br>8.3.2. | Endpoint / Variables | |
| | | 8.3.2.<br>8.3.3. | Summary Measure | |
| | | 6.3.3.<br>8.3.4. | Population of Interest | |
| | | 0.3.4. | 8.3.4.1. Statistical Methodology Specification | |
| | 8.4. | Evolorato | ory Efficacy Analyses (Not from HRCT Analyses) | |
| | 0.4. | 8.4.1. | Endpoint / Variables | |
| | | 8.4.2. | Summary Measure | |
| | | 8.4.3. | Population of Interest | |
| | | 8.4.4. | Statistical Analyses / Methods | |
| | | 0.4.4. | Oldibliodi / Widiyooo / Widiiodo | |
| 9. | RELAT | IONSHIP | BETWEEN THE PHARMACODYNAMIC AND | |
| | | | ATA AND THE HRCT DATA | 36 |
| | 9.1. | | ship between the mRNA data and the HRCT data | |
| | | | • | |
| | | | 'SES | |
| | 10.1. | | Events Analyses | |
| | 10.2. | | aboratory Analyses | |
| | 10.3. | Other Sa | fety Analyses | 37 |
| | | | IETIO ANALYOFO | |
| | | | IETIC ANALYSES | |
| | 11.1. | | ry Pharmacokinetic Analyses | |
| | | 11.1.1. | Endpoint / Variables | 38 |
| | | | 11.1.1.1. Drug Concentration Measures | |
| | | 44.4.0 | 11.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 11.1.2. | Summary Measure | |
| | | 11.1.3. | Population of Interest | 38 |
| 10 | DEEE | DENICES | | 20 |
| 12. | KEFE | KENCES. | | 39 |
| 13 | APPEN | IDICES | | 40 |
| 10. | 7.1. L.<br>13.1 | Annendix | 1: Protocol Deviation Management | 40 |
| | 10.1. | 13.1.1. | Important Protocol Deviations | 40 |
| | 13.2. | | c 2: Schedule of Activities | |
| | | 13.2.1. | Protocol Defined Schedule of Events | |
| | 13.3. | | 3: Assessment Windows | |
| | | 13.3.1. | Definitions of Assessment Windows for Analyses | |
| | 13.4. | | 4: Study Phases and Treatment Emergent Adverse | |
| | | Events | | 46 |
| | | 13.4.1. | Study Phases | |
| | | | 13.4.1.1. Study Phases for Concomitant Medication | |
| | | 13.4.2. | Treatment States for Adverse Events | 46 |
| | 13.5. | Appendix | c 5: Data Display Standards & Handling Conventions | |
| | | 13.5.1. | Reporting Process | |
| | | 13.5.2. | Reporting Standards | |

| | | | 201928 |
|--------|----------|-------------------------------------------------|--------|
| | 13.5.3. | Reporting Standards for Pharmacokinetic | 48 |
| 13.6. | Appendix | x 6: Derived and Transformed Data | |
| | 13.6.1. | General | |
| | 13.6.2. | Study Population | |
| | 13.6.3. | Efficacy | |
| | 13.6.4. | Safety | 52 |
| | 13.6.5. | Pharmacodynamic and Biomarker | 52 |
| 13.7. | Appendix | x 7: Reporting Standards for Missing Data | |
| | 13.7.1. | Premature Withdrawals | |
| | 13.7.2. | Handling of Missing Data | |
| | | 13.7.2.1. Handling of Missing and Partial Dates | 65 |
| 13.8. | Appendix | x 8: Values of Potential Clinical Importance | 66 |
| | 13.8.1. | Laboratory Values | 66 |
| | 13.8.2. | ECG | 67 |
| | 13.8.3. | Vital Signs | 67 |
| 13.9. | Appendix | x 9: Abbreviations & Trade Marks | 68 |
| | 13.9.1. | Abbreviations | 68 |
| | 13.9.2. | Trademarks | 70 |
| 13.10. | Appendix | k 10: List of Data Displays | 71 |
| | 13.10.1. | Data Display Numbering | 71 |
| | 13.10.2. | Deliverables | 71 |
| | 13.10.3. | Study Population Tables | 72 |
| | 13.10.4. | Efficacy Tables | 74 |
| | 13.10.5. | Efficacy Figures | 92 |
| | 13.10.6. | Safety Tables | 93 |
| | 13.10.7. | Pharmacokinetic Tables | 95 |
| | | Pharmacokinetic Figures | |
| | 13.10.9. | Pharmacodynamic and Biomarker Tables | 99 |
| | 13.10.10 | .ICH Listings | 104 |
| | 13.10.11 | Non-ICH Listings | 107 |

201928

#### 1. **INTRODUCTION**

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| GlaxoSmithKline Document Number | Date | Version |
| 2014N218070_00 | 2015-JUN-04 | Original |
| 2014N218070_01 | 2015-NOV-30 | Amendment No. 1 |
| Remove the specific equations for the predictio | n of percent predicted from spire | ometry |
| from the inclusion criteria and in Section 7.7.2. | At screening it may not be poss | ible to |
| identify which correction method was used, or r | nodify the correction method us | ed, at the |
| time. It therefore is not valid to stipulate that lun | g function values be corrected | using any |
| particular method. Both FEV <sub>1</sub> and FVC measur | ements (which are not entry crit | eria for |
| the study) collected during the study will be coll | ected as absolute values (unco | rrected), so |
| that consistency will be obtained across all sites | s in the study, and percent pred | icted will |
| be calculated using a standard approach in hou | se at the end of the study. | |
| 2014N218070_02 | 2016-JAN-26 | Amendment No. 2 |
| Increase the body mass index (BMI) range in the inclusion criteria from 18-32 kg/m <sup>2</sup> | | |
| (inclusive) to 16-35 kg/m <sup>2</sup> (inclusive). The origi | nal BMI range from 18-32 kg/m² | is a |
| typical range used in both healthy volunteer stu | dies and general subject popula | ations. The |
| revised range is more appropriate for a COPD | patient population. | |
| 2014N218070_03 | | |
| To remove photo toxicity from the protocol and | to include minor administrative | and |
| clarification changes. | | |
| 2014N218070_04 | 2017-MAR-2 | Amendment No. 4 |
| Replace the administration of GSK2269557 via the DISKUS™ device (1000 µg) by a | | |
| comparable dose administered via the ELLIPTA™ device (700 µg). GSK2269557 is no | | |
| longer manufactured for use with the DISKUS device which will be replaced with | | |

ELLIPTA Device. To increase the number of patients to be recruited to obtain sufficient completers. Minor updates and clarifications.

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

#### **Changes to the Protocol Defined Statistical Analysis Plan** 2.1.

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

201928

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Total lung capacity and lung lobar<br>volumes included in HRCT<br>secondary endpoint parameters | Total lung capacity and lung lobar<br>volumes dropped from HRCT<br>secondary endpoint parameters<br>included as an exploratory<br>endpoint parameter instead | The clinically relevant HRCT parameters are still to be decided. However, there was no clinical benefit seen in the comparison between GSK2269557 1000 mcg and Placebo in these parameters. |
| Analysis population: All Subject All randomised subjects who receive at least one dose of the study treatment. This population will be based on the treatment the subject actually received. Pharmacokinetic Subjects in the 'All subject' population for whom a pharmacokinetic sample was obtained and analysed. | Analysis population: All Subject All randomised subjects who receive at least one dose of the study treatment. This population will be based on the treatment the subject actually received. Pharmacokinetic Subjects in the 'All subject' population for whom a pharmacokinetic sample was obtained and analysed. Note: The two subjects who were not compliant with inhaler instructions will be excluded from the outcome summaries if they received active treatment but will be included if they received placebo | 2 subjects were not compliant with inhaler instructions and may not have received the full dose in amendment 4. Therefore, these subjects will be excluded from the outcome summaries if they received active treatment but will be included if they received placebo. Sensitivity analyses may be conducted including these subjects. |

# 2.2. Study Objective(s) and Endpoint(s)

| Ob | Objectives | | dpoints |
|---|---|---|---|
| Pri | Primary Objectives | | mary Endpoints |
| <ul> <li>To establish the PI3Kδ-dependent<br/>changes in previously identified immune<br/>cell mechanisms specifically related to<br/>neutrophil function using mRNA in sputum<br/>from patients with an exacerbation of<br/>COPD, with or without treatment with<br/>GSK2269557.</li> </ul> | | • | Alterations in previously identified immune cell mechanisms specifically related to neutrophil function as determined by changes in mRNA transcriptomics in induced sputum after 12, 28 and 84 days of treatment. |
| Sec | condary Objectives | Sec | condary Endpoints |
| • | To evaluate the effect of once daily repeat inhaled doses of GSK2269557 on lung parameters derived from HRCT scans in subjects with acute exacerbation of COPD, compared to placebo. | • | Change from baseline in siVaw, iVaw, iRaw, siRaw, total lung capacity, lung lobar volumes, trachea length and diameter at FRC and TLC after 12 days of treatment and after 28 days of treatment. |
| • | To assess the safety and tolerability of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. | • | Adverse events Haematology, clinical chemistry Vital signs 12-lead ECG |

201928

| Objectives | Endpoints |
|---|---|
| To evaluate the plasma PK of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD. To evaluate the effect of once daily repeat | <ul> <li>Day 1 plasma Cmax and trough (24 hours) post dose for inpatients.</li> <li>Trough concentration after 12 days, 28 days, 56 days and 84 days of treatment.</li> <li>To evaluate the effect of once daily repeat inhaled doses of</li> </ul> |
| inhaled doses of GSK2269557 on lung function parameters in subjects with acute exacerbation of COPD compared to placebo. | GSK2269557 on lung function parameters in subjects with acute exacerbation of COPD compared to placebo. |
| Exploratory Objectives | Exploratory Endpoints |
| <ul> <li>To establish any other PI3Kδ-dependent changes in mRNA in sputum or blood from patients with an exacerbation of COPD, with or without treatment with GSK2269557.</li> <li>To explore the pharmacodynamic effects in induced sputum of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo.</li> </ul> | <ul> <li>To establish any other PI3Kδ-dependent changes in mRNA in sputum or blood from patients with an exacerbation of COPD, with or without treatment with GSK2269557.</li> <li>To explore the pharmacodynamic effects in induced sputum of once daily repeat inhaled doses of GSK2269557 qPCR.</li> </ul> |
| To assess the changes in other CT parameters such as low attenuation score after once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. | Change from baseline for other CT parameters including low attenuation score after 12 days of treatment and after 28 days of treatment |

201928

# 2.3. Study Design



# 2.4. Statistical Analyses

# 2.4.1. Primary Analyses

To estimate differences in mRNA intensities within and between treatment groups, a repeated measures model will be fitted to the results of the analysis of each probe set at

201928

Day 12, Day 28 and Day 84 following a loge transformation of the data. The Day 1 response will be fitted as a baseline covariate.

Back transformed ratios versus screening along with 95% confidence intervals will be calculated for each treatment group and timepoint. Additionally, baseline adjusted ratios of the change between active treatment and placebo will be calculated along with 95% confidence intervals.

Further details are provided in Section 7.1.

201928

# 3. PLANNED ANALYSES

# 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Participants<br>Enrolled (APE) | All subjects who were screened for eligibility | Study Population |
| All Subject | Comprised of all subjects who were randomised. This population will be based on the treatment the subject actually received. If participants receive >1 treatment, then they will be summarised according to the most frequently dosed treatment. In cases where the frequency is equal, the participant will be assigned the lowest dose strength of nemiralisib. If participants receive no treatment, then they will be summarised according to "No Treatment" | <ul> <li>Study Population</li> <li>Pharmacodynamics<br/>and Biomarker</li> <li>Safety</li> <li>Efficacy</li> </ul> |
| Pharmacokinetic (PK) | Subjects in the 'All Subject' population for whom a pharmacokinetic sample was obtained and analysed. | • PK |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

Note: The two subjects who were not compliant with inhaler instructions will be excluded from the outcome summaries if they received active treatment but will be included if they received placebo

#### 4.1. Protocol Deviations

During the course of the study it was noted that two subjects did not complete dosing instructions as required. The primary plan is if the subjects received active treatment they will be excluded from the study outcome summaries; if the subject received placebo treatment, they will be included in the study outcome summaries. It has not yet been identified if they received placebo or active treatment. A footnote will be applied to all relevant displays stating the rationale, subject number, treatment and if they were excluded, e.g. "Subjects X & Y did not complete dosing instructions as required; subject X received nemiralisib and was therefore excluded, subject Y received placebo and was therefore included." The footnote may be tweaked for aesthetic purposes.

201928

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan, refer to Appendix 1.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

201928

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order in TLF |
| This will be derived as subjects who did not receive any treatment | | No Treatment | 1 |
| This will b | pe derived as subjects in RandALL<br>or C | All Placebo | 2 |
| This will be derived as subjects in RandALL codes B or D | | All NEMI | 3 |
| Α | Placebo | Placebo Diskus | 4 |
| B GSK2269557 1000 mcg | | NEMI Diskus | 5 |
| С | Placebo via Ellipta | Placebo Ellipta | 6 |
| D GSK2269557 700 mcg | | NEMI Ellipta | 7 |

#### NOTES:

- The following footnote will be presented on displays which use the "Placebo Diskus", "NEMI Diskus", "Placebo Ellipta" or "NEMI Ellipta" treatment groups:
  - NEMI Diskus = 1000 mcg Nemiralisib administered via the Diskus device; NEMI Ellipta =700 mcg Nemiralisib administered via the Ellipta device
- 2. Order represents treatments being presented in TFL, as appropriate

Treatment groups "Placebo" and "Placebo via Ellipta" (RandAll NG codes A and C) will be combined into "All Placebo" treatment group. Similarly, treatment groups "GSK2269557 700 mcg" and "GSK2269557 1000 mcg" (RandAll NG codes B and D) will be combined into "All NEMI" treatment group.

Treatment comparisons will be displayed as follows using the descriptors as specified:

#### 1. All NEMI vs All Placebo

#### Notes:

- The "All Placebo" and "All NEMI" groups and "All NEMI vs All Placebo" treatment comparison will be presented for Pharmacodynamic and biomarker, efficacy and study population summaries unless otherwise specified.
- The "Placebo Diskus", "NEMI Diskus", "Placebo Ellipta" or "NEMI Ellipta" treatment groups will be presented for Pharmacokinetic and safety summaries unless otherwise specified.
- The "Placebo Diskus", "NEMI Diskus", "Placebo Ellipta" or "NEMI Ellipta" treatment groups will be presented for all listings

201928

# 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | S | tudy Assessmer | nts Considered as Bas | Baseline | |
|---|---|---|---|---|---|
| | Screening | Day 1<br>(Pre-<br>Treatment) | Day 2<br>Within<br>48H/discharge<br>(On Treatment) | Day 12<br>(On<br>Treatment) | Used in Data<br>Display |
| Safety | | | | | |
| Labs including<br>Haematology | X | X | | | Day 1 |
| ECG | X | Χ | | | Day 1 |
| Vitals | Х | Χ | | | Day 1 |
| Efficacy | | | | | |
| HRCT Untrimmed | Х | | | | Screening |
| HRCT Scan<br>Trimmed | | | | | |
| Screening&Day12 | Х | | | | Screening |
| Screening&Day28 | Х | | | | Screening |
| Day12&Day28 | | | | Х | Day 12 |
| FEV₁ and FVC | | Χ | Χ | | Day 1 <sup>[1]</sup> |
| Daily PEF [2] | | Х | | | Day 1 |
| | | | | | Mean of Days<br>1 to 3 |
| | | | | | Maximum of Days 1 to 3 |
| Pharmacodynamic | | | | | |
| Sputum and Blood | Х | | | | Screening |
| Genetic sample (PGx) [3] | | | Х | | |

# NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- [1] Baseline will be investigated to ensure there is sufficient data and will be footnoted as appropriate
- [2] For PEF 3 different baselines will be calculated: Day 1, mean of Days 1 to 3 and Maximum of Days 1 to 3. TFLs will be footnoted with the relevant baseline.
- [3] Collected at any time after randomisation

201928

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Examination of Covariates and Subgroups

#### 5.3.1. Covariates and Other Strata

The list of covariates may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates of clinical interest may also be considered.

| Category | Details |
|------------|-------------------------------------------------------|
| Covariates | Age, Sex, BMI, Country, Primary exacerbation severity |

# 5.3.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories |
|-------------------------------|------------------------|
| Primary exacerbation severity | Moderate or Severe [1] |
| Country | Country |

#### NOTES:

[1] Exacerbations are defined as severe if they require hospitalisation, otherwise they are defined as moderate

# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 13.3 | Appendix 3: Assessment Windows |
| 13.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 13.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 13.6 | Appendix 6: Derived and Transformed Data |
| 13.7 | Appendix 7: Reporting Standards for Missing Data |
| 13.8 | Appendix 8: Values of Potential Clinical Importance |

201928

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "All Subject" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

201928

# 7. PHARMACODYNAMIC AND BIOMARKER ANALYSES

# 7.1. Primary Pharmacodynamic and Biomarker Analyses

# 7.1.1. Endpoint / Variables

Sputum RNA will be extracted and hybridised using a balanced batch design. An appropriate microarray platform will be determined at the time of hybridisation, to allow for improvements in technology. The quality of the data will be assessed and then normalised using appropriate methodologies and software.

Microarray mRNA data will be normalised using gcRMA or RMA in Array Studio v5.0 or later. After normalisation, the data will be quality assessed and any samples deemed as QC fails will be excluded from any further analysis. This quality assessment will involve looking for outlying signals in both the normalised expression data and the MAS5 QC metrics generated from each sample. If any samples are excluded, the remaining data will be re-normalised. The output from the normalisation will be log2 transformed mRNA intensity data (measured in arbitrary units).

Since the data will be log2 transformed prior to the analysis the treatment effects will be expressed as ratios after back transformation (2<sup>^</sup>). These ratios can be converted from treatment ratios to fold change values as follows:

- If ratio ≥ 0 then fold change = ratio
- If ratio <0 then fold change = -1/ratio

Microarray data consists of expression values (log2-transformed) derived from individual probe sets designed against coding regions of individual genes. More than one probe set can exist per gene. This analysis will be conducted at the probe set level.

The mRNA data gives results from  $\sim 14000$  genes encoded by  $\sim 54000$  probe sets. To establish the PI3K $\delta$ -dependent changes in previously identified immune cell mechanisms specifically related to neutrophil function using mRNA, we identified 258 gene to subset our data on, refer to Section 13.6.5. The gene names were converted to Affymetrix probe IDs, this resulted in 638 probes refer to Section 13.6.5.

To compare the expression value between treatments for each probe set, linear repeated measures mixed effects model will be fitted to each probe set, with log2 (intensity) as the response variable. Note: log2 (intensity) may also be referred to as mRNA intensities (logarithm base 2 scale). Alteration in previously identified immune cell mechanisms specifically related to neutrophil function will be determined by changes in mRNA transcriptomics in induced sputum after 12, 28 and 84 days of treatment by the analysis of mRNA intensities (logarithm base 2 scale) subset by the 638 probes identified in Section 13.6.5.

201928

# 7.1.2. Summary Measure

A repeated measures modelling analysis will be performed on the subset of 638 probes which have previously identified immune cell mechanisms specifically related to neutrophil function.

The model will be used to estimate the baseline adjusted fold changes for active treatment and placebo calculated for Day 12, Day 28 and Day 84 along with the corresponding 95% confidence intervals and unadjusted P-values. Additionally, baseline adjusted ratios of the change between active treatment and placebo will be calculated along with 95% confidence intervals and unadjusted P-values.

# 7.1.3. Population of Interest

The primary pharmacodynamic analyses will be based on the "All Subject" population, unless otherwise specified.

# 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 7.1.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

 Alterations in the previously identified immune cell mechanisms specifically related to neutrophil function as determined by changes in mRNA transcriptomics in induced sputum after 12, 28 and 84 days of treatment. The response variable will be mRNA intensities (logarithm base 2 scale).

#### **Model Specification**

The mRNA data gives results from ~14000 genes encoded by ~54000 probe sets. A subset of 638 probe sets specifically relating to the cell mechanisms of neutrophil function is specified in Section 13.6.5 This subset will comprise the primary statistical analysis dataset.

The repeated measures modeling analysis will be performed for each probe set separately.

To estimate differences in mRNA intensities between treatment groups, a repeated measures model will be fitted to mRNA intensities at Screening, Day 12, Day 28 and Day 84. The Screening time point will be considered Baseline. The model will include terms for treatment group (All Placebo or All NEMI), time and a treatment group by time interaction. An unstructured (UN) covariance structure will be fitted, however, in the event that this structure results in a model failing to converge then attempts will be made to fit a model that converges i.e. alternative covariance structures may be considered. The denominator degrees of freedom for use in significance testing

201928

will be computed using the Kenward Rogers approximation.

Back transformed baseline-adjusted means along with 95% CIs will be calculated for each treatment group and time-point. Additionally, baseline adjusted fold changes between All NEMI and All Placebo will be calculated for Day 12, Day 28 and Day 84 as well as the ratio between the baseline adjusted fold changes for All NEMI vs. All Placebo at day 12, 28 and 84, along with 95% CI and two-sided unadjusted p-values. Additionally, the fold change between All NEMI vs. All Placebo at day 84 may be investigate along with 95% CI and two-sided unadjusted p-values and other comparisons of interest.

To enable review by the study team a spreadsheet will be created containing the output for all probe sets in scope for the primary statistical analysis will be generated and ranked by p-value for the comparison All NEMI vs. All Placebo at day 12, 28 and 84 in separate tabs. A separate spreadsheet will be created containing only probe sets where the p-value for the comparison All NEMI vs. All Placebo is <0.05, with day 12, 28 and 84 in separate tabs. Such probe sets will be ranked by fold change, with the expectation that, in general, a greater than a 1.5-fold change is scientifically meaningful. To comply with guidance regarding QC, each tab will be stored as a SAS dataset to ensure QC can be audited.

Following review by the study team of the results, a subset of probe sets will be identified and may be used for further reporting.

# **Model Checking & Diagnostics**

- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - In the event that this model fails to converge, alternative correlation structures may be considered

#### **Model Results Presentation**

The subset of probe sets where the p-value for the comparison All NEMI vs. All Placebo at day 12, 28 and 84, is <0.05 will be reported as described below:

Output from the repeated measures modelling detailed above will be tabulated. In particular, the estimated baseline adjusted fold changes, 95% CI, standard error (on the logarithm base 2 scale), unadjusted p-values at each time point and for the active treatment comparison with placebo. The probe set, gene/gene description will be included in the outputs.

# 7.2. Exploratory Pharmacodynamic and Biomarker Analyses

# 7.2.1. Endpoint / Variables

In addition to the primary analysis, there is an exploratory objective to establish any other PI3K $\delta$ -dependent changes in mRNA in sputum or blood from patients with an exacerbation of COPD, with or without treatment with GSK2269557. To address this blood and sputum mRNA data, as described in Section 7.1, but analyses will be conducted

201928

on the complete mRNA data, i.e. the results from  $\sim$ 14000 genes encoded by  $\sim$ 54000 probe sets.

To explore the pharmacodynamic effects in induced sputum of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. Endpoints may include, but not limited to, cytokines (IL-6, IL-8, TNFα), microbiome (by 16SrRNA), bacterial qPCR, total cell counts and PMNs differentials.

To explore the pharmacodynamic effects in blood of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. Endpoints may include, but not limited to, total cell counts and PMNs differentials

# 7.2.2. Summary Measure

To establish any other PI3K $\delta$ -dependent changes in mRNA in sputum or blood from patients with an exacerbation of COPD, with or without treatment with GSK2269557. A repeated measures modelling analysis will be performed on the complete probe set. The model will be used to estimate the baseline adjusted fold changes for active treatment and placebo calculated for Day 12, Day 28 and Day 84 along with the corresponding 95% confidence intervals and unadjusted P-values. Additionally, baseline adjusted ratios of the change between active treatment and placebo will be calculated along with 95% confidence intervals and unadjusted P-values.

To explore the pharmacodynamic effects in induced sputum of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. Summary statistics of endpoints may include, but not limited to, cytokines (IL-6, IL-8, TNFα), microbiome (by 16SrRNA), bacterial qPCR, total cell counts and PMNs differentials.

To explore the pharmacodynamic effects in blood of once daily repeat inhaled doses of GSK2269557 administered to subjects with acute exacerbation of COPD, compared to placebo. Summary statistics of endpoints may include, but not limited to, total cell counts and PMNs differentials.

#### 7.2.3. Population of Interest

The exploratory pharmacodynamic analyses will be based on the "All Subjects" population, unless otherwise specified.

As previously discussed for the two subjects that did not follow inhalation instructions, if the subjects received active treatment they will be excluded from the study outcome summaries; if the subject received placebo treatment, they will be included in the study outcome summaries.

201928

# 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Refer to Section 7.1.4.1 for statistical methodology specification, however, for the exploratory analysis, the models will be fitted but on the complete dataset ~14000 genes encoded by ~54000 probe sets; sputum and blood data will be analysed separately.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed. For each endpoint, the values will be inspected to determine whether a data transformation is required. It is expected that: cytokines may require a transformed on the natural logarithm scale

201928

# 8. EFFICACY ANALYSES

# 8.1. Secondary Efficacy Analyses (Not From HRCT Analyses)

# 8.1.1. Endpoint / Variables

To evaluate the effect of once daily repeat inhaled doses of nemiralisib on lung function parameters in subjects with acute exacerbation of COPD compared to placebo. Lung function parameters including:

- PEF
- FEV<sub>1</sub> and FVC at clinic prior to sputum induction
- reliever usage

# 8.1.2. Summary Measure

For PEF, summary statistics for the change from baseline PEF will be presented in tabular form, mean and 95% CIs of AM PEF readings will be plotted by study treatment vs. Study Day.

For FEV<sub>1</sub> (mL) and FVC (mL), a change from baseline statistical analysis will be conducted and presented via tables of predicted adjusted medians for each Treatment arm at each visit, and the difference between treatment arms at each visit.

For reliever use, bronchodilator use recorded in the diary will be summarised as the mean number of occasions of rescue use per day and the percentage of rescue-free days in four-week interval periods as described in Section 13.6.3, where a rescue-free day is defined as a 24-hour period in which the number of occasions bronchodilator taken is zero. Summary tables will display estimates for each 4-weekly period for mean number of occasions of rescue use per day and percentage of rescue-free days separately.

# 8.1.3. Population of Interest

The primary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

# 8.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8.1.4.1. Statistical Methodology Specification

NOTE: The description below describes the current thinking of how to analyse these endpoints. The proposed models will be assessed, and if not appropriate alternative models could be used.

201928

#### **Endpoint / Variables**

FEV1 (ml), FVC(ml)

# **Model Specification**

- The data will be inspected during statistical analysis to determine whether a data transformation is required. It is likely no transformations will be required
- The analysis will include all available values. If there are values which were recorded within 4h
  after the subject had taken relief medication, a sensitivity analysis may be done which excludes
  these values.
- The endpoints (FEV<sub>1</sub> and FVC) will be analysed in separate models. The change from baseline in the endpoint will be analysed in a Bayesian repeated measures model, with a baseline by Visit covariate and Treatment by Visit class parameter. Note that the model will not include an intercept. The Treatment will have two levels: All NEMI and All Placebo, and the Visit will have two levels: Day 28 and Day 84. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e. covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The change from baseline at each of the Visits will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in a tabular format.
- The difference between the treatment arms, for the change from baseline will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular format.
- The probabilities that the treatment difference is greater or less than 0 (depending on direction
  of the endpoint), in addition to other values appropriately selected based on the data, will also
  be computed for each Visit. These results will be presented in tabular format.

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data. For example, if data do not approximately follow a normal distribution then attempt will be made to find a suitable transformation.
- A comprehensive investigation into a suitable model should be initiated. For example, additional covariates will be investigated
- An unstructured covariance structure will be used. However, in the event that this model fails to converge, alternative correlation structures may be considered.
- Models with a Bayesian Framework will use vague priors. If appropriate, conjugate priors will be used. For example, for a multivariate model, the prior for the variance covariance matrix will be an inverse Wishart distribution.

#### **Model Results Presentation**

 Output from the repeated measures modelling detailed above will be tabulated. In particular, the estimated change from baseline, 95% CI, standard error, and posterior probabilities at each time point and for the active treatment comparison with placebo.

201928

# **Subgroup Analyses**

- For FEV1, a subgroup analysis will be conducted by index exacerbation severity (refer to Section 5.3 Examination of Covariates and Subgroups). A similar model as described in Model specification will be fitted but will also include a Severity\*Treatment\*Visit term within the model.
- The results of the subgroup analysis will be reported in a separate table.

# 8.2. Secondary Efficacy Analyses (From HRCT Analyses)

# 8.2.1. Endpoint / Variables

To evaluate the effect of once daily repeat inhaled doses of nemiralisib on lung parameters derived from HRCT scans in subjects with acute exacerbation of COPD, compared to placebo. Ratio from baseline in siVaw, iVaw, iRaw, siRaw, trachea length and diameter at FRC and TLC after 12 days of treatment and after 28 days of treatment.

# 8.2.2. Summary Measure

Each HRCT scan will be conducted at two lung volumes: total lung capacity (TLC) and functional residual capacity (FRC); these will be referred to as scan conditions. The HRCT images will be processed to derive the HRCT parameters at FRC and TLC, however these conditions are not applicable for all parameters.

The HRCT scans will be conducted at Screening, Day 12 and Day 28. The 3 HRCT images will then be processed to derive the HRCT parameters at each scan; this data will be referred to as the untrimmed data. The untrimmed data measures all airways that are present in each scan.

However partially due to positioning of subjects whilst taking a scan, it can be that some airways are visible in some scans and not in other scans. For these reasons, some HRCT imaging endpoints will be calculated to include only airways that are visible in both scans. Therefore, the scans were grouped into three scan trimming pairs where, within each scan trimming pair, the airways that were not present in both scans were removed/trimmed.

The three scan trimming pairs, and subsequent timepoints, are:

- The scan trimming pair SCRD28, which contains the Screening (SCRD28:SCR) and Day 28 (SCRD28:D28) timepoints, where only airways that were present in both screening and day 28 scans are accounted for.
- The scan trimming pair SCRD12, which contains the Screening (SCRD12:SCR) and Day 12 (SCRD12:D12) timepoints where only airways that were present in both screening and day 12 scan are accounted for.
- The scan trimming pair (D12D28), which contains the Day 12 (D12D28:D12) and Day 28 (D12D28:D28) timepoints, where only airways that were present in both day 12 and day 28 scans are accounted for.

These 6 HRCT images were then processed to derive the HRCT parameters at each of these scan-trimming pair time points; this data will be referred to as the scan trimmed

201928

data. The scan trimmed data considers only airways that were present in both scans within the scan trimming pair. This ensures the airway models are the same length although the cross-sectional area of the airway may vary. For example, the schematic below shows visible airways on Screening alone and Day 12 alone. It then shows the airways that are visible on both Screening & Day 12 scans, through removing/trimming airways that are not present in both scans.



The HRCT scans can identify the 5 different lobes of the lungs and these lobes can then be categorized into and up to 5 regions depending on the endpoint. The 5 lobes are Right Upper Lobe (RUL), Left Upper Lobe (LUL), Right Middle Lobe (RML), Right Lower Lobe (RLL) and Left Lower Lobe (LLL). The 5 regions are Upper (comprising of RUL, RML and LUL), Lower (comprising of RLL and LLL), Central (the main bronchi between the lobes and the trachea), Distal (comprising of Upper and Lower) and Total (comprising of Distal and Central).

The endpoints for which the 5 regions apply include:

- Specific imaging airway volume (siVaw)
- Imaging airway volume (iVaw)
- Specific imaging airway resistance (siRaw)
- Imaging airway resistance (iRaw)
- Specific imaging airway wall volume (siVaww)
- Imaging airway wall volume (iVaww)

The endpoints for which only 3 regions (upper, lower & total) apply include:

- Imaging lobe volume (iVlobe)
- Percent predicted lobar volume (iVlobepred)
- Low attenuation score (LAS)
- Air trapping score (AT)
- Blood vessel density (BVD)

The endpoint for which only 2 regions (upper & lower) apply is:

• Internal airflow lobar distribution (IALD)

For the measures iVaw, iRaw and iVaww, standardization within a subject for the size of the lobar volume was conducted. These specific measures can be adjusted for the individual's lobar volume by correcting for the corresponding lobe/region. Note the central region is not applicable for lobar volumes, instead the corresponding region for the central, distal and total regions is the total lobar volume region. For example:

 To calculate siVaw, the lobes/regions of iVaw being divided by the corresponding lobes/regions of iVlobe to calculate the lobes/regions of siVaw, thus siVaw can be

201928

defined as a measure of volume in an individual's airways, corrected for the individual's lobar volume.

- To calculate siRaw, the lobes/regions of iRaw were multiplied by the corresponding lobes/regions of iVlobe.
- To calculate siVaww, the lobes/regions of iVaww were divided by the corresponding lobes/regions of iVlobe.

For such reasons, the table below shows the HRCT endpoints and the results that will be captured:

Table 2 HRCT Endpoints (and results that will be captured)

| | | Untrimmed | | Scan Trimming, based on: | | | |
|---|---|---|---|---|---|---|---|
| Endpoints | Units | Screening | Day<br>12 | Day 28 | Screening<br>and Day 12<br>scans | Screening<br>and Day 28<br>scans | Day 12 and<br>Day 28 scans |
| iVaw | mL | Х | Х | Х | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| siVaw | mL/L | Х | Х | Х | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| iRaw | KPa*s/L | | | | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| siRaw | KPa*s | | | | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| iVlobe | L | Х | Х | Х | | | |
| Percent<br>Predicted iVlobe | % of<br>Predicted<br>value | Х | х | Х | | | |
| IALD <sup>[3]</sup> | % | Х | х | х | | | |
| LAS [1] | % of iVlobe | х | х | Х | | | |
| AT [2] | % of iVlobe | Х | Х | Х | | | |
| BVD [1] | % of iVlobe | Х | Х | Х | | | |
| iVaww <sup>[1]</sup> | mL | Х | Х | Х | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |
| siVaww [1] | mL/L | Х | Х | х | x (Screening)<br>x (Day 12) | x (Screening)<br>x (Day 28) | x (Day 12)<br>x (Day 28) |

201928

| | | Untrimmed | | | Scan Trimming, based on: | | |
|---|---|---|---|---|---|---|---|
| Endpoints | Units | Screening | Day<br>12 | Day 28 | Screening<br>and Day 12<br>scans | Screening<br>and Day 28<br>scans | Day 12 and<br>Day 28 scans |
| Trachea length | mm | х | х | х | | | |
| Trachea<br>Diameter | mm | Х | х | х | | | |
| Trachea<br>Length/Diameter | mm/mm | Х | х | х | | | |

All these endpoints will be measured at TLC and FRC, except:

- [1] These endpoints will only be measured at TLC
- [2] This endpoint will be measured only at FRC
- [3] The state (TLC/FRC) is not applicable

For the endpoints siVaw, iVaw, iRaw and siRaw appropriate transformations will be applied prior to summaries and statistical analyses, likely a log transformation. Summary statistics will be presented for absolute data and change from baseline. An attempt will be made to fit separate statistical models for each endpoint, scan trimming condition (Untrimmed or Scan Trimmed), lung volume (FRC or TLC) and Lobes (RUL, LUL, RML, RLL and LLL) or Regions (Upper, Lower, Central, Distal and Total) combination as appropriate. The primary plan for statistical analyses will be to fit separate statistical models for:

#### siVaw

- o Untrimmed at FRC for all lobes, i.e. RUL, LUL, RML, RLL and LLL in one model.
- o Untrimmed at FRC for all regions, i.e. Upper, Lower, Central, Distal and Total in one model.
- o Scan Trimmed at FRC for Distal region only.

#### siRaw

o Scan Trimmed at FRC for Distal region only.

For untrimmed data, the ratio from baseline across the different Regions (accounting for the average baseline associated to the Region of interest) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). In addition, the placebo-adjusted ratio from baseline across the different Regions will be represented via adjusted posterior medians, as well as their associated 95% HPD-tailed credible intervals and posterior probabilities. These results will be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

For scan trimmed data, the change from baseline across the different Regions (accounting for the average baseline associated to the Region of interest) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated

201928

95% HPD-tailed credible intervals. These results will be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). In addition, the placebo-adjusted change from baseline across the different Regions will be represented via adjusted posterior medians, as well as their associated 95% HPD-tailed credible intervals and posterior probabilities. These results will be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

For the tracheal endpoints, absolute data and change from baseline summary statistics will be provided for each lung volume (FRC or TLC) for trachea length, diameter and length/diameter.

# 8.2.3. Population of Interest

The primary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

# 8.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 8.2.4.1. Statistical Methodology Specification

NOTE: The description below describes the current thinking of how to analyse these endpoints. The proposed models will be assessed, and if not appropriate alternative models could be used.

# **Endpoint / Variables**

Imaging Untrimmed endpoint siVaw at FRC

#### **Model Specification**

- The data will be inspected prior to analysis to determine whether a data transformation is required. It is likely that the data will approximately follow a log normal distribution; however, the most appropriate distribution should be used.
- It is thought that the use of bronchodilators could affect the HRCT results. The database will contain information on whether relief medication was used in the 4 hours prior to each scan, and this information may be used in the sensitivity analyses of the HRCT results.
- An attempt will be made to fit a statistical model for all Lobes (RUL, LUL, RML, RLL and LLL) and a separate statistical model for all Regions (Upper, Lower, Central, Distal and Total), i.e. two models; one for lobes, one for regions. However, should this model fail to converge or be deemed unsuitable potentially due to sample size, separate statistical models will be fitted for each Lobe/Region (RUL, LUL, RML, RLL, LLL, Upper, Lower, Central, Distal and Total), i.e. ten models in total, one for each lobe/region endpoint.

201928

- The log of (or other transformation as appropriate) the ratio from baseline will be analysed in a multivariate model), under a Bayesian framework. The model will include a Baseline\*Region term and a Treatment\*Visit\*Region term, as well as any co-variates of interest. Note that the model will not include an intercept. The Visit will consist of two levels: Day 12 and Day 28, and the Treatment will consist of two levels: All NEMI and All Placebo. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e. covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The change from baseline (accounting for the average baseline) across the different Visits will
  be represented via adjusted posterior medians for each of the Treatment Arms, as well as their
  associated 95% HPD-tailed credible intervals. These results will also be presented within
  tabular form, and will be presented after the data have been appropriately back transformed (if
  applicable).
- The difference between the treatment arms, for the change from baseline across the different
  Visits will be represented via adjusted medians, as well as their associated 95% HPD-tailed
  credible intervals. These results will also be presented within tabular form, and will be
  presented after the data have been appropriately back transformed (if applicable)
- The probabilities that the treatment ratio is greater than 1 (depending on direction of the
  endpoint), in addition to other values appropriately selected based on the data, will also be
  computed for each Visit. These results will be presented in tabular format

# **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data. For example, if data do not approximately follow a normal distribution then attempt will be made to find a suitable transformation.
  - Note: Should parameters require a log transformation with an offset, for each posterior sample (i) appropriately back transformed values will be calculated for each treatment arm, and then (ii) using these back transformed values, the ratio of the treatment arms (All NEMI/All Placebo) will be calculated for each posterior sample, and finally summarised accordingly
- A comprehensive investigation into a suitable model should be initiated. For example, additional covariates will be investigated such as age, BMI, gender etc. Note: when investigating fitting separate statistical models for Lobes (RUL, LUL, RML, RLL and LLL) and Regions (Upper, Lower, Central, Distal and Total), i.e. two models; one for lobes, one for regions. If there are convergence issues an alternative structure of fitting separate statistical models for each Lobe (RUL, LUL, RML, RLL and LLL) and each Region (Upper, Lower, Central, Distal and Total), i.e. ten models; five for lobes, five for regions. a similar model as described in Model Specification should be tested but will include a baseline and a Treatment\*Visit term instead of a Baseline\*Region term and a Treatment\*Visit\*Region term, respectively.

Note: It may also be prudent to investigate a model fitting baseline as a timepoint in which case the log of (or other transformation as appropriate) the absolute results will be analysed in a multivariate model, under a Bayesian framework. The model could include a Treatment\*Visit\*Region parameter, as well as any co-variates of interest. Note that this model would not include an intercept. The Visit would consist of three levels: Baseline, Day 12 and Day 28, and the Treatment would consist of three levels: Null (when Visit = Screening), NEMI

201928

- and Placebo. With assumptions as described in Model Specification.
- An unstructured covariance structure will be used. However, in the event that this model fails to converge, alternative correlation structures may be considered.
- Models with a Bayesian Framework will use vague priors. If appropriate, conjugate priors will be used. For example, for a multivariate model, the prior for the variance covariance matrix will be an inverse Wishart distribution.

#### **Model Results Presentation**

Output from the repeated measures modelling detailed above will be tabulated. In particular,
the estimated ratio to baseline (or change from baseline if appropriate), 95% CI, standard error
(on the appropriate scale, likely logarithm base e), and posterior probabilities at each time point
and for the active treatment comparison with placebo. The scan trimming condition, lung
volume and lobe or region description will be included in the outputs.

### **Sensitivity and Supportive Analyses**

It is thought that the use of bronchodilators could affect the HRCT results. The database will
contain information on if relief medication was used in the 4 hours prior to each scan, and this
information may be used in the sensitivity analyses of the HRCT results including only those
who did not take bronchodilator relief medication in the 4 hours prior to HRCT scan.

# **Endpoint / Variables**

Imaging Scan Trimmed endpoints siVaw and siRaw at FRC in the Distal Region only.

# **Model Specification**

- It is likely that the data will approximately follow a log normal distribution; however, the most appropriate distribution should be used.
- Separate statistical models will be fitted for each endpoint, i.e. two models; one for siVaw (scan trimmed at FRC in Distal region), one for siRaw (scan trimmed at FRC in Distal region).
- The responses of interest are the change from baseline based on (i) Airways present on scans taken at Screening and Day 12, (ii) Airways present on scans taken at Screening and Day 28, and (iii) Airways present on scans taken at Day 12 and Day 28. The baselines for each of these endpoints are provided in the table below.

| | 1 | | (iii) Day 12 & Day 28<br>Scan trimming |
|---|---|---|---|
| Screening Result | ✓ (baseline) | ✓ (baseline) | |
| Day 12 Result | ✓ (post dose) | | ✓ (baseline) |
| Day 28 Result | | ✓ (post dose) | ✓ (post dose) |

 The modelling below assumes that the Scan trimming endpoints (Screening&Day12, Screening&Day28 and Day12&Day28) will be analysed in a single multivariate model. This is subject to sensitivity analysis.

201928

- The log of (or other transformation as appropriate) the change from baseline (where baseline is defined in the table above) will be analysed in a multivariate model to account for the correlation between the multiple Scan Trimmings (Screening&Day12, Screening&Day28 and Day12&Day28), under a Bayesian framework. The model will have a separate intercept for each Scan Trimming combination (by fitting a class parameter Scan Trimming, and having no overall intercept), and will also include a baseline\*Scan Trimming and a Treatment\*Scan Trimming parameter. The Visit will consist of two levels: Day 12 and Day 28, the scan trimming will consist of three levels Screening&Day12, Screening&Day28 and Day12&Day28, and the Treatment will consist of two levels: All NEMI and All Placebo. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e. covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The change from baseline across the different Scan Trimming pairs (accounting for the
  average baseline) will be represented via adjusted posterior medians for each of the Treatment
  Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be
  presented within tabular form, and will be presented after the data have been appropriately
  back transformed (if applicable).
- The difference between the treatment arms, for the change from baseline across the different Scan Trimming pairs will be represented via adjusted medians, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (if applicable). For parameters that require a log transformation with an offset, for each posterior sample (i) appropriately back transformed values will be calculated for each treatment arm, and then (ii) using these back transformed values, the ratio of the treatment arms (Active/Placebo) will be calculated for each posterior sample, and finally summarised accordingly.

The probabilities that the treatment ratio is greater than 1 (for siVaw) and less than 1 (for siRaw), in addition to other values appropriately selected based on the data, will also be computed for each Visit. These results will be presented in tabular format.

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments maybe made based on the
  data. For example if data do not approximately follow a normal distribution then an attempt will
  be made to find a suitable transformation.
  - Note: Should parameters require a log transformation with an offset, for each posterior sample (i) appropriately back transformed values will be calculated for each treatment arm, and then (ii) using these back transformed values, the ratio of the treatment arms (All NEMI/All Placebo) will be calculated for each posterior sample, and finally summarised accordingly
- A comprehensive investigation into a suitable model should be initiated. For example, additional covariates will be investigated
- An unstructured covariance structure will be used. However, in the event that this model fails to converge, alternative correlation structures may be considered.
- Models with a Bayesian Framework will use vague priors. If appropriate, conjugate priors will be used. For example, for a multivariate model, the prior for the variance covariance matrix will be an inverse Wishart distribution.

201928

#### **Model Results Presentation**

Output from the repeated measures modelling detailed above will be tabulated. In particular,
the estimated ratio to baseline (or change from baseline if appropriate), 95% CI, standard error
(on the appropriate scale, likely logarithm base e), and posterior probabilities at each time point
and for the active treatment comparison with placebo. The scan trimming condition, lung
volume and lobe or region description will be included in the outputs.

# Sensitivity and Supportive Analyses

It is thought that the use of bronchodilators could affect the HRCT results. The database will
contain information on if relief medication was used in the 4 hours prior to each scan, and this
information may be used in the sensitivity analyses of the HRCT results including only those
who did not take bronchodilator relief medication in the 4 hours prior to HRCT scan.

# 8.3. Exploratory Efficacy Analyses (From HRCT Analyses)

#### 8.3.1. Endpoint / Variables

To assess the changes in other HRCT parameters such as low attenuation score after once daily repeat inhaled doses of nemiralisib administered to subjects with acute exacerbation of COPD, compared to placebo. Change from baseline for other CT parameters including low attenuation score after 12 days of treatment and after 28 days of treatment.

# 8.3.2. Summary Measure

The structure of HRCT endpoints is as described in Section 8.2.2, exploratory endpoints include:

- iVlobe
- Percent Predicted iVlobe
- IALD
- LAS
- AT
- BVD
- iVaww
- siVaww

For all endpoints, the data will be inspected prior to analyses to determine whether a data transformation is required. Appropriate transformations will be applied prior to summaries and statistical analyses. It is likely a log transformation will be required for iVlobe, LAS, IALD, BVD iVaww and siVaww, and that no transformation will be required for Percent Predicted iVlobe and AT, however, the most appropriate distribution should be used

Summary statistics will be presented for absolute data and change from baseline. Separate statistical models will be fitted for each scan trimming condition (Untrimmed or Scan Trimmed), lung volume (FRC or TLC) and Regions (Upper, Lower, Central, Distal

201928

and Total) combination as appropriate, note: statistical analyses will only be conducted on:

- IALD for upper and lower regions only (within the same model)
- LAS at TLC for total region only
- AT at FRC for total region only
- BVD at TLC for total region only
- siVaww untrimmed data at TLC for distal region only

For the endpoints: LAS, AT and BVD, separate statistical models will be fitted for the Total region only. The change from baseline (accounting for the average baseline associated to the region) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). The difference between the treatment arms, for the change from baseline will be represented via adjusted medians, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

For the endpoint IALD, a statistical model will be fitted for both the Upper and Lower regions. The change from baseline across the different regions (accounting for the average baseline associated to the region of interest) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). The difference between the treatment arms, for the change from baseline across the different regions will be represented via adjusted medians, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

For the endpoint siVaww, a statistical model will be fitted for the distal region using untrimmed data. The change from baseline (accounting for the average baseline associated to the region) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented within tabular form, and will be presented after the data have been appropriately back transformed (if applicable). The difference between the treatment arms, for the change from baseline will be represented via adjusted medians, as well as their associated 95% HPD-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios (or median differences if applicable).

# 8.3.3. Population of Interest

The secondary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

201928

# 8.3.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.3.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 8.3.4.1. Statistical Methodology Specification

For statistical analyses of IALD in the upper and lower regions refer to Section 8.2.4.1 for the analysis of untrimmed siVaw but note that it is likely only 1 statistical model would be fitted for the upper and lower regions only. If appropriate this could be adapted into two models; one for upper, one for lower. The probability that the treatment ratio is greater than 1 will be presented for the lower region and the probability that the treatment ratio is less than 1 will be presented for the upper region, in addition to other values appropriately selected based on the data.

For statistical analyses of LAS at TLC in the total region only, refer to Section 8.2.4.1 for the analysis of untrimmed siVaw but note only 1 statistical model would be fitted for the Total regions only. The probability that the treatment ratio is less than 1 will be presented, in addition to other values appropriately selected based on the data.

For statistical analyses of AT at FRC in the total region only, refer to Section 8.2.4.1 for the analysis of untrimmed siVaw however it is likely that no transformation will be required for this endpoint in which case the absolute change from baseline will be fitted and probabilities that the true treatment difference is less than 1, in addition to other values appropriately selected based on the data, will also be computed for each Visit. Note only 1 statistical model would be fitted for the Total regions only.

For statistical analyses of BVD at TLC in the total region only, refer to Section 8.2.4.1 for the analysis of untrimmed siVaw but note only 1 statistical model would be fitted for the Total regions only.

For statistical analyses of siVaww at TLC in the distal region only, refer to Section 8.2.4.1 for the analysis of untrimmed siVaw but note only 1 statistical model would be fitted for the Distal regions only. The probability that the treatment ratio is less than 1, in addition to other values appropriately selected based on the data will be presented.

# 8.4. Exploratory Efficacy Analyses (Not from HRCT Analyses)

# 8.4.1. Endpoint / Variables

Additional exploratory endpoints include the severity of index exacerbation, where exacerbations requiring hospitalisations are defined as severe and those not requiring hospitalisation are defined as moderate.

#### 8.4.2. Summary Measure

For the severity of index exacerbation, a summary table detailing the number and percentage of subjects who had moderate or severe index exacerbations. Note:

201928

exacerbations requiring hospitalisations are defined as severe and those not requiring hospitalisation are defined as moderate.

If available, data on exacerbations occurring during the study will be summarised. This may include investigator defined exacerbations (including information on moderate or severe) and concomitant medication defined exacerbations. Concomitant medication defined exacerbations will be defined as treatment with systemic/oral corticosteroids and/or antibiotics where the exacerbation is deemed to have ended if no additional treatment with systemic/oral corticosteroids and/or antibiotics is required within < 7days from the end of treatment for the primary exacerbation.

# 8.4.3. Population of Interest

The secondary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

# 8.4.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.4.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

201928

# 9. RELATIONSHIP BETWEEN THE PHARMACODYNAMIC AND BIOMARKER DATA AND THE HRCT DATA

# 9.1. Relationship between the mRNA data and the HRCT data

The relationship between a selection of the mRNA data and the HRCT data may be performed as an exploratory analysis. This may include scatter plots of individual participant data, linear regression lines, Pearson's correlation coefficient and 95% confidence intervals plots as appropriate. This data will be produced following SAC.
201928

## 10. SAFETY ANALYSES

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

## 10.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 10.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

## 10.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

201928

## 11. PHARMACOKINETIC ANALYSES

## 11.1. Secondary Pharmacokinetic Analyses

## 11.1.1. Endpoint / Variables

## 11.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3 Reporting Standards for Pharmacokinetic)

#### 11.1.1.2. Derived Pharmacokinetic Parameters

No non-compartmental analysis will be conducted for this study as such there will be no derived pharmacokinetic parameters.

## 11.1.2. Summary Measure

The concentrations of the samples will be summarised.

## 11.1.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

201928

# 12. REFERENCES

Quanjer Ph.H, Tammeling G.J, Cotes J.E., Pedersen O.F, Peslin R, Yernault J-C. Lung volumes and forced ventilatory flows; *European Respiratory Journal* 1993 6: 5-40

201928

## 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management

## 13.1.1. Important Protocol Deviations

Based on an assessment of the important protocol deviations listed in the PDMP, partial data exclusions or time-point exclusions may occur which may not remove a subject from the analysis population, but may exclude a portion of the subject's data.

201928

# 13.2. Appendix 2: Schedule of Activities

## 13.2.1. Protocol Defined Schedule of Events

## **Screening and Follow Up Visits**

| | Screening (up to 3 days prior to Visit 1) | Follow-up (7-14 days post-last dose) | Notes |
|---|---|---|---|
| Procedure | | | |
| Informed consent | X | | |
| Demography | X | | |
| Inclusion and exclusion criteria | X | | |
| Full physical exam, including height and weight | Х | | |
| Brief physical examination, including weight | | X | |
| Chest X-Ray | Х | | To be done before baseline HRCT to exclude significant pneumonia and other incidental serious underlying pathology. |
| Medical history (includes substance usage and Family history of premature CV disease) | X | | Substances: Drugs, Alcohol, tobacco via history. No drug, alcohol screening is required. |
| Past and current medical conditions (including cardiovascular medical history and therapy history) | Х | | |
| Laboratory assessments (include Hematology and biochemistry) <sup>1</sup> | X | Х | Historical values analysed by local lab to be used for eligibility assessment. Another sample must be collected and sent to central lab as soon as informed consent is obtained. |
| Hep B and Hep C screen <sup>2</sup> | X | | |
| Urine pregnancy test (only WCBP) | X | | Before conducting the HRCT. Done locally at the site. |
| 12-lead ECG | X | X | Single assessment |
| Vital signs | X | X | Single assessment |
| HRCT (at TLC and FRC) | Х | | Within 48 h of diagnosis, if subject otherwise eligible. Includes electronic monitoring of breathing (if applicable). Baseline HRCT will be reviewed by the local site's radiologist to identify any significant occurring underlying medical conditions that require further clinical management or monitoring. |

| Procedure | Screening (up to 3 days prior to Visit 1) | Follow-up<br>(7-14 days post-last dose) | Notes |
|---|---|---|---|
| Induced Sputum <sup>3</sup> | X <sup>4</sup> | | To include sputum culture pre-first dose. Culture to be done by the local site laboratory. |
| Blood sample for mRNA Analysis | X <sup>4</sup> | | Collected at any time on specified days |
| AE/SAE collection and review | | X | |
| Concomitant medication review | X | X | |

- 1. Due to the short screening window, central laboratory analysis results will not be available on time. Therefore, the local laboratory results should be used for eligibility assessment (to exclude severe subjects and underlying medical conditions). If local laboratory results are already available from diagnosis of current exacerbation, there is no need to take another sample for local analysis. A sample for central laboratory analysis should also be obtained. See Section 7.8.6 of Protocol Amendment 4 for further details.
- 2. If test otherwise performed within 3 months prior to first dose of study freatment, testing at screening is not required. Because of the short window for screening, treatment with GSK2269557 may start before receiving the result of the hepatitis tests. If subsequently the test is found to be positive, the subject may be withdrawn, as judged by the Principal Investigator in consultation with the Medical Monitor.
- 3. Induced sputum collection may be attempted on several occasions if an adequate sample is not produced at the first attempt.
- 4. To be collected at any time point before randomisation.

201928

## **Treatment Period**

| Procedure | Treatment Period | | | Notes | | | |
|---|---|---|---|---|---|---|---|
| Visit | 1 | 21 | 3 | 4 | 5 | 6 | |
| Day | 1 | Within 48h<br>/ discharge | 12 | 28 | 56 | 84 | |
| Visit window | N/A | ±1 days | ±2 days | ±2 days | - 4 / +2 days | - 4 / +2 days | |
| SAFETY ASSESSMENTS | | | | | | | |
| AE/SAE collection and review | <b>←===</b> = | ======= | ======= | ======= | ======== | :====→ | |
| Concomitant medication review | <del>-===</del> | ======== | ======= | ======= | ======== | :==== <del>&gt;</del> | |
| Reliever usage | <b>←===</b> | | | ., | | :==== <del>&gt;</del> | |
| Brief physical exam, including weight | X2 | | Χ | Х | Х | X | Pre-dose |
| Laboratory assessments (include haematology and biochemistry) | X <sup>2</sup> | | Χ | Х | X | Χ | Pre-dose |
| 12-lead ECG | X2 | | Χ | X | X | Χ | Pre-dose. Single assessment |
| Vital signs | X2 | | Χ | Х | Х | Χ | Pre-dose. Single assessment |
| Urine pregnancy test (only WCBP) | | | Χ | Х | | | Before conducting the HRCT |
| STUDY TREATMENT | | | | _ | | | |
| ELLIPTA™ Inhaler Training | Х | | | | | | Training conducted by reviewing the<br>Patient Information Leaflet with the<br>subject (no device will be used).<br>Additional training may be conducted at<br>the discretion of the investigator |
| Randomisation | X | | | | | | |
| Study drug administration | <b>←===</b> | ======== | ======= | | ======== | ====→ | Daily in the morning before breakfast, (with the exception of days when the subjects have a planned visit to the clinic. On those days, they will be dosed at the clinic). |
| Assessment of study treatment compliance | | | Х | X | Х | Χ | |
| Diary Card dispense and review at clinic | Х | | Х | Х | Х | Х | Refer to SRM for details. |

| Procedure | | Treatment Period | | | | | | Notes |
|---|---|---|---|---|---|---|---|---|
| | Visit | 1 | 21 | 3 | 4 | 5 | 6 | |
| | Day | 1 | Within 48h<br>/ discharge | 12 | 28 | 56 | 84 | |
| | Visit window | N/A | ±1 days | ±2 days | ±2 days | - 4 / +2 days | - 4 / +2 days | |
| EFFICACY ASSESSMENTS | | | | | | | | |
| HRCT (at TLC and FRC) | | | | Х | X | | | At any time on specified days. Includes electronic monitoring of breathing (if applicable). The radiologist may review any of the scan(s) if they wish, but this is NOT required for the study. A formal review is required at screening only by the radiologist. |
| FEV <sub>1</sub> and FVC | | Х | Х | Х | Х | Х | Х | In clinic only for all visits where possible. |
| PEF | | <del>(</del> ==== | | ====== | | ======= | | Daily before drug administration at home. If subject in hospital, this may be collected using the handheld device provided prior to drug administration. |

| OTHER ASSESSMENTS | | | | | | | |
|---|---|---|---|---|---|---|---|
| Blood sample for PK | Х | | Х | Х | Х | Х | Day 1: 5 min and 24 h post-dose. The 24 h post-dose time-point is optional for subjects not hospitalised. Pre-dose at all other time-points. |
| Sputum induction <sup>3</sup> | | | Х | Х | | Х | |
| Blood sample for mRNA analysis | | | Х | X | | Х | |
| Genetic sample (PGx) <sup>4</sup> | | Х | | | | | Collected at any time after randomisation |

- On discharge if the subject was hospitalized. Within 48 hours of first dose administration if the subject was not hospitalised. See Section 4.2 of Protocol Amendment 4
   Assessments do not need to be completed if screening assessments conducted within 48 hours
   Induced sputum collection may be repeated on several occasions if an adequate sample is not produced at the first attempt

- 4. Informed consent for optional sub-studies (e.g. genetics research) must be obtained before collecting a sample. May be obtained at any visits.

201928

# 13.3. Appendix 3: Assessment Windows

# 13.3.1. Definitions of Assessment Windows for Analyses

| Population | Target | Analysis V | Vindow | Analysis |
|---|---|---|---|---|
| | | Beginning Timepoint | Ending Timepoint | Timepoint |
| Screening | NA | 3 days prior to Visit 1<br>(Day 1) | Day 1 | Screening |
| Safety, | NA – Day of first dose | NA | NA | Visit 1 |
| Efficacy, Study<br>population and<br>all other<br>assessments | If subject was hospitalised: Target = On discharge If subject wasn't hospitalised: Target = Within 48 hours of first dose administration | Target -1 day | Target +1 day | Visit 2 |
| | Day 12 | Target -2 day | Target +2 day | Visit 3 |
| | Day 28 | Target -2 day | Target +2 day | Visit 4 |
| | Day 56 | Target -4 day | Target +2 day | Visit 5 |
| | Day 84 | Target -4 day | Target +2 day | Visit 6 |
| Follow-up | NA | 1 week following last day of dose | 2 weeks following the last day of dose | Follow-up |

201928

# 13.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 13.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the study treatment, unless otherwise specified

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

## 13.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 13.4.2. Treatment States for Adverse Events

| Flag | Definition |
|---|---|
| Pre-Treatment | If AE onset date is before the treatment start date. |
| | AE Start Date < Study Treatment Start Date |
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after treatment start date &amp; on or before treatment stop<br/>date.</li> </ul> |
| (On-Treatment) | • Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date. |
| Post-Treatment | If AE onset date is after the treatment stop date. |
| | AE Start Date > Study Treatment Stop Date |
| Onset Time Since | If Treatment Start Date > AE Onset Date, then |
| 1st Dose (Days) | Onset Time = AE Onset Date - Treatment Start Date |
| | <ul> <li>If Treatment Start Date ≤ AE Onset Date, then</li> </ul> |
| | Onset Time = AE Onset Date - Treatment Start Date +1 |
| | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing]. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

201928

# 13.5. Appendix 5: Data Display Standards & Handling Conventions

## 13.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently supply | The currently supported versions of SAS software (version 9.4) will be used. |
| Reporting Area | |
| HARP Server | : UK1SALX00175.corpnet2.com |
| HARP Compound | : ARPROD/GSK2269557/mid201928 |
| | Note: the current planned reporting effort is final_01, this may be superseded. |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to Legacy GSK A&amp;R dataset standards and Integrated Data<br/>Standards Library</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be get a second control of the second control | RTF files will be generated for all tables |

## 13.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- A project wide decision was made to present GSK2269557 as Nemiralisib (abbreviated to NEMI) refer to Section 5.1 for further details.

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

201928

| | <ul> <li>Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be<br/>included in listings but omitted from figures, summaries and statistical analyses.</li> </ul> |
|---|---|
| Unscheduled Visits | · |
| Unscheduled visit | s will not be included in summary tables. |
| <ul> <li>Unscheduled visit</li> </ul> | s will not be included in summary figures |
| All unscheduled v | isits will be included in listings. |
| Descriptive Summar | y Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |
| All graphics will b | e done using the SGPLOT/SGPANEL/SG template procedures |

# 13.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. Note: Use the separate NEMI DISKUS and NEMI ELLIPTA treatment groups |
| NONMEM/Pop PK<br>File | Not applicable. |
| NONMEM/PK/PD<br>File | Not applicable. |

201928

## 13.6. Appendix 6: Derived and Transformed Data

#### 13.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 13.3.1) the value closest to the target day
  for that window will be used. If values are the same distance from the target, then the mean will be
  taken
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety
  parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of
  related summary tables. This will also be applicable to relevant Potential Clinical Importance summary
  tables.

## **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing
    - → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 13.6.2. Study Population

#### **Treatment Compliance**

• Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

- Treatment compliance could be greater than 100% if there are events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.
- Planned Treatment Duration is defined as 84 days.

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

## Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### Demographics

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - o Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### Body Mass Index (BMI)

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

201928

## 13.6.3. **Efficacy**

#### **HRCT**

#### **Endpoints provided by FluidDA**

Y = Endpoints will be provided by FluidDA.

| | | | | | | | Lobes | & Regions | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | LLL | LUL | RML | RUL | RLL | LL | UL | CENTRAL | DISTAL | TOTAL | TRACHEA |
| iVaw | Υ | Υ | Υ | Υ | Υ | С | С | Υ | С | С | N/A |
| siVaw | С | С | С | С | С | С | С | С | С | С | N/A |
| iRaw | Υ | Υ | Υ | Υ | Υ | C | С | Υ | Υ | Υ | N/A |
| siRaw | С | С | С | С | С | С | С | С | С | С | N/A |
| iVlobe | Υ | Υ | Υ | Υ | Υ | С | С | N/A | N/A | С | N/A |
| iVlobepred | Υ | Υ | Υ | Υ | Υ | Υ | Υ | N/A | N/A | Υ | N/A |
| LAS | Υ | Υ | Υ | Υ | Υ | Υ | Υ | N/A | N/A | Υ | N/A |
| IALD | С | С | С | С | С | С | С | N/A | N/A | N/A | N/A |
| AT | Υ | Υ | Υ | Υ | Υ | Υ | Υ | N/A | N/A | Υ | N/A |
| BVD | Υ | Υ | Υ | Υ | Υ | Υ | Υ | N/A | N/A | Υ | N/A |
| iVaww | Υ | Υ | Υ | Υ | Υ | C | С | Υ | С | С | N/A |
| siVaww | С | С | С | С | С | С | С | С | С | С | N/A |
| Diameter | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | Υ |
| Length | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | Υ |
| Length/Diameter | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | N/A | С |

C = Endpoints will be Calculated by GSK (see Derived Data below)

#### Imaging Endpoints Calculated by GSK

iVaw LL = iVaw RLL + iVaw LLL

iVaw UL = iVaw RUL + iVaw RML + iVaw LUL

iVaw DISTAL = iVaw LL + iVaw UL

iVaw TOTAL = iVaw CENTRAL + iVaw DISTAL

iRaw LL = 1/ (1/iRaw RLL + 1/iRaw LLL)

iRaw UL = 1/ (1/iRaw RUL + 1/iRaw RML + 1/iRaw LUL)

iVlobe LL = iVlobe RLL + iVlobe LLL

iVlobe UL = iVlobe RUL + iVlobe RML + iVlobe LUL

iVlobe TOTAL = iVlobe LL + iVlobe UL

iVaww LL = iVaww RLL + iVaww LLL

iVaww UL = iVaww RUL + iVaww RML + iVaww LUL

iVaww DISTAL = iVaww LL + iVaww UL

iVaww TOTAL = iVaww CENTRAL + iVaww DISTAL

siVaw LLL = iVaw LLL / iVlobe LLL

siVaw LUL = iVaw LUL / iVlobe LUL

siVaw RML = iVaw RML / iVlobe RML

siVaw RUL = iVaw RUL / iVlobe RUL siVaw RLL = iVaw RLL / iVlobe RLL

siVaw LL = iVaw LL / iVlobe LL

siVaw UL = iVaw UL / iVlobe UL

siVaw CENTRAL = iVaw CENTRAL / iVlobe TOTAL

siVaw DISTAL = iVaw DISTAL / iVlobe TOTAL

siVaw TOTAL = iVaw TOTAL / iVlobe TOTAL

siRaw LLL = iRaw LLL \* iVlobe LLL

siRaw LUL = iRaw LUL \* iVlobe LUL

siRaw RML = iRaw RML \* iVlobe RML

siRaw RUL = iRaw RUL \* iVlobe RUL

siRaw RLL = iRaw RLL \* iVlobe RLL

siRaw LL = iRaw LL \* iVlobe LL

siRaw UL = iRaw UL \* iVlobe UL

201928

## **HRCT**

siRaw CENTRAL = iRaw CENTRAL \* iVlobe TOTAL

siRaw DISTAL = iRaw DISTAL \* iVlobe TOTAL

siRaw TOTAL = iRaw TOTAL \* iVlobe TOTAL

siVaww LLL = iVaww LLL / iVlobe LLL

siVaww LUL = iVaww LUL / iVlobe LUL

siVaww RML = iVaww RML / iVlobe RML

siVaww RUL = iVaww RUL / iVlobe RUL

siVaww RLL = iVaww RLL / iVlobe RLL

siVaww LL = iVaww LL / iVlobe LL

siVaww UL = iVaww UL / iVlobe UL

siVaww CENTRAL = iVaww CENTRAL / iVlobe TOTAL

siVaww DISTAL = iVaww DISTAL / iVlobe TOTAL

siVaww TOTAL = iVaww TOTAL / iVlobe TOTAL

IALD LLL = 100 \* (iVlobe LLL TLC - iVlobe LLL FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD LUL = 100 \* (iVlobe LUL TLC - iVlobe LUL FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD RML = 100 \* (iVlobe RML TLC - iVlobe RML FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD RUL = 100 \* (iVlobe RUL TLC - iVlobe RUL FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD RLL = 100 \* (iVlobe RLL TLC - iVlobe RLL FRC) / (iVlobe TOTAL TLC - iVlobe TOTAL FRC)

IALD LL = IALD RLL + IALD LLL

IALD UL = IALD RUL + IALD RML + IALD LUL

#### **Lung Function Parameters**

## **Lung Function Parameters Calculated by GSK**

- FEV1 % Predicted (Men) = 4.30\*Height 0.029\*Age 2.49
- FEV1 % Predicted (Women) = 3.95\*Height 0.025\*Age 2.60

Formulas have been taken from Quanjer, 1993 Lung volumes and forced ventilator flows [accessed: 23rd July 2015] where height is measured in metres and age in years at screening.

#### **Rescue Medication Endpoints**

#### Number of occasions bronchodilator taken in the last 24 per hours 4-week period derived by GSK

- Number of occasions bronchodilator taken in the last 24 hours were collected in the daily diary
- The table below shows which daily diary records are used to calculate the daily diary endpoints for each analysis time period. Any diary data collected in the post-treatment phase of the study will not be slotted.

| Daily Record | | |
|---------------------------|------------------------|----------------------|
| Beginning Timepoint (day) | Ending Timepoint (day) | Analysis Time Period |
| 1 | 28 | Weeks 1 – 4 |
| 29 | 56 | Weeks 5 – 8 |
| 57 | 84 | Weeks 9 – 12 |

Note: There is no Day 0. Any records with actual day>84 will not be assigned to a time period. Any records with actual day<0 may be assigned to a Week -1 (Baseline) time period

Note: Daily diary records that were not assigned to a time period will not be used in calculation of daily diary endpoints.

- For a subject to be counted in any time period for a given endpoint they must have at least one diary entry recorded for that endpoint during that time period.
- Any daily diary data that were collected post-study treatment discontinuation will be excluded from analysis, including four weekly period data summaries.
- If a subject has more than one daily diary record for any given day, the worst-case

201928

#### **Rescue Medication Endpoints**

response on that day for each endpoint will be used in the summaries and analyses. i.e. the maximum number of occasions of bronchodilator use reported will be counted for the day in question and used to determine if it was a rescue-free day

• The mean number of occasions of rescue use per day and percentage of rescue-free days, will be calculated for each subject during the four weekly periods defined above.

## 13.6.4. Safety

#### **ECG Parameters**

#### **RR Interval**

IF RR interval (msec) is not provided directly, then RR can be derived as:

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^2 \right] * 1000$$

If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value then
do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas
  will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

## 13.6.5. Pharmacodynamic and Biomarker

| Biomarker Category | Analyte | Method | Lab | Matrix | Total samples |
|---|---|---|---|---|---|
| Inflammatory Cytokine | IL-8 | MSD | Quest | Sputum | 4 |
| | IL-6 | MSD | Quest | Sputum | 4 |
| | $TNF\alpha$ | MSD | Quest | Sputum | 4 |
| Microbiome | Bacterial DNA | 16SRNA | GSK-RTP | Sputum | 4 |
| | Bacterial DNA | qPCR | GSK-RTP | Sputum | 4 |
| | Viral DNA | qPCR | GSK-RTP | Sputum | 4 |
| Transcriptomics | Human RNA | Affymetrix | Expression<br>Analysis | Blood | 4 |

## NOTES:

- Sampling times: Screening, day 12, day 28 and day 84
- Inflammatory cytokine biomarkers are elevated in COPD patients. Expected to reduce with treatment.
- · Microbiome biomarkers are drivers of exacerbations in COPD and are inhibited in preclinical disease studies
- PI3Kδ transcriptome analysis in FTIH study has 16 genes identified (sputum) showing a consistent response with dose – all are down regulated.

201928

#### Pharmacodynamic and Biomarker

#### Pharmacodynamic

#### **PMNs Differentials**

- Percentage data may be arc-sine transformed especially if many of the percentage values are smaller than 20% or larger than 80%. The response variable, y, measured in radians, is sin-1sqrt{0.01\*p} where p is the differential percentage.
- If transformations are used then the results will be reported on the back-transformed scale, except where a transformed value:
  - exceeds 0.01\*p/2 then the back-transformed value will be set equal to 100%
  - o is less than 0 then the back-transformed value will be set equal to 0%.

#### **Biomarkers**

#### **Inflammatory Cytokines**

- In general, it is assumed that biomarker endpoints will require variance stabilising transformations, such as taking a
  loge transformation prior to analysis (and that summary statistics appropriate to loge normally distributed data will
  apply for all summaries). However, this assumption will be considered for each endpoint Individually prior to the
  generation of summary tables or statistical analysis, and if deemed more appropriate, a loge transformation will not
  be applied, or non-parametric methods may be employed.
- If transformations are used, then the results will be reported on the back-transformed scale unless otherwise stated.

#### **RNA transcriptome**

- Affymetrix microarray mRNA data will be normalised using RMA in ARRAY STUDIO v8.0 or later by the Statistical
  Consultancy Group (SCG) within GSK. After normalisation, the data will be quality assessed and any samples
  deemed as QC fails will be excluded from any further analysis. This quality assessment will involve looking for
  outlying signals in both the normalised expression data and the MAS5 QC metrics generated from each sample. If
  any samples are excluded, the remaining data will be re-normalised. The output from the normalization will be log2
  transformed mRNA intensity data.
- Summary mRNA data will be reviewed and a decision made on which probe sets are to be included in the SI
  dataset.
- Treatment ratios from the statistical analyses of mRNA intensity data will be converted to fold changes as follows:
  - o If ratio ≥ 1 then fold change = ratio
  - If ratio < 1 then fold change = -1/ratio</li>

The primary pharmacodynamic endpoint is based on a subset of probe sets defined as those that have previously identified immune cell mechanisms specifically related to neutrophil function.

The gene list that meets this criterion based on PII115119 D14 vs D1 gene changes, PII115117 and Metacore neutrophil pathways identified in PII115119 study. This gene list identified 258 genes in total after filtering for redundancy and was agreed by the study team is presented in Table 3.

Table 3 Gene List that have previously identified immune cell mechanisms specifically related to neutrophil function

| Gene | Source | Gene | Source |
|---|---|---|---|
| CD177 | PII115119 - Neutrophil migration | ITGAL | Metacore: IL8 Neutrophil migration |
| CXCR1 | PII115119 - Neutrophil migration | ADAM17 | Metacore: Inhibition of neutrophil migration |
| CXCR2 | PII115119 - Neutrophil migration | C5 | Metacore: Inhibition of neutrophil migration |
| FPR2 | PII115119 - Neutrophil migration | C5AR1 | Metacore: Inhibition of neutrophil migration |
| LTB4R | PII115119 - Neutrophil migration | CCR5 | Metacore: Inhibition of neutrophil migration |
| PAK1 | PII115119 - Neutrophil migration | CD34 | Metacore: Inhibition of neutrophil migration |
| PXN | PII115119 - Neutrophil migration | CALM1 | Metacore: Inhibition of neutrophil migration |
| PREX1 | PII115119 - Neutrophil migration | CALM2 | Metacore: Inhibition of neutrophil migration |
| TLN1 | PII115119 - Neutrophil migration | CALM3 | Metacore: Inhibition of neutrophil migration |
| SSH2 | PII115119 - Neutrophil migration | FPR1 | Metacore: Inhibition of neutrophil migration |
| F2RL1 | PII115119 - Neutrophil infection response | ICAM2 | Metacore: Inhibition of neutrophil migration |
| TLR10 | PII115119 - Neutrophil infection response | IL1B | Metacore: Inhibition of neutrophil migration |
| CEACAM3 | PII115119 - Neutrophil infection response | IL1R1 | Metacore: Inhibition of neutrophil migration |
| TREML2 | PII115119 - Neutrophil infection response | ITPR1 | Metacore: Inhibition of neutrophil migration |
| DEFB124 | PII115119 - Neutrophil infection response | ITPR2 | Metacore: Inhibition of neutrophil migration |
| CLEC4C | PII115119 - Neutrophil infection response | ITPR3 | Metacore: Inhibition of neutrophil migration |
| IFITM1 | PII115119 - Neutrophil infection response | SELL | Metacore: Inhibition of neutrophil migration |
| CR1 | PII115119 - Neutrophil infection response | MSN | Metacore: Inhibition of neutrophil migration |
| PMAIP1 | FTIH - GSK'557 response | NFKB1 | Metacore: Inhibition of neutrophil migration |
| S100P | FTIH - GSK'557 response | NFKB2 | Metacore: Inhibition of neutrophil migration |
| PTGS2 | FTIH - GSK'557 response | REL | Metacore: Inhibition of neutrophil migration |
| CCL20 | FTIH - GSK'557 response | RELA | Metacore: Inhibition of neutrophil migration |
| EGR3 | FTIH - GSK'557 response | RELB | Metacore: Inhibition of neutrophil migration |
| H1F0 | FTIH - GSK'557 response | PECAM1 | Metacore: Inhibition of neutrophil migration |
| NCOA3 | FTIH - GSK'557 response | PRKCA | Metacore: Inhibition of neutrophil migration |
| TARP | FTIH - GSK'557 response | PRKCB | Metacore: Inhibition of neutrophil migration |
| CEACAM1 | FTIH - GSK'557 response | PRKCD | Metacore: Inhibition of neutrophil migration |
| TTPAL | FTIH - GSK'557 response | PRKCE | Metacore: Inhibition of neutrophil migration |
| VPS37B | FTIH - GSK'557 response | PRKCG | Metacore: Inhibition of neutrophil migration |
| SYAP1 | FTIH - GSK'557 response | PRKCH | Metacore: Inhibition of neutrophil migration |
| SPTBN1 | FTIH - GSK'557 response | PRKCI | Metacore: Inhibition of neutrophil migration |
| EGR1 | FTIH - GSK'557 response | PRKCQ | Metacore: Inhibition of neutrophil migration |
| OSM | FTIH - GSK'557 response | PRKD1 | Metacore: Inhibition of neutrophil migration |
| TBC1D22A | FTIH - GSK'557 response | PRKD2 | Metacore: Inhibition of neutrophil migration |
| AKT1 | Metacore: IL8 Neutrophil migration | PRKD3 | Metacore: Inhibition of neutrophil migration |
| AKT2 | Metacore: IL8 Neutrophil migration | PLCB2 | Metacore: Inhibition of neutrophil migration |
| AKT3 | Metacore: IL8 Neutrophil migration | PTAFR | Metacore: Inhibition of neutrophil migration |
| ACTA1 | Metacore: IL8 Neutrophil migration | TLR2 | Metacore: Inhibition of neutrophil migration |
| ACTA2 | Metacore: IL8 Neutrophil migration | TLR4 | Metacore: Inhibition of neutrophil migration |

| Gene | Source | Gene | Source |
|---|---|---|---|
| ACTB | Metacore: IL8 Neutrophil migration | TNFRSF1A | Metacore: Inhibition of neutrophil migration |
| ACTC1 | Metacore: IL8 Neutrophil migration | TNFRSF1B | Metacore: Inhibition of neutrophil migration |
| ACTG1 | Metacore: IL8 Neutrophil migration | TNF | Metacore: Inhibition of neutrophil migration |
| ACTG2 | Metacore: IL8 Neutrophil migration | VAV1 | Metacore: Inhibition of neutrophil migration |
| MYH1 | Metacore: IL8 Neutrophil migration | EZR | Metacore: Inhibition of neutrophil migration |
| MYH10 | Metacore: IL8 Neutrophil migration | VCL | Metacore: Inhibition of neutrophil migration |
| MYH11 | Metacore: IL8 Neutrophil migration | ITGAM | Metacore: Inhibition of neutrophil migration |
| MYH13 | Metacore: IL8 Neutrophil migration | ABL1 | Metacore: Inhibition of neutrophil migration |
| MYH14 | Metacore: IL8 Neutrophil migration | JUN | Metacore: Inhibition of neutrophil migration |
| MYH15 | Metacore: IL8 Neutrophil migration | FOS | Metacore: Inhibition of neutrophil migration |
| MYH16 | Metacore: IL8 Neutrophil migration | MAPK11 | Metacore: Inhibition of neutrophil migration |
| MYH2 | Metacore: IL8 Neutrophil migration | MAPK12 | Metacore: Inhibition of neutrophil migration |
| MYH3 | Metacore: IL8 Neutrophil migration | MAPK13 | Metacore: Inhibition of neutrophil migration |
| MYH4 | Metacore: IL8 Neutrophil migration | MAPK14 | Metacore: Inhibition of neutrophil migration |
| MYH6 | Metacore: IL8 Neutrophil migration | BDKRB1 | Metacore: Neutrophil migration in Asthma |
| MYH7 | Metacore: IL8 Neutrophil migration | CCL15 | Metacore: Neutrophil migration in Asthma |
| MYH8 | Metacore: IL8 Neutrophil migration | CCL2 | Metacore: Neutrophil migration in Asthma |
| MYH9 | Metacore: IL8 Neutrophil migration | CCL5 | Metacore: Neutrophil migration in Asthma |
| MYL1 | Metacore: IL8 Neutrophil migration | CCL7 | Metacore: Neutrophil migration in Asthma |
| MYL12A | Metacore: IL8 Neutrophil migration | CCR1 | Metacore: Neutrophil migration in Asthma |
| MYL12B | Metacore: IL8 Neutrophil migration | CCR2 | Metacore: Neutrophil migration in Asthma |
| MYL2 | Metacore: IL8 Neutrophil migration | CCR3 | Metacore: Neutrophil migration in Asthma |
| MYL3 | Metacore: IL8 Neutrophil migration | CXCL5 | Metacore: Neutrophil migration in Asthma |
| MYL4 | Metacore: IL8 Neutrophil migration | CXCL1 | Metacore: Neutrophil migration in Asthma |
| MYL5 | Metacore: IL8 Neutrophil migration | CXCL2 | Metacore: Neutrophil migration in Asthma |
| MYL6 | Metacore: IL8 Neutrophil migration | CXCL3 | Metacore: Neutrophil migration in Asthma |
| MYL6B | Metacore: IL8 Neutrophil migration | HSPA14 | Metacore: Neutrophil migration in Asthma |
| MYL7 | Metacore: IL8 Neutrophil migration | HSPA1A | Metacore: Neutrophil migration in Asthma |
| MYL9 | Metacore: IL8 Neutrophil migration | HSPA1B | Metacore: Neutrophil migration in Asthma |
| MYLPF | Metacore: IL8 Neutrophil migration | HSPA1L | Metacore: Neutrophil migration in Asthma |
| ACTN1 | Metacore: IL8 Neutrophil migration | HSPA2 | Metacore: Neutrophil migration in Asthma |
| ACTN2 | Metacore: IL8 Neutrophil migration | HSPA4 | Metacore: Neutrophil migration in Asthma |
| ACTN3 | Metacore: IL8 Neutrophil migration | HSPA5 | Metacore: Neutrophil migration in Asthma |
| ACTN4 | Metacore: IL8 Neutrophil migration | HSPA6 | Metacore: Neutrophil migration in Asthma |
| ACTR2 | Metacore: IL8 Neutrophil migration | HSPA7 | Metacore: Neutrophil migration in Asthma |
| ACTR3 | Metacore: IL8 Neutrophil migration | HSPA8 | Metacore: Neutrophil migration in Asthma |
| ACTR3B | Metacore: IL8 Neutrophil migration | HSPA9 | Metacore: Neutrophil migration in Asthma |
| ARPC1A | Metacore: IL8 Neutrophil migration | MIF | Metacore: Neutrophil migration in Asthma |
| ARPC1B | Metacore: IL8 Neutrophil migration | CCL3 | Metacore: Neutrophil migration in Asthma |
| ARPC2 | Metacore: IL8 Neutrophil migration | PGF | Metacore: Neutrophil migration in Asthma |
| ARPC3 | Metacore: IL8 Neutrophil migration | TAC1 | Metacore: Neutrophil migration in Asthma |

| Gene | Source | Gene | Source |
|---|---|---|---|
| ARPC4 | Metacore: IL8 Neutrophil migration | TACR1 | Metacore: Neutrophil migration in Asthma |
| ARPC5 | Metacore: IL8 Neutrophil migration | KLK1 | Metacore: Neutrophil migration in Asthma |
| CFL1 | Metacore: IL8 Neutrophil migration | KLK10 | Metacore: Neutrophil migration in Asthma |
| CFL2 | Metacore: IL8 Neutrophil migration | KLK11 | Metacore: Neutrophil migration in Asthma |
| MAPK1 | Metacore: IL8 Neutrophil migration | KLK12 | Metacore: Neutrophil migration in Asthma |
| MAPK3 | Metacore: IL8 Neutrophil migration | KLK13 | Metacore: Neutrophil migration in Asthma |
| GNAI1 | Metacore: IL8 Neutrophil migration | KLK14 | Metacore: Neutrophil migration in Asthma |
| GNAI2 | Metacore: IL8 Neutrophil migration | KLK15 | Metacore: Neutrophil migration in Asthma |
| GNAI3 | Metacore: IL8 Neutrophil migration | KLK2 | Metacore: Neutrophil migration in Asthma |
| GNAO1 | Metacore: IL8 Neutrophil migration | KLK3 | Metacore: Neutrophil migration in Asthma |
| GNAZ | Metacore: IL8 Neutrophil migration | KLK4 | Metacore: Neutrophil migration in Asthma |
| GNB1 | Metacore: IL8 Neutrophil migration | KLK5 | Metacore: Neutrophil migration in Asthma |
| GNB2 | Metacore: IL8 Neutrophil migration | KLK6 | Metacore: Neutrophil migration in Asthma |
| GNB3 | Metacore: IL8 Neutrophil migration | KLK7 | Metacore: Neutrophil migration in Asthma |
| GNB4 | Metacore: IL8 Neutrophil migration | KLK8 | Metacore: Neutrophil migration in Asthma |
| GNB5 | Metacore: IL8 Neutrophil migration | KLK9 | Metacore: Neutrophil migration in Asthma |
| GNG10 | Metacore: IL8 Neutrophil migration | FLT1 | Metacore: Neutrophil migration in Asthma |
| GNG11 | Metacore: IL8 Neutrophil migration | RUNX1 | Metacore: Transcription regulation of granulocytes |
| GNG12 | Metacore: IL8 Neutrophil migration | CEBPA | Metacore: Transcription regulation of granulocytes |
| GNG13 | Metacore: IL8 Neutrophil migration | CEBPE | Metacore: Transcription regulation of granulocytes |
| GNG2 | Metacore: IL8 Neutrophil migration | ANPEP | Metacore: Transcription regulation of granulocytes |
| GNG3 | Metacore: IL8 Neutrophil migration | PTPRC | Metacore: Transcription regulation of granulocytes |
| GNG4 | Metacore: IL8 Neutrophil migration | E2F1 | Metacore: Transcription regulation of granulocytes |
| GNG5 | Metacore: IL8 Neutrophil migration | CSF3 | Metacore: Transcription regulation of granulocytes |
| GNG7 | Metacore: IL8 Neutrophil migration | CSF3R | Metacore: Transcription regulation of granulocytes |
| GNG8 | Metacore: IL8 Neutrophil migration | GATA1 | Metacore: Transcription regulation of granulocytes |
| GNGT1 | Metacore: IL8 Neutrophil migration | JAK1 | Metacore: Transcription regulation of granulocytes |
| GNGT2 | Metacore: IL8 Neutrophil migration | JAK2 | Metacore: Transcription regulation of granulocytes |
| ICAM1 | Metacore: IL8 Neutrophil migration | LRG1 | Metacore: Transcription regulation of granulocytes |
| CXCL8 | Metacore: IL8 Neutrophil migration | LTF | Metacore: Transcription regulation of granulocytes |
| ITGB2 | Metacore: IL8 Neutrophil migration | ELANE | Metacore: Transcription regulation of granulocytes |
| LIMK1 | Metacore: IL8 Neutrophil migration | LYZ | Metacore: Transcription regulation of granulocytes |
| MYLK | Metacore: IL8 Neutrophil migration | MXD1 | Metacore: Transcription regulation of granulocytes |
| MYLK2 | Metacore: IL8 Neutrophil migration | MAX | Metacore: Transcription regulation of granulocytes |
| MYLK3 | Metacore: IL8 Neutrophil migration | PRTN3 | Metacore: Transcription regulation of granulocytes |
| PPP1CB | Metacore: IL8 Neutrophil migration | MPO | Metacore: Transcription regulation of granulocytes |
| PPP1R12A | Metacore: IL8 Neutrophil migration | SPI1 | Metacore: Transcription regulation of granulocytes |
| PDPK1 | Metacore: IL8 Neutrophil migration | RARA | Metacore: Transcription regulation of granulocytes |
| PIK3CG | Metacore: IL8 Neutrophil migration | RXRA | Metacore: Transcription regulation of granulocytes |
| PIK3R5 | Metacore: IL8 Neutrophil migration | SOCS3 | Metacore: Transcription regulation of granulocytes |
| PIP5K1A | Metacore: IL8 Neutrophil migration | STAT3 | Metacore: Transcription regulation of granulocytes |

201928

| Gene | Source | Gene | Source |
|---|---|---|---|
| PIP5K1B | Metacore: IL8 Neutrophil migration | STAT5A | Metacore: Transcription regulation of granulocytes |
| PIP5K1C | Metacore: IL8 Neutrophil migration | STAT5B | Metacore: Transcription regulation of granulocytes |
| PRKCZ | Metacore: IL8 Neutrophil migration | FES | Metacore: Transcription regulation of granulocytes |
| PLD1 | Metacore: IL8 Neutrophil migration | MYB | Metacore: Transcription regulation of granulocytes |
| PLPP6 | Metacore: IL8 Neutrophil migration | MYC | Metacore: Transcription regulation of granulocytes |
| RAC1 | Metacore: IL8 Neutrophil migration | CYBB | Metacore: Transcription regulation of granulocytes |
| RAC2 | Metacore: IL8 Neutrophil migration | NCF1 | Metacore: Transcription regulation of granulocytes |
| TLN2 | Metacore: IL8 Neutrophil migration | NCF2 | Metacore: Transcription regulation of granulocytes |

Gene names converted to Affymetrix probe ID, resulted in 638 probes in total, these are presented in Table 4.

Table 4 Probe Set that have previously identified immune cell mechanisms specifically related to neutrophil function

| Gene | Probe ID | Gene | Probe ID |
|-------|-------------------------|--------|--------------|
| ABL1 | 202123_s_at | KLK7 | 239381_at |
| ACTA1 | 203872_at | KLK8 | 1552319_a_at |
| ACTA2 | 200974_at | KLK8 | 206125_s_at |
| ACTA2 | 215787_at | KLK9 | 233687_s_at |
| ACTA2 | 243140_at | LIMK1 | 204356_at |
| ACTB | 200801_x_at | LIMK1 | 204357_s_at |
| ACTB | 213867_x_at | LIMK1 | 208372_s_at |
| ACTB | 224594_x_at | LRG1 | 228648_at |
| ACTB | AFFX-HSAC07/X00351_3_at | LTB4R | 210128_s_at |
| ACTB | AFFX-HSAC07/X00351_5_at | LTB4R | 216388_s_at |
| ACTB | AFFX-HSAC07/X00351_M_at | LTB4R | 236172_at |
| ACTC1 | 205132_at | LTF | 202018_s_at |
| ACTG1 | 201550_x_at | LYZ | 1555745_a_at |
| ACTG1 | 211970_x_at | LYZ | 213975_s_at |
| ACTG1 | 211983_x_at | MAPK1 | 1552263_at |
| ACTG1 | 211995_x_at | MAPK1 | 1552264_a_at |
| ACTG1 | 212363_x_at | MAPK1 | 208351_s_at |
| ACTG1 | 212988_x_at | MAPK1 | 212271_at |
| ACTG1 | 213214_x_at | MAPK1 | 224620_at |
| ACTG1 | 221607_x_at | MAPK1 | 224621_at |
| ACTG1 | 224585_x_at | MAPK1 | 229847_at |
| ACTG2 | 202274_at | MAPK11 | 206040_s_at |
| ACTG2 | 241148_at | MAPK11 | 211499_s_at |
| ACTN1 | 208636_at | MAPK11 | 211500_at |
| ACTN1 | 208637_x_at | MAPK12 | 1556340_at |
| ACTN1 | 211160_x_at | MAPK12 | 1556341_s_at |
| ACTN1 | 237401_at | MAPK12 | 206106_at |
| ACTN2 | 203861_s_at | MAPK13 | 210058_at |
| ACTN2 | 203862_s_at | MAPK13 | 210059_s_at |
| ACTN2 | 203863_at | MAPK14 | 202530_at |
| ACTN2 | 203864_s_at | MAPK14 | 210449_x_at |
| ACTN3 | 206891_at | MAPK14 | 211087_x_at |
| ACTN4 | 200601_at | MAPK14 | 211561_x_at |
| ACTR2 | 1554390_s_at | MAPK3 | 212046_x_at |

| Gene | Probe ID | Gene | Probe ID |
|--------|--------------|--------|--------------------|
| ACTR2 | 1558015_s_at | MAX | 208403_x_at |
| ACTR2 | 200727_s_at | MAX | 209331_s_at |
| ACTR2 | 200728_at | MAX | 209332_s_at |
| ACTR2 | 200729_s_at | MAX | 210734_x_at |
| ACTR2 | 234210 x at | MAX | 214108_at |
| ACTR2 | 234212_at | MIF | 217871_s_at |
| ACTR3 | 200996_at | MPO | 203948 s_at |
| ACTR3 | 213101_s_at | MPO | 203949 at |
| ACTR3 | 213102_at | MSN | 200600_at |
| ACTR3 | 228603 at | MSN | 233749 at |
| ACTR3 | 239170 at | MXD1 | 206877_at |
| ACTR3B | 1555487 a at | MXD1 | 226275 at |
| ACTR3B | 218868_at | MXD1 | 228846_at |
| ADAM17 | 205745 x at | MYB | 204798 at |
| ADAM17 | 205746_s_at | MYB | 215152_at |
| ADAM17 | 213532 at | MYC | 202431_s_at |
| ADAM17 | 237897_at | MYH1 | 205951_at |
| AKT1 | 207163 s_at | MYH10 | 212372_at |
| AKT2 | 1560689_s_at | MYH10 | 213067_at |
| AKT2 | 203808_at | MYH11 | 1568760_at |
| AKT2 | 203809_s_at | MYH11 | 201495_x_at |
| AKT2 | 211453 s_at | MYH11 | 201496 x at |
| AKT2 | 225471_s_at | MYH11 | 201497_x_at |
| AKT2 | 226156_at | MYH11 | 207961 x at |
| AKT2 | 236664 at | MYH11 | 228133_s_at |
| AKT3 | 212607_at | MYH11 | 228134_at |
| AKT3 | 212609_s_at | MYH11 | 239307_at |
| AKT3 | 219393 s_at | MYH13 | 208208_at |
| AKT3 | 222880 at | MYH14 | 217545_at |
| AKT3 | 224229_s_at | MYH14 | 217660_at |
| AKT3 | 242876 at | MYH14 | 219946_x_at |
| AKT3 | 242879_x_at | MYH14 | 226988_s_at |
| ANPEP | 202888_s_at | MYH14 | 232977_x_at |
| ANPEP | 234458_at | MYH14 | 234290_x_at |
| ANPEP | 234576_at | MYH15 | 215331_at |
| ARPC1A | 200950 at | MYH16 | 1564072_at |
| ARPC1B | 201954_at | MYH2 | 204631_at |
| ARPC2 | 207988_s_at | MYH3 | 205940_at |
| ARPC2 | 208679_s_at | MYH4 | 208148 at |
| ARPC2 | 213513_x_at | MYH6 | 214468 at |
| ARPC3 | 208736 at | MYH7 | 204737_s_at |
| ARPC4 | 211672_s_at | MYH7 | 216265_x_at |
| ARPC4 | 217817_at | MYH8 | 206717_at |
| ARPC4 | 217818_s_at | MYH8 | 34471 at |
| ARPC5 | 1555797_a_at | MYH9 | 211926 s at |
| ARPC5 | 1569325_at | MYL1 | 209888_s_at |
| ARPC5 | 211963_s_at | MYL12A | 1555976 s at |
| ARPC5 | 237387_at | MYL12A | 1555977_at |
| BDKRB1 | 207510 at | MYL12A | 1555978 s at |
| C5 | 205500 at | MYL12A | 201318_s_at |
| C5AR1 | 220088_at | MYL12A | 201319_at |
| CCL15 | 210390_s_at | MYL12B | 221474_at |
| CCL2 | 216598 s at | MYL2 | 209742 s at |
| CCL20 | 205476_at | MYL3 | 205589 at |
| 00120 | -00 11 0_at | IVIILO | 1 = 0 0 0 0 0 _ ut |

| Gene | Probe ID | Gene | Probe ID |
|---------|--------------|--------|--------------|
| CCL3 | 205114_s_at | MYL4 | 210088_x_at |
| CCL5 | 1405_i_at | MYL4 | 210395_x_at |
| CCL5 | 1555759_a_at | MYL4 | 216054_x_at |
| CCL5 | 204655_at | MYL4 | 217274_x_at |
| CCL7 | 208075_s_at | MYL5 | 205145_s_at |
| CCR1 | 205098_at | MYL6 | 212082_s_at |
| CCR1 | 205099_s_at | MYL6 | 214002_at |
| CCR2 | 206978_at | MYL6B | 204173_at |
| CCR2 | 207794_at | MYL7 | 219942_at |
| CCR3 | 208304_at | MYL9 | 201058_s_at |
| CCR5 | 206991_s_at | MYL9 | 244149_at |
| CD177 | 219669_at | MYLK | 1563466_at |
| CD34 | 209543_s_at | MYLK | 1568770_at |
| CEACAM1 | 206576_s_at | MYLK | 1569956_at |
| CEACAM1 | 209498_at | MYLK | 202555_s_at |
| CEACAM1 | 210610_at | MYLK | 224823_at |
| CEACAM1 | 211883_x_at | MYLK2 | 231792_at |
| CEACAM1 | 211889_x_at | MYLK3 | 1562411_at |
| CEACAM3 | 208052_x_at | MYLK3 | 1568925_at |
| CEACAM3 | 210789_x_at | MYLK3 | 1568926_x_at |
| CEACAM3 | 217209_at | MYLK3 | 217623_at |
| CEBPA | 204039_at | MYLK3 | 238834_at |
| CEBPE | 214523_at | MYLPF | 205163_at |
| CFL1 | 1555730_a_at | NCF1 | 204961_s_at |
| CFL1 | 200021_at | NCF1 | 214084_x_at |
| CFL1 | 230870_at | NCF2 | 209949_at |
| CFL1 | 236792_at | NCOA3 | 1562439_at |
| CFL2 | 224352_s_at | NCOA3 | 207700_s_at |
| CFL2 | 224663_s_at | NCOA3 | 209060_x_at |
| CFL2 | 233496_s_at | NCOA3 | 209061_at |
| CLEC4C | 1552552_s_at | NCOA3 | 209062_x_at |
| CLEC4C | 1555687_a_at | NCOA3 | 211352_s_at |
| CR1 | 206244_at | NFKB1 | 209239_at |
| CR1 | 208488_s_at | NFKB2 | 207535_s_at |
| CR1 | 217484_at | NFKB2 | 209636_at |
| CR1 | 217552_x_at | NFKB2 | 211524_at |
| CR1 | 244313_at | OSM | 214637_at |
| CSF3 | 207442_at | OSM | 230170_at |
| CSF3R | 1553297_a_at | PAK1 | 1565772_at |
| CSF3R | 203591_s_at | PAK1 | 209615_s_at |
| CXCL1 | 204470_at | PAK1 | 226507_at |
| CXCL2 | 1569203_at | PAK1 | 230100_x_at |
| CXCL2 | 209774_x_at | PDPK1 | 204524_at |
| CXCL2 | 230101_at | PDPK1 | 221244_s_at |
| CXCL3 | 207850_at | PDPK1 | 224986_s_at |
| CXCL5 | 207852_at | PDPK1 | 244629_s_at |
| CXCL5 | 214974_x_at | PDPK1 | 244630_at |
| CXCL5 | 215101_s_at | PDPK1 | 32029_at |
| CXCL8 | 202859_x_at | PECAM1 | 1558397_at |
| CXCL8 | 211506_s_at | PECAM1 | 1559921_at |
| CXCR1 | 207094_at | PECAM1 | 208981_at |
| CXCR2 | 207008_at | PECAM1 | 208982_at |
| CYBB | 203922_s_at | PECAM1 | 208983_s_at |
| CYBB | 203923_s_at | PGF | 209652_s_at |

| Gene | Probe ID | Gene | Probe ID |
|---------|--------------|----------|--------------|
| CYBB | 217431_x_at | PGF | 215179_x_at |
| CYBB | 233538_s_at | PIK3CG | 206369_s_at |
| DEFB124 | 1568375_at | PIK3CG | 206370_at |
| DEFB124 | 1568377_x_at | PIK3CG | 239294_at |
| E2F1 | 2028_s_at | PIK3R5 | 220566_at |
| E2F1 | 204947_at | PIK3R5 | 227553_at |
| EGR1 | 201693_s_at | PIK3R5 | 227645_at |
| EGR1 | 201694_s_at | PIP5K1A | 207391_s_at |
| EGR1 | 227404_s_at | PIP5K1A | 210256_s_at |
| EGR3 | 206115_at | PIP5K1A | 211205_x_at |
| ELANE | 206871_at | PIP5K1B | 205632_s_at |
| EZR | 208621_s_at | PIP5K1B | 217477_at |
| EZR | 208622_s_at | PIP5K1C | 212518_at |
| EZR | 208623_s_at | PLCB2 | 204046_at |
| EZR | 217230_at | PLCB2 | 210388_at |
| EZR | 217234_s_at | PLD1 | 1557126_a_at |
| FES | 205418_at | PLD1 | 177_at |
| FLT1 | 204406_at | PLD1 | 205203_at |
| FLT1 | 210287_s_at | PLD1 | 215723_s_at |
| FLT1 | 222033_s_at | PLD1 | 215724_at |
| FLT1 | 226497_s_at | PLD1 | 226636_at |
| FLT1 | 226498_at | PLD1 | 232530_at |
| FLT1 | 232809_s_at | PLPP6 | 227385_at |
| FOS | 209189_at | PMAIP1 | 204285_s_at |
| FPR1 | 205118_at | PMAIP1 | 204286_s_at |
| FPR1 | 205119_s_at | PPP1CB | 201407_s_at |
| FPR2 | 210772_at | PPP1CB | 201408_at |
| FPR2 | 210773_s_at | PPP1CB | 201409_s_at |
| GATA1 | 1555590_a_at | PPP1CB | 228222_at |
| GATA1 | 210446_at | PPP1R12A | 201602_s_at |
| GNAI1 | 209576_at | PPP1R12A | 201603_at |
| GNAI1 | 227692_at | PPP1R12A | 201604_s_at |
| GNAI2 | 201040_at | PREX1 | 224909_s_at |
| GNAI2 | 215996_at | PREX1 | 224925_at |
| GNAI2 | 217271_at | PRKCA | 1560074_at |
| GNAI3 | 201179_s_at | PRKCA | 206923_at |
| GNAI3 | 201180_s_at | PRKCA | 213093_at |
| GNAI3 | 201181_at | PRKCA | 215194_at |
| GNAO1 | 204762_s_at | PRKCA | 215195_at |
| GNAO1 | 204763_s_at | PRKCB | 207957_s_at |
| GNAO1 | 215912_at | PRKCB | 209685_s_at |
| GNAO1 | 231951_at | PRKCB | 227817_at |
| GNAZ | 204993_at | PRKCB | 227824_at |
| GNB1 | 200744_s_at | PRKCB | 228795_at |
| GNB1 | 200745_s_at | PRKCB | 230437_s_at |
| GNB1 | 200746_s_at | PRKCD | 202545_at |
| GNB2 | 200852_x_at | PRKCE | 206248_at |
| GNB3 | 206047_at | PRKCE | 226101_at |
| GNB4 | 223487_x_at | PRKCE | 234089_at |
| GNB4 | 223488_s_at | PRKCE | 236459_at |
| GNB4 | 225710_at | PRKCE | 239011_at |
| GNB5 | 1554346_at | PRKCG | 206270_at |
| GNB5 | 204000_at | PRKCG | 236195_x_at |
| GNB5 | 207124_s_at | PRKCH | 206099_at |

| Gene | Probe ID | Gene | Probe ID |
|---|---|---|---|
| GNB5 | 211871_x_at | PRKCH | 218764_at |
| GNB5 | 242404_at | PRKCH | 230124_at |
| GNG10 | 201921_at | PRKCI | 209677_at |
| GNG11 | 204115_at | PRKCI | 209678_s_at |
| GNG11 | 239942_at | PRKCI | 213518_at |
| GNG12 | 1555240_s_at | PRKCQ | 210038_at |
| GNG12 | 212294_at | PRKCQ | 210039_s_at |
| GNG12 | 222834_s_at | PRKCZ | 1569748_at |
| GNG13 | 220806_x_at | PRKCZ | 202178_at |
| GNG2 | 1555766_a_at | PRKD1 | 205880_at |
| GNG2 | 223943_s_at | PRKD1 | 217705_at |
| GNG2 | 224964_s_at | PRKD2 | 209282_at |
| GNG2 | 224965_at | PRKD2 | 241669_x_at |
| GNG3 | 222005_s_at | PRKD2 | 38269_at |
| GNG4 | 1555765_a_at | PRKD3 | 1554910_at |
| GNG4 | 1555867_at | PRKD3 | 211084_x_at |
| GNG4 | 1566513_a_at | PRKD3 | 218236_s_at |
| GNG4 | 205184_at | PRKD3 | 222565_s_at |
| GNG5 | 207157_s_at | PRKD3 | 242549_at |
| GNG7 | 206896_s_at | PRTN3 | 207341_at |
| GNG7 | 214227_at | PTAFR | 206278_at |
| GNG7 | 228831_s_at | PTAFR | 211661_x_at |
| GNG7 | 232043_at | PTAFR | 227184_at |
| GNG8 | 233416_at | PTGS2 | 1554997_a_at |
| GNG8 | 234284_at | PTGS2 | 204748_at |
| GNGT1 | 207166_at | PTPRC | 1552480_s_at |
| GNGT2 | 235139_at | PTPRC | 1569830_at |
| H1F0 | 208886_at | PTPRC | 207238_s_at |
| HSPA14 | 219212_at | PTPRC | 212587_s_at |
| HSPA14 | 226887_at | PTPRC | 212588_at |
| HSPA14 | 227650_at | PXN | 201087_at |
| HSPA1L | 210189_at | PXN | 211823_s_at |
| HSPA1L | 233694_at | RAC1 | 1567457_at |
| HSPA2 | 211538_s_at | RAC1 | 1567458_s_at |
| HSPA4 | 208814_at | RAC1 | 208640_at |
| HSPA4 | 208815_x_at | RAC1 | 208641_s_at |
| HSPA4 | 211015_s_at | RAC2 | 207419_s_at |
| HSPA4 | 211016_x_at | RAC2 | 213603_s_at |
| HSPA5 | 211936_at | RARA | 1565358_at |
| HSPA5 | 230031_at<br>117 at | RARA | 203749_s_at |
| HSPA6 | | RARA | 203750_s_at |
| HSPA6 | 213418_at | RARA | 211605_s_at |
| HSPA8<br>HSPA8 | 208687_x_at<br>210338_s_at | RARA<br>REL | 216300_x_at<br>206035_at |
| HSPA8 | 221891_x_at | REL | 206035_at 206036_s_at |
| HSPA8 | 224187_x_at | REL | 228812_at |
| HSPA9 | 200690_at | REL | 235242_at |
| HSPA9 | 200691_s_at | REL | 239486_at |
| HSPA9 | 200692 s at | RELA | 201783_s_at |
| HSPA9 | 232200 at | RELA | 209878_s_at |
| ICAM1 | 202637_s_at | RELA | 230202_at |
| ICAM1 | 202638_s_at | RELB | 205205_at |
| ICAM1 | 215485 s at | RXRA | 202426_s_at |
| ICAM2 | 204683 at | RXRA | 202420_s_at |
| 10/11/12 | 20 1000_at | IVIIVI | 102 1 10_0_at |

| Gene | Probe ID | Gene | Probe ID |
|--------|--------------|----------|--------------|
| ICAM2 | 213620_s_at | S100P | 204351_at |
| IFITM1 | 201601_x_at | SELL | 204563_at |
| IFITM1 | 214022_s_at | SOCS3 | 206359_at |
| IL1B | 205067_at | SOCS3 | 206360_s_at |
| IL1B | 39402_at | SOCS3 | 214105_at |
| IL1R1 | 202948_at | SOCS3 | 227697_at |
| IL1R1 | 215561_s_at | SPI1 | 205312_at |
| ITGAL | 1554240_a_at | SPTBN1 | 200671_s_at |
| ITGAL | 213475_s_at | SPTBN1 | 200672_x_at |
| ITGAM | 205785_at | SPTBN1 | 212071_s_at |
| ITGAM | 205786_s_at | SPTBN1 | 213914_s_at |
| ITGB2 | 1555349_a_at | SPTBN1 | 214856_at |
| ITGB2 | 202803_s_at | SPTBN1 | 215918_s_at |
| ITGB2 | 236988_x_at | SPTBN1 | 226342_at |
| ITPR1 | 1562373_at | SPTBN1 | 226765_at |
| ITPR1 | 203710_at | SPTBN1 | 228246_s_at |
| ITPR1 | 211323_s_at | SPTBN1 | 230540_at |
| ITPR1 | 216944_s_at | SPTBN1 | 242220_at |
| ITPR1 | 240052_at | SSH2 | 1554114_s_at |
| ITPR2 | 202660_at | SSH2 | 1555423_at |
| ITPR2 | 202661_at | SSH2 | 1555425_x_at |
| ITPR2 | 202662_s_at | SSH2 | 1560306_at |
| ITPR2 | 211360_s_at | SSH2 | 226080_at |
| ITPR3 | 201187_s_at | STAT3 | 208991_at |
| ITPR3 | 201188_s_at | STAT3 | 208992_s_at |
| ITPR3 | 201189_s_at | STAT3 | 225289_at |
| ITPR3 | 239542_at | STAT3 | 243213_at |
| JAK1 | 1552610_a_at | STAT5A | 203010_at |
| JAK1 | 1552611_a_at | STAT5B | 1555086_at |
| JAK1 | 201648_at | STAT5B | 1555088_x_at |
| JAK1 | 239695_at | STAT5B | 205026_at |
| JAK1 | 240613_at | STAT5B | 212549_at |
| JAK2 | 1562031_at | STAT5B | 212550_at |
| JAK2 | 205841_at | SYAP1 | 225154_at |
| JAK2 | 205842_s_at | TAC1 | 206552_s_at |
| JUN | 201464_x_at | TACR1 | 208048_at |
| JUN | 201465_s_at | TACR1 | 208049_s_at |
| JUN | 201466_s_at | TACR1 | 210637_at |
| JUN | 213281_at | TACR1 | 230908_at |
| KLK1 | 216699_s_at | TARP | 211144_x_at |
| KLK10 | 209792_s_at | TARP | 216920_s_at |
| KLK10 | 215808_at | TARP | 217381_s_at |
| KLK11 | 205470_s_at | TBC1D22A | 209650_s_at |
| KLK12 | 220782_x_at | TBC1D22A | 210144_at |
| KLK12 | 233586_s_at | TBC1D22A | 33778_at |
| KLK12 | 234316_x_at | TLN1 | 203254_s_at |
| KLK13 | 205783_at | TLN1 | 232763_at |
| KLK13 | 216670_at | TLN1 | 236132_at |
| KLK13 | 217315_s_at | TLN2 | 212701_at |
| KLK14 | 220573_at | TLN2 | 212703_at |
| KLK15 | 221462_x_at | TLN2 | 232625_at |
| KLK15 | 233477_at | TLR10 | 223750_s_at |
| KLK15 | 234495_at | TLR10 | 223751_x_at |
| KLK15 | 234966_at | TLR2 | 204924_at |

| Gene | Probe ID | Gene | Probe ID |
|------|--------------|----------|--------------|
| KLK2 | 1555545_at | TLR4 | 1552798_a_at |
| KLK2 | 209854_s_at | TLR4 | 221060_s_at |
| KLK2 | 209855_s_at | TLR4 | 224341_x_at |
| KLK2 | 210339_s_at | TLR4 | 232068_s_at |
| KLK3 | 204582_s_at | TNF | 1563357_at |
| KLK3 | 204583_x_at | TNF | 207113_s_at |
| KLK3 | 231629_x_at | TNFRSF1A | 207643_s_at |
| KLK4 | 1555697_at | TNFRSF1B | 203508_at |
| KLK4 | 1555737_a_at | TREML2 | 219748_at |
| KLK4 | 224062_x_at | TTPAL | 219633_at |
| KLK4 | 231782_s_at | TTPAL | 228031_at |
| KLK4 | 233854_x_at | VAV1 | 206219_s_at |
| KLK5 | 222242_s_at | VCL | 200930_s_at |
| KLK6 | 204733_at | VCL | 200931_s_at |
| KLK7 | 205778_at | VPS37B | 221704_s_at |

201928

# 13.7. Appendix 7: Reporting Standards for Missing Data

## 13.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as Subject whom have completed their final visit (day 84).</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 13.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> </li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| PD | <ul> <li>Any values below the Lower Limit of Quantification (LLQ) will be assigned a value of ½ LLQ for display purposes in Figures and for computation of summary statistics. Any values above the Upper Limit of Quantification (ULQ) will be assigned to the ULQ for display purposes in Figures and for computation of summary statistics. If multiple LLQ and /or ULQ values are available per assay (for example if multiple runs with different standard curves are utilised) then the LLQ and/or ULQ value used for the above imputation shall be the minimum of the available LLQs and/or the maximum of the ULQs. Where biomarker concentrations are from an assay of an increased dilution factor the LLQ and ULQ will be multiplied by this factor.</li> <li>If the number of LLQ (and/or ULQ) values is large for an individual biomarker then an alternative analysis method, such as TOBIT analysis, may be required. "Large" is hard to define prospectively and may depend upon the dataset in question. Any such methodology will be documented in the statistical contributions to the study report.</li> <li>Imputed values will be used in tables and figures, unless the proportion of imputed values at a given time point is large, in which case the summary statistics may not be presented for that time point and/or alternative actions will be taken and documented in the study report.</li> <li>Where values are imputed, the number of such imputations will be included as a summary statistic in the relevant summary tables.</li> </ul> |
| HRCT | <ul> <li>No missing data imputation methods will be used.</li> <li>Note that for the HRCT data, there may be instances such that measurements from a particular Lobe cannot be distinguished between another Lobe, for example the iVlobe may be measured from both the LLL and LUL lobes. In such a case, the Lobe will be denoted as LLL + LUL. Therefore, for the statistical analysis purpose, since analysis is performed on a lobar level, the LLL and LUL Lobes will be set to missing and will</li> </ul> |

201928

| Element | Reporting Detail | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | efore not be included in the analysis. Below is a table of all possible scenarios, re the data is set to missing and not used in the statistical analysis: | | | | | | |
| | | | | Lobes | | | Label | |
| | RUL RML RLL LUL LLL | | | | Labei | | | |
| | | Χ | Χ | | | | RUL + RML | |
| | | | Х | Х | | | RML + RLL | |
| | | x x RUL + RLL | | | | | | |
| | | Χ | Х | Х | | | RUL + RML + RLL | |
| | | | | | Х | Х | LUL + LLL | |
| | | | | | | | | - |

# 13.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be<br/>recorded for AE start and end dates; that is, the day of the month may be missing. In<br/>such a case, the following conventions will be applied for calculating the time to onset<br/>and the duration of the event:</li> </ul> |
| | <ul> <li>Missing Start Day: First of the month will be used unless this is before the start<br/>date of study treatment; in this case the study treatment start date will be used and<br/>hence the event is considered On-treatment as per Appendix 4: Study Phases and<br/>Treatment Emergent Adverse Events.</li> </ul> |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop<br/>date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
| Concomitant<br>Medications/ | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |
| Medical<br>History | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be<br/>used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent<br/>on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

201928

# 13.8. Appendix 8: Values of Potential Clinical Importance

# 13.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Hematocrit | Ratio of | Male | | 0.54 |
| Петнагості | 1 | Female | | 0.54 |
| Haemoglobin | g/L | Male | | 180 |
| Haemoglobin | | Female | | 180 |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

201928

## 13.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-----------------------|-------|------------------------|-----------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 500 [1] |
| Absolute PR Interval | msec | < 110 [1] | > 220 [2] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [2] |

## NOTES:

# 13.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

<sup>[1]</sup> An upper limit of 450 would represent standard ECG values of PCI for HV studies, this has been extended to 500 as often with exacerbations the treatment can result in a short term prolongation of QTc up to 500.

<sup>[2]</sup> Represent standard ECG values of PCI for HV studies

201928

# 13.9. Appendix 9: Abbreviations & Trade Marks

## 13.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| A&R | Analysis and Reporting |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| AT | Air Trapping Score (% of iVlobe) |
| BVD | Blood Vessel Density (% of iVlobe) |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CENTRAL | Central lung region |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CT | Computed tomography |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| Diameter | Diameter |
| DISTAL | Distal lung region |
| DLco | Diffusion capacity |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FEV <sub>1</sub> | Forced expiratory volume in 1 second |
| FRI | Functional respiratory imaging |
| FRC | Functional residual capacity |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| HRCT | High Resolution Computed Tomography |
| IA | Interim Analysis |
| IALD | Internal Airflow Lobar Distribution |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IL-8 | Interleukin 8 |
| IL-6 | Interleukin 6 |

| Abbreviation | Description |
|---|---|
| IMMS | International Modules Management System |
| IP | Investigational Product |
| iRaw | Imaging Airway Resistance |
| ITT | Intent-To-Treat |
| iVlobe | Lobar Volume |
| iVlobepred | Percent Predicted Lobar Volume |
| iVaw | Imaging Airway Volume |
| iVaww | Airway Wall Volume |
| LAS | Low Attenuation Score (% of iVlobe) |
| Length | Length |
| LL | Lung, lower lobes |
| LLL | Lung, left lower lobe |
| LOC | Last Observation Carries Forward |
| LUL | Lung, left upper lobe |
| LUL+LLL | Lung, left upper and lower lobe |
| MMP9 | 0 11 |
| MMRC | Matrix metallopeptidase 9 Modified Medical Research Council |
| MMRM | |
| | Mixed Model Repeated Measures |
| NQ | Non-quantifiable |
| OTU | Operational Taxonomic Unit |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PEF | peak expiratory flow |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| qPCR | Quantitative polymerase chain reaction |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RLL | Lung, right lower lobe |
| RML | Lung, right middle lobe |
| RML+RLL | Lung, right middle and lower lobe |
| RUL | Lung, right upper lobe |
| RUL+RLL | Lung, right upper and lower lobe |
| RUL+RML | Lung, right upper and middle lobe |
| RUL+RML+RLL | Lung, right upper, middle and lower lobe |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| sGaw | Specific conductance |
| siRaw | Specific Imaging Airway Resistance |

201928

| Abbreviation | Description |
|--------------|--------------------------------|
| siVaw | Specific Imaging Airway Volume |
| siVaww | Specific Airway Wall Volume |
| SoC | Standard of Care |
| SOP | Standard Operation Procedure |
| sRaw | Specific Resistance |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TLC | Total lung capacity |
| TNFα | Tumor necrosis factor alpha |
| TOTAL | Total lung region |
| TRACHEA | Trachea |
| UL | Lung, upper lobes |

# 13.9.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| ELLIPTA |
| HARP |
| RAMOS NG |
| RANDALL NG |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| FluidDA |
| Quest |
| SAS |
| WinNonlin |

201928

# 13.10. Appendix 10: List of Data Displays

# 13.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|---------|
| Study Population | 1.1 to 1.17 | N/A |
| Efficacy | 2.1 to 2.68 | 2.1 |
| Safety | 3.1 to 3.20 | N/A |
| Pharmacokinetic | 4.1 to 4.4 | 4.1 |
| Pharmacodynamic and / or Biomarker | 6.1 to 6.21 | 6.1 |
| Section | List | ings |
| ICH Listings | 1 to 34 | |
| Other Listings | 35 t | o 49 |

## 13.10.2. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

201928

## 13.10.3. Study Population Tables

| Study | Study Population Tables | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | | | | |
| Subjec | Subject Disposition | | | | | | | | |
| 1.1. | All Subject | ES1 | Summary of Subject Disposition | ICH E3, FDAAA, EudraCT | SAC | | | | |
| 1.2. | All Subject | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC | | | | |
| 1.3. | APE | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC | | | | |
| 1.4. | All Subject | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations | SAC | | | | |
| Protoc | Protocol Deviation | | | | | | | | |
| 1.5. | All Subject | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC | | | | |
| Popula | Population Analysed | | | | | | | | |
| 1.6. | APE | SP1 | Summary of Study Populations | IDSL | SAC | | | | |
| 1.7. | All Subject | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | SAC | | | | |
| Demog | raphic and Bas | eline Characteris | tics | | | | | | |
| 1.8. | All Subject | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC | | | | |
| 1.9. | APE | DM11 | Summary of Age Ranges | EudraCT | SAC | | | | |
| 1.10. | All Subject | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC | | | | |
| 1.11. | All Subject | DM6 | Summary of Race and Racial Combinations Details | | SAC | | | | |
| 1.12. | All Subject | PII116678/final/<br>Table 2.109 | Summary of Index Exacerbation Severity | | | | | | |
| Study F | Study Population Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | | | |
| Prior a | nd Concomitan | t Medications | | | | | | |
| 1.13. | All Subject | MH1 | Summary of Current Medical Conditions | ICH E3 | SAC | | | |
| 1.14. | All Subject | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC | | | |
| 1.15. | All Subject | CM1 | Summary of Prior Medications | ICH E3 | SAC | | | |
| 1.16. | All Subject | CM1 | Summary of Concomitant Medications | ICH E3 | SAC | | | |
| Exposu | ire and Treatme | ent Compliance | | | | | | |
| 1.17. | All Subject | EX1 | Summary of Exposure to Study Treatment | ICH E3 Include Daily Dose, Cumulative does and Days on study drug per template. | SAC | | | |

201928

# 13.10.4. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| HRCTI | maging Endpo | ints | | | |
| 2.1. | All subjects | PII116678/ final/<br>Table 2.1 | Summary of iVaw (mL) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used | SAC |
| 2.2. | All subjects | PII116678/ final/<br>Table 2.2 | Summary of iVaw (mL) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.3. | All subjects | PII116678/ final/<br>Table 2.3 | Summary of iVaw (mL) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used | SAC |
| 2.4. | All subjects | PII116678/ final/<br>Table 2.4 | Summary of iVaw (mL) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.5. | All subjects | PII116678/ final/<br>Table 2.9 | Summary of siVaw (mL/L) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used | SAC |
| 2.6. | All subjects | PII116678/ final/<br>Table 2.10 | Summary of siVaw (mL/L) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.7. | All subjects | PII116678/final/<br>Table 2.11 | Summary of siVaw (mL/L) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used | SAC |
| 2.8. | All subjects | PII116678/final/<br>Table 2.12 | Summary of siVaw (mL/L) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.9. | All subjects | PII116678/final/<br>Table 2.17 | Summary of iRaw (kPa*s/L) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No longitudinal endpoints Footnote any transformations used | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.10. | All subjects | PII116678/final/<br>Table 2.18 | Summary of iRaw (kPa*s/L) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No longitudinal endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.11. | All subjects | PII116678/final/<br>Table 2.19 | Summary of iRaw (kPa*s/L) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page No longitudinal endpoints Footnote any transformations used | SAC |
| 2.12. | All subjects | PII116678/final/<br>Table 2.20 | Summary of iRaw (kPa*s/L) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page No longitudinal endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.13. | All subjects | PII116678/final/<br>Table 2.25 | Summary of siRaw (kPa*s) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No longitudinal endpoints Footnote any transformations used | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.14. | All subjects | PII116678/final/<br>Table 2.26 | Summary of siRaw (kPa*s) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No longitudinal endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.15. | All subjects | PII116678/final/<br>Table 2.27 | Summary of siRaw (kPa*s) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page No longitudinal endpoints Footnote any transformations used | SAC |
| 2.16. | All subjects | PII116678/final/<br>Table 2.28 | Summary of siRaw (kPa*s) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page No longitudinal endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.17. | All subjects | PII116678/final/<br>Table 2.33 | Summary of iVlobe (L) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.18. | All subjects | PII116678/final/<br>Table 2.34 | Summary of iVlobe (L) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.19. | All subjects | PII116678/final/<br>Table 2.35 | Summary of iVlobe (L) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.20. | All subjects | PII116678/final/<br>Table 2.36 | Summary of iVlobe (L) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.21. | All subjects | PII116678/final/<br>Table 2.41 | Summary of Percent Predicted iVlobe (%) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Note in HARP to output (%) it may be necessary to input (%%) | SAC |
| 2.22. | All subjects | PII116678/final/<br>Table 2.42 | Summary of Percent Predicted iVlobe (%) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline Note in HARP to output (%) it may be necessary to input (%%) | SAC |
| 2.23. | All subjects | PII116678/final/<br>Table 2.43 | Summary of Percent Predicted iVlobe (%) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Note in HARP to output (%) it may be necessary to input (%%) | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.24. | All subjects | PII116678/final/<br>Table 2.44 | Summary of Percent Predicted iVlobe (%) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline Note in HARP to output (%) it may be necessary to input (%%) | SAC |
| 2.25. | All subjects | PII116678/final/<br>Table 2.49 | Summary of LAS (% of iVlobe) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.26. | All subjects | PII116678/final/<br>Table 2.50 | Summary of LAS (% of iVlobe) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.27. | All subjects | PII116678/final/<br>Table 2.51 | Summary of LAS (% of iVlobe) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.28. | All subjects | PII116678/final/<br>Table 2.52 | Summary of LAS (% of iVlobe) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.29. | All subjects | PII116678/final/<br>Table 2.55 | Summary of IALD (%) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.30. | All subjects | PII116678/final/<br>Table 2.56 | Summary of IALD (%) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.31. | All subjects | PII116678/final/<br>Table 2.57 | Summary of IALD (%) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central, Distal and Total do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.32. | All subjects | PII116678/final/<br>Table 2.58 | Summary of IALD (%) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central, Distal and Total do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.33. | All subjects | PII116678/final/<br>Table 2.61 | Summary of AT (% of iVlobe) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.34. | All subjects | PII116678/final/<br>Table 2.62 | Summary of AT (% of iVlobe) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.35. | All subjects | PII116678/final/<br>Table 2.63 | Summary of AT (% of iVlobe) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.36. | All subjects | PII116678/final/<br>Table 2.64 | Summary of AT (% of iVlobe) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.37. | All subjects | PII116678/final/<br>Table 2.67 | Summary of BVD (% of iVlobe) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.38. | All subjects | PII116678/final/<br>Table 2.68 | Summary of BVD (% of iVlobe) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.39. | All subjects | PII116678/final/<br>Table 2.69 | Summary of BVD (% of iVlobe) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used | SAC |
| 2.40. | All subjects | PII116678/final/<br>Table 2.70 | Summary of BVD (% of iVlobe) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Regions Central and Distal do not exist No Scan Trimming endpoints Footnote any transformations used Footnote baseline | SAC |
| 2.41. | All subjects | PII116678/final/<br>Table 2.73 | Summary of iVaww (mL) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used | SAC |
| 2.42. | All subjects | PII116678/final/<br>Table 2.74 | Summary of iVaww (mL) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used Footnote baseline | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.43. | All subjects | PII116678/final/<br>Table 2.75 | Summary of iVaww (mL) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used | SAC |
| 2.44. | All subjects | PII116678/final/<br>Table 2.76 | Summary of iVaww (mL) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.45. | All subjects | PII116678/final/<br>Table 2.79 | Summary of siVaww (mL/L) (Absolute), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used | SAC |
| 2.46. | All subjects | PII116678/final/<br>Table 2.80 | Summary of siVaww (mL/L) (Change from Baseline), for Individual Lobes | Ensure no overlapping information across pages for each Lobe, hence if required start each Lobe on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.47. | All subjects | PII116678/final/<br>Table 2.81 | Summary of siVaww (mL/L) (Absolute), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.48. | All subjects | PII116678/final/<br>Table 2.82 | Summary of siVaww (mL/L) (Change from Baseline), for Individual Regions | Ensure no overlapping information across pages for each Region, hence if required start each Region on a separate page Footnote any transformations used Footnote baseline | SAC |
| 2.49. | All subjects | PII116678/final/<br>Table 2.85 | Summary of Trachea Length (mm), Diameter (mm) and Length /Diameter (mm/mm) (Absolute) | Footnote any transformations used | SAC |
| 2.50. | All subjects | PII116678/final/<br>Table 2.86 | Summary of Trachea Length (mm), Diameter (mm) and Length /Diameter (mm/mm) (Change from Baseline) | Footnote any transformations used Footnote baseline | SAC |
| 2.51. | All subjects | PII116678/final/<br>Table 2.14 | Summary of Statistical Analysis for siVaw (mL/L), for Individual Lobes at FRC using Untrimmed Data | Ensure no overlapping information across pages for each Lobe Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.52. | All subjects | PII116678/final/<br>Table 2.16 | Summary of Statistical Analysis for siVaw (mL/L), for Individual Regions at FRC using Untrimmed Data | Ensure no overlapping information across pages for each Lobe Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.53. | All subjects | Refer to:<br>PII116678/final/<br>Table 2.16<br>Note: there will<br>be less regions | Summary of Statistical Analysis for siVaw (mL/L), for Distal Region at FRC using Scan Trimmed Data | Ensure no overlapping information across pages for each Lobe Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.54. | All subjects | Refer to:<br>PII116678/final/<br>Table 2.29<br>Note: there will<br>be less regions | Summary of Statistical Analysis for siRaw (kPa*s), for Distal Region at FRC | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.55. | All subjects | Refer to: PII116678/final/ Table 2.54 Note: there will be less regions | Summary of Statistical Analysis for LAS (% of iVlobe), for Total Region at TLC | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.56. | All subjects | Refer to:<br>PII116678/final/<br>Table 2.60<br>Note: there will<br>be less regions | Summary of Statistical Analysis for IALD (%), for Upper and Lower Regions | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.57. | All subjects | Refer to:<br>PII116678/final/<br>Table 2.66<br>Note: there will<br>be less regions | Summary of Statistical Analysis for AT (% of iVlobe), for Total Region at FRC | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.58. | All subjects | Refer to:<br>PII116678/final/<br>Table 2.72<br>Note: there will<br>be less regions | Summary of Statistical Analysis for BVD (% of iVlobe), for Total Region at TLC | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.59. | All subjects | Refer to:<br>PII116678/final/<br>Table 2.84<br>Note: there will<br>be less regions | Summary of Statistical Analysis for siVaww (mL/L), for Distal Region at TLC using Untrimmed Data | Ensure no overlapping information across pages for each Region No longitudinal endpoints Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| Lung F | unction | | | | |
| 2.60. | All subjects | PII115119/<br>Part_A /Table<br>3.18 | Summary of FEV1 (ml) and FVC (ml) (Absolute Values) | Summaries by Visit<br>Footnote any transformations used | SAC |
| 2.61. | All subjects | PII115119/<br>Part_A /Table<br>3.19 | Summary of FEV1 (ml) and FVC (ml) (Change from Baseline) | Summaries by Visit Footnote any transformations used Footnote Baseline | SAC |
| 2.62. | All subjects | PII116678/ final<br>/Table 2.88 | Summary of Statistical Analysis for FEV1 (ml) (Change from Baseline) | Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| 2.63. | All subjects | PII116678/<br>postcsr_2017_01<br>/Table 2.1 | Sub Group Analysis: by Index Exacerbation Severity<br>Summary of Statistical Analysis for FEV1 (ml) (Change from<br>Baseline) | Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.64. | All subjects | PII116678/ final<br>/Table 2.88 | Summary of Statistical Analysis for FVC (ml) (Change from Baseline) | Footnote to include the statistical analysis conducted, including covariates, co-variance matrix and prior assumptions. Footnote any transformations used Footnote baseline | SAC |
| Relief I | Medication | | | | |
| 2.65. | All subjects | Refer to<br>programming<br>notes | Summary of Rescue Medication Free Days | Use the standard tu_sumstatsinrows to summarise Rescue Medication Free days by time period and treatment. Include columns for time period, treatment, N, n, mean, 95% CI, SD, median, min and max | SAC |
| 2.66. | All subjects | Refer to programming notes | Summary of Mean Number of Occasions of Rescue Use per<br>Day | Use the standard tu_sumstatsinrows to summarise Mean Number of Occasions of Rescue Use per Day by time period and treatment. Include columns for timeperiod, treatment, N, n, mean, 95% CI, SD, median, min and max | SAC |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Exacer | bations | | | | |
| 2.67. | All subjects | Refer to PII116678/ final /Table 2.97 And programming notes | Summary of Investigator Defined Exacerbations | Update rows to be consistent with data i.e. include 6, 7, etc exacerbations as appropriate | SAC |
| 2.68. | All subjects | Refer to PII116678/ final /Table 2.116 And programming notes | Summary of Concomitant Medication Defined Exacerbations | Update rows to be consistent with data i.e. include 6, 7, etc exacerbations as appropriate | SAC |

201928

# 13.10.5. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Lung Fı | unction | | | | |
| 2.1. | All subjects | Refer to PII116678/final/ Table 2.2 but update the number of plots based on the data as appropriate | Summary of PEF (morning) | X-axis to contain each Day, with<br>Means and confidence intervals,<br>grouped by Treatment.<br>Include baseline as a subheading<br>per example shell | SAC |

201928

# 13.10.6. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events (AEs) | | | | |
| 3.1. | All Subject | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.2. | All Subject | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | ICH E3 | SAC |
| 3.3. | All Subject | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3<br>Include flag for serious | SAC |
| 3.4. | All Subject | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT | SAC |
| Serious | and Other Sig | nificant Adverse I | Events | | |
| 3.5. | All Subject | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC |
| 3.6. | All Subject | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | IDSL | SAC |
| Labora | tory: Chemistry | / | | | |
| 3.7. | All Subject | LB1 | Summary of Chemistry | ICH E3 | SAC |
| 3.8. | All Subject | LB15 | Summary of Worst Case Emergent Laboratory Chemistry<br>Results Relative to Normal Range | | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Labora | tory: Hematolo | gy | | | |
| 3.9. | All Subject | LB1 | Summary of Hematology | ICH E3 | SAC |
| 3.10. | All Subject | LB15 | Summary of Worst Case Emergent Laboratory Hematology Results Relative to Normal Range | | SAC |
| Labora | tory: Urinalysis | <b>3</b> | | | · |
| 3.11. | All Subject | LB1 | Summary of Urine Concentration | ICH E3 | SAC |
| 3.12. | All Subject | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | · |
| 3.13. | All Subject | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC |
| 3.14. | All Subject | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC |
| ECG | | | | | · |
| 3.15. | All Subject | EG1 | Summary of ECG Findings | IDSL | SAC |
| 3.16. | All Subject | EG2 | Summary of ECG Values by Visit | | SAC |
| 3.17. | All Subject | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC |
| Vital Si | gns | | | | |
| 3.18. | All Subject | VS1 | Summary of Vital Signs | | SAC |
| 3.19. | All Subject | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3<br>Includes Baseline Values | SAC |
| 3.20. | All Subject | VS7 | Summary of Emergent Vital Sign Results by Potential Clinical Importance (PCI) Criteria | | SAC |

201928

## 13.10.7. Pharmacokinetic Tables

| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Plasma | Concentration | n | | | |
| 4.1 | DIV | PK01 | Summary of Plasma Nemiralisib Pharmacokinetic Concentration | All visits/timepoints, include a column for visit. Summarise PK data on original scale. Produce 95% CIs Note: Use the separate NEMI | CAC |
| 4.1. | PK | PII116678/final/Table<br>4.1 | – Time Ďata (ng/mL) | Diskus and NEMI ELLIPTA treatment groups Excluding the two subjects who were noted to not comply with inhalation instructions – include | SAC |

| Pharma | acokinetic: Tak | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| | | | | All visits/timepoints, include a column for visit. Summarise PK data on original scale. Produce 95% CIs | |
| 4.2. | PK | PK01<br>PII116678/final/Table<br>4.2 | Summary of Plasma Nemiralisib Pharmacokinetic Concentration – Time Data (ng/mL) Including All PK Concentrations Analysed | Note: Use the separate NEMI<br>Diskus and NEMI ELLIPTA<br>treatment groups | SAC |
| | | | | Including the two subjects who were noted to not comply with inhalation instructions – include footnote | |
| | | | | All visits/timepoints, include a column for visit and planned time. Summarise PK data on original scale. Produce n, No. imputed, geometric mean and corresponding 95% Cis SD Logs and %CVb | |
| 4.3. | PK | PII116678/final/Table<br>4.3 | ble Summary of Log-Transformed Plasma Nemiralisib Pharmacokinetic Concentration – Time Data (ng/mL) | Note: Use the separate NEMI<br>Diskus and NEMI ELLIPTA<br>treatment groups | SAC |
| | | | | Excluding the two subjects who were noted to not comply with inhalation instructions – include footnote | |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.4. | PK | PII116678/final/Table<br>4.4 | Summary of Log-Transformed Plasma Nemiralisib<br>Pharmacokinetic Concentration – Time Data (ng/mL)<br>Including All PK Concentrations Analysed | All visits/timepoints, include a column for visit and planned time. Summarise PK data on original scale. Produce n, No. imputed, geometric mean and corresponding 95% Cis SD Logs and %CVb Note: Use the separate NEMI Diskus and NEMI ELLIPTA treatment groups Including the two subjects who were noted to not comply with inhalation instructions – include footnote | SAC |

201928

# 13.10.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Plasma | Concentration | i | | | |
| 4.1. | PK | Refer to PII116678/ final/ Figure 4.1 But include additional timepoints per programming notes | Box and Whisker Plot of Plasma Concentration | Two figures to be created: 1st: Plasma Concentration at Day 1 (5 min and 24 hours post-dose) and Day 12 2nd: Plasma Concentration at Day 12, Day 28, Day 56 and Day 84 Note: Use the separate NEMI Diskus and NEMI ELLIPTA | SAC |

201928

# 13.10.9. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| MRNa | • | | | | |
| 6.1. | All subjects | PII115119/<br>Part A/<br>Listing 40 | Summary of Statistical Analysis of mRNA Transcriptome in Induced Sputum (Selected Probe Sets Related to Neutrophil Function) | Summarise fold changes, 95% CI and p-values. Rank by p-value and fold change within timepoint. | SAC |
| 6.2. | All subjects | PII115119/<br>Part A/<br>Listing 40 | Summary of Statistical Analysis of mRNA Transcriptome in Blood (All Probe Sets) | Summarise fold changes, 95% CI and p-values. Rank by p-value and fold change within timepoint. | SAC |
| 6.3. | All subjects | PII115119/<br>Part A/<br>Listing 40 | Summary of Additional Statistical Analysis of mRNA<br>Transcriptome in Induced Sputum (All Probe Sets) | Summarise fold changes, 95% CI and p-values. Rank by p-value and fold change within timepoint. | SAC |
| Cell Co | unt Data and P | MN Differentials | | | |
| 6.4. | All subjects | PII115119/<br>Part A/Table<br>5.7 | Summary Statistics (Absolute): Total Cell Count Data in Sputum by Treatment and Time. | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.5. | All subjects | PII115119/<br>Part A/Table<br>5.8 | Summary Statistics (Change from Baseline): Total Cell Count Data in Sputum by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.6. | All subjects | PII115119/<br>Part A/Table<br>5.9 | Summary Statistics (Absolute): PMNs Differentials in Sputum by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.7. | All subjects | PII115119/<br>Part A/Table<br>5.10 | Summary Statistics (Change from Baseline): PMNs Differentials in Sputum by Treatment and Time | Appropriate transformation should<br>be used prior to summarising data.<br>Ensure transformation is clearly<br>documented and update column<br>labels as appropriate | SAC |
| 6.8. | All subjects | PII115119/<br>Part A/Table<br>5.11 | Summary Statistics (Absolute): Total Cell Count Data in Blood by Treatment and Time. | Appropriate transformation should<br>be used prior to summarising data.<br>Ensure transformation is clearly<br>documented and update column<br>labels as appropriate | SAC |
| 6.9. | All subjects | PII115119/<br>Part A/Table<br>5.12 | Summary Statistics (Change from Baseline): Total Cell Count Data in Blood by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.10. | All subjects | PII115119/<br>Part A/Table<br>5.13 | Summary Statistics (Absolute): PMNs Differentials in Blood by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |

| Pharma | codynamic and | d Biomarker: Tabl | es | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.11. | All subjects | PII115119/<br>Part A/Table<br>5.14 | Summary Statistics (Change from Baseline): PMNs Differentials in Blood by Treatment and Time | Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| Inflamn | natory Biomark | ers | | | |
| 6.12. | All subjects | PII115119/<br>Part A/Table<br>5.17 | Summary Statistics (Absolute): Inflammatory Biomarkers by Treatment and Time | It is expected that no transformation will be required for this Table (6.12) and a log transformation will be required for Table 6.14. However appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.13. | All subjects | PII115119/<br>Part A/Table<br>5.18 | Summary Statistics (Change from Baseline): Inflammatory Biomarkers by Treatment and Time | It is expected that no transformation will be required for this Table (6.13) and a log transformation will be required for Table 6.15. However appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |

| Pharma | acodynamic and | d Biomarker: Tabl | es | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.14. | All subjects | PII115119/<br>Part A/Table<br>5.19 | Summary Statistics (Log-Transformed Absolute) Inflammatory Biomarkers by Treatment and Time | It is expected that no transformation will be required for Table 6.12 and a log transformation will be required for this Table (6.14). However appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.15. | All subjects | PII115119/<br>Part A/Table<br>5.20 | Summary Statistics (Log-Transformed Change from Baseline)<br>Inflammatory Biomarkers by Treatment and Time | It is expected that no transformation will be required for Table 6.13 and a log transformation will be required for this Table (6.15). However appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| Microb | iome (16S rRNA | A) and qPCR | | | |
| 6.16. | All subjects | PD4<br>and Refer to<br>programming<br>notes | Summary Statistics (Absolute): Microbiome (16S rRNA) Relative Abundance by Treatment and Time | If Data available Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.17. | All subjects | PD4<br>and Refer to<br>programming<br>notes | Summary Statistics (Percentage Change from Baseline): Microbiome (16S rRNA) Relative Abundance by Treatment and Time | If Data available. Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.18. | All subjects | PII115119/<br>Part A/Table<br>5.24 | Summary Statistics (Absolute): qPCR delta Ct by Treatment and Time | If Data available. Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| 6.19. | All subjects | PII115119/<br>Part A/Table<br>5.25 | Summary Statistics (Log-Transformed Absolute): qPCR fold change by Treatment and Time | If Data available. Appropriate transformation should be used prior to summarising data. Ensure transformation is clearly documented and update column labels as appropriate | SAC |
| Bacteri | al Culture | | | | |
| 6.20. | All subjects | PII115119/<br>Part A/Table<br>5.26 | Frequency Table of Bacterial Culture (Presence) by Treatment and Time | | SAC |

201928

# 13.10.10. ICH Listings

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1. | APE | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | All Subjects | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | All Subjects | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 4. | All Subjects | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| 5. | All Subjects | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 6. | All Subjects | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | All Subjects | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 8. | APE | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | All Subjects | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 10. | All Subjects | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | All Subjects | CM3 | Listing of Concomitant Medications | IDSL | SAC |
| Exposi | ure and Treatme | ent Compliance | | | |
| 12. | All Subjects | EX3 | Listing of Exposure Data | ICH E3 | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events | | | | • |
| 13. | All Subjects | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| 14. | All Subjects | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 15. | All Subjects | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Serious | and Other Sig | nificant Adverse I | Events | | • |
| 16. | All Subjects | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| 17. | All Subjects | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| 18. | All Subjects | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 19. | All Subjects | AE8 | Listing of Adverse Events Leading to Withdrawal from Study or<br>Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | <u> </u> |
| 20. | All Subjects | MH2 | Listing of Medical Conditions for Participants with Liver Stopping<br>Events | IDSL | SAC |
| 21. | All Subjects | SU2 | Listing of Substance Use for Participants with Liver Stopping<br>Events | IDSL | SAC |
| 22. | All Subjects | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC |
| 23. | All Subjects | LIVER7 | Listing of Liver Biopsy Details | | SAC |
| 24. | All Subjects | LIVER8 | Listing of Liver Imaging Details | | SAC |
| All Lab | oratory | | | | |
| 25. | All Subjects | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 26. | All Subjects | LB5 | Listing of Laboratory Values of Potential Clinical Importance | | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 27. | All Subjects | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| 28. | All Subjects | UR2A | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| ECG | | | | | |
| 29. | All Subjects | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 30. | All Subjects | EG3 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC |
| 31. | All Subjects | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |
| 32. | All Subjects | EG5 | Listing of Abnormal ECG Findings | IDSL | SAC |
| Vital Si | gns | | | | |
| 33. | All Subjects | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 34. | All Subjects | VS4 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC |

201928

# 13.10.11. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Demog | Demography and Baseline Characteristics | | | | |
| 35. | All Subjects | FH1 | Summary of Family History of Cardiovascular Risk Factors | | SAC |
| 36. | All Subjects | Refer to<br>Programming<br>notes | COPD Disease duration and Exacerbation Duration | Include investigator ID, subject ID, country, treatment group, COPD Disease Duration (in years and months) and Exacerbation History (number requiring oral/systemic corticosteroids and/or antibiotics and number requiring hospitalisation) as columns | SAC |
| 37. | All Subjects | PREG1a | Listing of Subjects Who Became Pregnant During the Study | Also indicate if the female partners of subjects became pregnant during the study | |
| Labs | | | | | |
| 38. | All Subjects | LB13 | Listing of Laboratory Reference Ranges | | SAC |
| 39. | All Subjects | CP_LB5 | Listing of Laboratory Values Outside Normal Reference Range | | SAC |
| ECG | | | | | |
| 40. | All Subjects | CP_EG5 | Listing of All ECG findings for Subjects with an Abnormal Finding | | SAC |
| PK | | | | | |
| 41. | PK | PK07 | Listing of Individual Subjects Plasma Concentrations at all time points | | SAC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| PD/Bio | markers | | | | |
| 42. | All subjects | PII115119/<br>Part A/Listing<br>25 | Listing of Sputum Collection | Include sample ID if available | SAC |
| 43. | All subjects | PII115119/<br>Part A/Listing<br>26 | Listing of Blood Collection for RNA | | SAC |
| 44. | All subjects | PII115119/<br>Part A/Listing<br>31 | Listing of Cell Count Data | | SAC |
| 45. | All subjects | PII115119/<br>Part A/Listing<br>32 | Listing of PMNs Differentials | | SAC |
| 46. | All subjects | PII115119/<br>Part A/Listing<br>34 | Listing of Individual Subject Inflammatory Cytokine Biomarker Data | | SAC |
| 47. | All subjects | PII115119/<br>Part A/Listing<br>35 | Listing of Microbiome (16S rRNA) Biomarker Data | | SAC |
| 48. | All subjects | PII115119/<br>Part A/Listing<br>36 | Listing of qPCR Data | | SAC |
| 49. | All subjects | PII115119/<br>Part A/Listing<br>37 | Listing of Bacterial Culture Data | | SAC |

#### The GlaxoSmithKline group of companies

201928

| Division | : Worldwide Development | |
|---|---|---|
| Information Type | : Reporting and Analysis Plan (RAP) - Critical Components | • |

| Title | : | Critical Components of Reporting and Analysis Plan for Study 201928: A randomised, double-blind, placebo-controlled study to evaluate the safety, efficacy and changes in induced sputum and blood biomarkers following daily repeat doses of inhaled GSK2269557 for 12 weeks in adult subjects diagnosed with an acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD) |
|---|---|---|
| Compound Number | : | GSK2269557 |
| Effective Date | : | 25-SEP-2015 |

#### **Description:**

The purpose of this CC-RAP (Critical Components of the Reporting and Analysis Plan) is to capture the following Critical Components, by First Subject First Visit:

- Analysis Population
- Protocol Deviations (Reflect the agreements from the plan for managing protocol deviations and define the reporting & analysis of all important deviations, as defined in the ICH guidelines)
- Statistical Evaluation (Primary/critical endpoints) and Statistical Analysis Considerations

#### Author's Name and Functional Area:

| PPD | | 25 CED 2015 |
|------------------------|-------------------------|-------------|
| Principal Statistician | n (Clinical Statistics) | 25-SEP-2015 |

Copyright 2015 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

201928

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | ANAL | YSIS PO | PULATIONS | 3 |
| | 1.1. | | ol Deviations | |
| _ | | | | |
| 2. | | IARY STA | ATISTICAL ANALYSES | 4 |
| | 2.1. | | acodynamic / Biomarker Analyses | 4 |
| | | 2.1.1. | Overview of Planned Pharmacodynamic / Biomarker | |
| | | | Analyses | 4 |
| | | 2.1.2. | Planned Pharmacodynamic / Biomarker Statistical | |
| | | | Analyses | 4 |
| 3. | SECO | ONDARY | STATISTICAL ANALYSES | 5 |
| Ο. | 3.1. | | acodynamic / Biomarker Analyses | |
| | 5.1. | 3.1.1. | | |
| | | 3.1.1. | Analyses | 5 |
| | | 3.1.2. | Planned Pharmacodynamic / Biomarker Statistical | |
| | | 3.1.2. | | _ |
| | 2.0 | C-f-t- | Analyses | 5 |
| | 3.2. | • | Analyses | |
| | 0.0 | 3.2.1. | - · | |
| | 3.3. | | acokinetic Analyses | |
| | | 3.3.1. | Overview of Planned Pharmacokinetic Analyses | |
| | 3.4. | | y Analyses | |
| | | 3.4.1. | | |
| | | 3.4.2. | Planned Efficacy Statistical Analyses | 9 |
| 4. | OTHE | R STATI | ISTICAL ANALYSES | 11 |
| ••• | 4.1. | | atory Pharmacodynamic / Biomarker Analyses | |
| | | 4.1.1. | Overview of Planned Exploratory Pharmacodynamic / | |
| | | | Biomarker Analyses | |
| | | 4.1.2. | Planned Exploratory Pharmacodynamic / Biomarker | |
| | | 4.1.2. | Statistical Analyses | 11 |
| | | | Statistical At 1817585 | |

201928

#### 1. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All subjects who were screened. | <ul> <li>Demography</li> <li>Screening failure details</li> <li>Eligibility criteria</li> <li>Protocol Deviations</li> <li>Serious adverse events</li> </ul> |
| All subject | <ul> <li>All randomised subjects who receive at least<br/>one dose of the study treatment.</li> <li>This population will be based on the<br/>treatment the subject actually received.</li> </ul> | <ul><li>Study Population</li><li>Pharmacodynamics</li><li>Safety</li><li>Efficacy</li></ul> |
| Pharmacokinetic | <ul> <li>Subjects in the 'All subject' population for<br/>whom a pharmacokinetic sample was<br/>obtained and analysed.</li> </ul> | • PK |

## 1.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

201928

#### 2. PRIMARY STATISTICAL ANALYSES

## 2.1. Pharmacodynamic / Biomarker Analyses

#### 2.1.1. Overview of Planned Pharmacodynamic / Biomarker Analyses

The pharmacodynamic analyses will be based on the "All Subjects" population, unless otherwise specified.

## 2.1.2. Planned Pharmacodynamic / Biomarker Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

 Alterations in the previously identified immune cell mechanisms specifically related to Neutrophil function as determined by changes in mRNA transcriptomics in induced sputum after 12, 28 and 84 days of treatment.

#### **Model Specification**

- The analyses proposed in this section may be adapted before database freeze, in the light of emerging findings from other studies.
- The analysis will be conducted by Target Sciences statistics, GSK.
- The mRNA data gives results from 54000 genes captured through >54000 probe sets. The subset of these 54000 genes which comprise the primary endpoint data will be specified in advance of DBF.
- For each probe set, repeated measures modelling (using measurements taken at Screening, Day 12, Day 28 and Day 84) will be used to estimate differences in mRNA intensities between treatment groups.
- Back transformed screening-adjusted means along with 95% CIs will be calculated for each treatment group and timepoint. Additionally, screening-adjusted fold changes between GSK2269557 1000 mcg and placebo will be calculated for Day 12, Day 28, and Day 84 along with 95% CI and p-values.
- A spreadsheet containing the output from each model for all probe sets in scope for the primary analysis will be generated and ranked by p-value for the comparison GSK2269557 1000 mcg vs. Placebo at Day 84. A separate tab in the spreadsheet will only include probe sets where the p-value for the comparison GSK2269557 1000mcg vs. placebo, is <0.05 (this cut-off criteria may be relaxed slightly if few probe sets are selected). Such probe sets will be ranked by fold change, with the expectation that, in general, a greater than a 1.5 fold change is scientifically meaningful.</p>
- Following review by the study team of the results, a subset of probe sets will be identified and included in an Excel file for further reporting.

#### **Model Checking**

• Details of Model Checking and Diagnostics for Statistical Analyses will be provided in the full RAP.

201928

## 3. SECONDARY STATISTICAL ANALYSES

## 3.1. Pharmacodynamic / Biomarker Analyses

## 3.1.1. Overview of Planned Pharmacodynamic / Biomarker Analyses

The pharmacodynamic analyses will be based on the "All Subjects" population, unless otherwise specified.

#### 3.1.2. Planned Pharmacodynamic / Biomarker Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

 Change from baseline in siVaw, iVaw, iRaw, siRAW, total lung capacity, lung lobar volumes, trachea length and diameter at FRC and TLC after 12 days of treatment and after 28 days of treatment.

The analyses proposed in this section may be adapted before database freeze, in the light of emerging findings from other studies.

#### Imaging:

The HRCT scans will be conducted at Screening, Day 12 and Day 28 (longitudinal in nature). However due to positioning of subjects whilst taking a scan, it can be that some airways are visible in some scans and not in other scans. For these reasons some HRCT imaging endpoints will be calculated to include only airways that are visible in both scans. For example the schematic below shows visible airways on Screening alone and Day 12 alone. It then shows the airways that are visible on both Screening & Day 12 scans, through removing/trimming airways that are not present in both scans.

#### Screening:



Scan Trimming Screening & Day 12:



For such reasons, the table below shows the HRCT endpoints and the results that will be captured

| | Lo | ongitudinal | | Scan Trimming, based on: | | |
|---|---|---|---|---|---|---|
| Endpoints | Screening | Day 12 | Day 28 | Screening and | Screening and | Day 12 and |
| | | | | Day 12 scans | Day 28 scans | Day 28 scans |
| iVaw | Х | Χ | Х | x (Screening) | x (Screening) | x (day12) |
| | | | | x (day 12) | x (day 28) | x (day 28) |
| siVaw | Х | Χ | Х | x (Screening) | x (Screening) | x (day12) |
| | | | | x (day 12) | x (day 28) | x (day 28) |
| iRaw | | | | x (Screening) | x (Screening) | x (day12) |
| | | | | x (day 12) | x (day 28) | x (day 28) |
| siRaw | | | | x (Screening) | x (Screening) | x (day12) |
| | | | | x (day 12) | x (day 28) | x (day 28) |
| iVlobe | X | Χ | Х | | | |
| iVlobe Pred | Х | Х | Х | | | |

201928

| Pla | Planned Statistical Analyses | | | |
|-----|------------------------------|---|---|---|
| | Trachea length | Х | х | Х |
| | Trachea<br>Diameter | X | Х | Х |

#### **Model Specification**

#### Imaging Endpoints with longitudinal data (iVaw, siVaw, iVlobe, ivlobe Pred)

- The data will be inspected during statistical analysis to determine whether a data transformation is required. It is likely that the data will approximately follow a lognormal distribution (for the iVaw and siVaw) and a log transformation with an offset (for the iRaw and siRaw); however the most appropriate distribution should be used.
- It is thought that the use of bronchodilators could affect the HRCT results. The database will
  contain information on whether or not relief medication was used in the 4h prior to each scan,
  and this information may be used in sensitivity analyses of the HRCT results.
- The FRC and TLC will be analysed in separate statistical models.
- The change from baseline (where baseline is screening) will be analysed in a multivariate model to account for the correlation between the multiple Regions (Total, Lower, Upper, Central and Distal), under a Bayesian framework. The model will have a separate intercept for each Region (by fitting a class parameter, and having no overall intercept) and will also include a baseline\*Visit\*Region and a Treatment\*Visit\*Region parameter. The Visit will consist of two levels: Day 12 and Day 28, and the Treatment will consist of two levels: GSK2269557 1000 mcg and Placebo. The Region will consist of 5 levels: Total, Lower, Upper, Central and Distal, however note that if one of the Regions is a linear combination of other Regions then only non linear combination Regions should be fitted, however all results (e.g Treatment medians and differences) for that particular Region should be retrospectively calculated though the known linear combination. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The change from baseline across the different Visits and Regions (accounting for the average baseline associated to the Region of interest) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% equi-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios if applicable.
- The difference between the treatment arms, for the change from baseline across the different Visits and Regions will be represented via adjusted posterior medians, as well as their associated 95% equi-tailed credible intervals. These results will be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios if applicable. For parameters that require a log transformation with an offset, for each posterior sample (i) appropriately back transformed values will be calculated for each treatment arms, and then (ii) using these back transformed values, the ratio of the treatment arms (Active/Placebo) will be calculated for each posterior sample, and finally summarised accordingly.
- The probabilities that the true treatment ratio is greater than 1, in addition to any other values

201928

#### **Planned Statistical Analyses**

appropriately selected based on the data, will also be computed for each Visit and Region. These results will be presented in tabular format.

## Imaging Endpoints with Scan Trimming (iVaw, siVaw, iRaw, siRaw)

- It is likely that the data will approximately follow a lognormal distribution (for the iVaw and siVaw) and a log transformation with an offset (for the iRaw and siRaw); however the most appropriate distribution should be used.
- The FRC and TLC will be analysed in separate statistical models.
- The responses of interest are the change from baseline based on (i) Airways present on scans taken at Screening and Day 12, (ii) Airways present on scans taken at Screening and Day 28, and (iii) Airways present on scans taken at Screening and Day 28. The baselines for each of these endpoints are provided in the table below.

| | (i) Screening &<br>Day12 Scan trimming | (ii) Screening &<br>Day28 Scan trimming | (iii) Day 12 & Day 28<br>Scan trimming |
|---|---|---|---|
| Screening Result | √ (baseline) | √ (baseline) | |
| Day 12 Result | √ (postdose) | | √ (baseline) |
| Day 28 Result | | √ (postdose) | √ (postdose) |

- The modeling below assumes that the Scan trimming endpoints (Screening&Day12, Screening&Day28 and Day12&Day28) will be analysed in a single multivariate model. This is subject to sensitivity analysis.
- The change from baseline (where baseline is defined in the table above) will be analysed in a multivariate model to account for the correlation between the multiple Scan Trimmings (Screening&Day12, Screening&Day28 and Day12&Day28) and Regions (Total, Lower, Upper, Central and Distal), under a Bayesian framework. The model will have a separate intercept for each Region and Scan Trimming combination (by fitting a class parameter Region\*ScanTrimming, and having no overall intercept), and will also include a baseline\*ScanTrimming\*Region and a Treatment\*ScanTrimming\*Region parameter. The Visit will consist of two levels: Day 12 and Day 28, the scan trimming will consist of three levels Screening&Day12, Screening&Day28 and Day12&Day28, and the Treatment will consist of two levels: GSK2269557 1000 mcg and Placebo. The Region will consist of 5 levels: Total, Lower, Upper, Central and Distal, however note that if one of the Regions is a linear combination of other Regions then only non linear combination Regions should be fitted, however all results (e.g. Treatment medians and differences) for that particular Region should be retrospectively calculated though the known linear combination. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e. covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The change from baseline across the different Scan Trimmings and Regions (accounting for the average baseline associated to the Region of interest) will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% equi-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios if applicable.

201928

## **Planned Statistical Analyses**

- The difference between the treatment arms, for the change from baseline across the different Scan Trimming and Regions will be represented via adjusted posterior medians, as well as their associated 95% equi-tailed credible intervals. These results will also be presented in tabular form, and will be presented after the data have been appropriately back transformed to give median ratios if applicable. For parameters that require a log transformation with an offset, for each posterior sample (i) appropriately back transformed values will be calculated for each treatment arm, and then (ii) using these back transformed values, the ratio of the treatment arms (Active/Placebo) will be calculated for each posterior sample, and finally summarised accordingly.
- The probabilities that the true treatment ratio is greater than 1, in addition to other values appropriately selected based on the data, will also be computed for each Visit and Region. These results will be presented in tabular format.

#### **Trachea Length and Diameter**

- The data will be inspected during statistical analysis to determine whether a data transformation is required.
- The FRC and TLC will be analysed in separate statistical models.
- The data will be analysed in a multivariate model to account for the correlation between the multiple endpoints ((i)Trachea length and (ii) Trachea Diameter), under a Bayesian framework. The model will have separate intercepts for each endpoint (by fitting a class variable "Endpoint", and having no overall intercept), and will also include a baseline\*Visit\*Endpoint and a Treatment\*Visit\*Endpoint parameter. The Visit will consist of two levels: Day 12 and Day 28, the Treatment will consist of two levels: GSK2269557 1000 mcg and Placebo, whilst the Endpoint will consist of two levels: Trachea Length and Diameter. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.
- The predicted values across the different Endpoints and Visits will be represented via adjusted
  posterior medians for each of the Treatment Arms, as well as their associated 95% equi-tailed
  credible intervals. These results will also be presented in a tabular format.
- The difference between the treatment arms across the different Endpoints and Visits will be represented via adjusted posterior medians, as well as their associated 95% equi-tailed credible intervals. These results will also be presented in a tabular format.
- Through the use of a Bayesian framework, for each posterior sample the following will be calculated:
  - The predicted Trachea Length (for each Visit and Treatment for an average baseline)
  - The predicted Trachea Diameter (for each Visit and Treatment for an average baseline)
- The predicted Trachea length (1.) for each Visit and Treatment will be divided by the predicted Diameter (2.). This will be summarised and represented through calculating a posterior median, with 95% equi-tailed credible intervals. These results will also be presented in a tabular format.
- The difference between Treatment Arms (at each Visit) for the predicted Trachea / Diameter Ratio will be calculated using the posterior samples (generated in the bullet point above). This

201928

#### **Planned Statistical Analyses**

will be summarised and represented through calculating a posterior median, with 95% equitailed credible intervals. These results will also be presented in a tabular format.

#### **Model Checking**

• Details of Model Checking and Diagnostics for Statistical Analyses will be provided in the full RAP.

## 3.2. Safety Analyses

## 3.2.1. Overview of Planned Analyses

The safety analyses will be based on the "All Subjects" population, unless otherwise specified. Details of the analyses of safety data will be included in the full RAP.

# 3.3. Pharmacokinetic Analyses

#### 3.3.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic" population, unless otherwise specified. Details of the analyses of PK data will be included in the full RAP.

## 3.4. Efficacy Analyses

## 3.4.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the "All Subjects" population, unless otherwise specified.

#### 3.4.2. Planned Efficacy Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

- FEV<sub>1 and</sub> FVC at clinic prior to sputum induction
- Daily PEF
- Daily reliever usage

# Model Specification

#### FEV<sub>1</sub> (L) and FVC (L) at clinic prior to sputum induction

- The data will be inspected prior to analysis to determine whether a data transformation is required.
- The analysis will include all available values. If there are values which were recorded within 4h
  after the subject had taken relief medication, a sensitivity analysis may be done which
  excludes these values.
- The endpoints (FEV<sub>1</sub>,and FVC) will be analysed in separate statistical models. The change from baseline in the endpoint will be analysed in a Bayesian repeated measures model, with a baseline by Visit covariate and Treatment by Visit class parameter. The Treatment will have

201928

## **Planned Statistical Analyses**

two levels: GSK2269557 1000 mcg and Placebo, and the Visit will have two levels: Day 12 and Day 28. No fixed assumption around the structure of the covariance matrix will be enforced. The priors for the mean vector for each of the parameters (i.e covariates) will each follow a normal distribution and the prior for the variance-covariance will follow an inverse Wishart distribution. Sensitivity analysis will be conducted to select appropriate parameters for both distributions such that the priors are non-informative with respect to the posterior.

- The change from baseline at each of the Visits will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% equi-tailed credible intervals. These results will also be presented in a tabular format.
- The difference between the treatment arms, for the change from baseline will be represented via adjusted posterior medians for each of the Treatment Arms, as well as their associated 95% equi-tailed credible intervals. These results will also be presented in a tabular format.
- The probabilities that the treatment difference is greater than 0 (or 1, if a lognormal distribution is used) will also be computed at each Visit, in addition to any other values appropriately selected based on the data. These results will be presented in tabular format.

#### **Daily PEF**

Mean and 95% CIs of AM PEF readings will be plotted by study treatment vs. Study Day

#### Reliever usage

- A reliever medication-free day is defined for statistical analysis as a 24-hour period in which the number of relief medication inhalations is zero.
- The number of occasions per day on which reliever medication was used will be averaged per
  day and plotted in the same way as the PEF daily endpoint above. If the data are non-normally
  distributed then the median and upper and lower quartiles will be plotted instead of the mean
  and 95% CIs. The percentage of reliever medication free days will be calculated over the
  treatment period and summarised by study treatment.

#### **Model Checking & Diagnostics**

Details of Model Checking and Diagnostics for Statistical Analyses will be provided in the full RAP.

201928

#### 4. OTHER STATISTICAL ANALYSES

## 4.1. Exploratory Pharmacodynamic / Biomarker Analyses

# 4.1.1. Overview of Planned Exploratory Pharmacodynamic / Biomarker Analyses

The exploratory pharmacodynamic/biomarker analyses will be based on the "All Subjects" population, unless otherwise specified.

# 4.1.2. Planned Exploratory Pharmacodynamic / Biomarker Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

- Alterations in immune cell mechanisms as determined by changes in mRNA transcriptomics in induced sputum or blood after 12, 28 and 84 days of treatment.
- Induced sputum endpoints may include, but are not limited to cytokines (IL-6, IL-8, TNFα), microbiome (by 16SrRNA), bacterial qPCR, viral qPCR.
- Change from baseline for other CT parameters including low attenuation score after 12 days of treatment and after 28 days of treatment.
- Correlations of sputum biomarker data with CT parameters.

The table below shows the exploratory HRCT endpoints and the results that will be captured:

| | Lo | ongitudinal | | Scan Trimming, based on: | | |
|---|---|---|---|---|---|---|
| Endpoints | Screening | Day 12 | Day 28 | Screening and<br>Day 12 scans | Screening and<br>Day 28 scans | Day 12 and<br>Day 28 scans |
| IALD | Х | Х | Х | | | |
| LAS | Х | Х | Х | | | |
| AT | X | Х | Χ | | | |
| BVD | Х | Х | Х | | | |
| iVaww | | | | x (Screening)<br>x (day 12) | x (Screening)<br>x (day 28) | x (day12)<br>x (day 28) |
| siVaww | | | | x (Screening)<br>x (day 12) | x (Screening)<br>x (day 28) | x (day12)<br>x (day 28) |

#### **Model Specification**

- Analyses for mRNA (from induced sputum and blood) and further CT endpoints will follow the
  methods outlined for the corresponding primary and secondary endpoints respectively, or as
  appropriate to the type of endpoint. Details will be covered in the full RAP. As noted in the
  above sections, the analyses proposed for these endpoints may be adapted before database
  freeze, in the light of emerging findings from other studies. The analysis of induced sputum
  parameters will be described in the full RAP.
- An outline plan for correlations of sputum biomarker data with CT parameters will be included in the full RAP.
- As these analyses are exploratory in nature, additional non-RAP-specified analyses may be performed.